## **Statistical Analysis Plan**

**Study ID:** 221853

Official Title of Study: A PHASE 1, 2-PART, OPEN-LABEL, FIXED-SEQUENCE STUDY EVALUATING THE EFFECT OF RIFAMPIN (PART 1) AND RABEPRAZOLE (PART 2) ON THE PHARMACOKINETICS OF A SINGLE DOSE OF CAMLIPIXANT (BLU-5937) 50 mg TABLET IN HEALTHY PARTICIPANTS UNDER FASTING CONDITIONS

**Date of Document:** 02-Nov-2023

## 16.1.2 Reporting and Analysis Plan

| Table of conter | ıts | |
|------------------|-----------------------------------------------------|----|
| 16.1.2 | Reporting and Analysis Plan | 1 |
| Table of conter | nts | 1 |
| Statistical Anal | ysis Plan 1.0 dated 04-OCT-2023 | 2 |
| Statistical Anal | ysis Plan (Table/Figure/Listing Shells) Version 1.0 | |
| dated 2 | S_OCT_2023 | 32 |

# Statistical Analysis Plan 1.0 dated 04-OCT-2023



## **Statistical Analysis Plan for Interventional Studies (Early Phase)**

Sponsor Name: Bellus Health

Protocol Number: 220254 (BUS-P1-11)

**Protocol Title:** A Phase 1, 2-Part, Open-label, Fixed-sequence Study Evaluating the Effect of Rifampin (Part 1) and Rabeprazole (Part 2) on the Pharmacokinetics of a Single Dose of Camlipixant (BLU-5937) 50 mg Tablet in Healthy Participants under Fasting Conditions

**Protocol Version and Date:** Final, 03-Apr-2023

Sponsor Study Number: BUS-P1-11

Authors: PPD , Senior Principal Biostatistician

, Technical Writer

## **Notice of Confidential and Proprietary Information:**

The information contained in this document is confidential belonging to Bellus Health. Acceptance of this document constitutes agreement by the recipient that no information contained herein will be published or disclosed without prior written authorization from an official of Bellus Health. However, this document may be disclosed to the appropriate Institutional Review Board and ethics committees or duly authorized representatives of a national regulatory authority under the condition that they are requested to keep it confidential. In the event of an actual or suspected breach of this obligation, Syneos Health should be notified promptly.

This document is confidential.

SAP Version: Final 1.0 04-Oct-2023

Controlled Document ID: 2805A.00, Effective Date 29-Jul-2019

Filing requirements: TMF 

## **Revision History**

| Version | Date<br>(DD-Mmm-YYYY) | <b>Document Owner</b> | Revision Summary |
|-----------|-----------------------|-----------------------|------------------|
| Final 1.0 | 04-Oct-2023 | PPD | Final version |

## Approvals

I confirm that I have reviewed this document and agree with the content.

| Syneos Health Approval | | |
|---|---|---|
| PPD , Senior Principal Biostatistician | PPD | 04-Oct-2023 |
| Name, Title<br>Lead Biostatistician | Signature PPD | Date<br>(DD-Mmm-YYYY) |
| PPD , Sr. Biostatistician | | 05-Oct-2023 |
| Name, Title<br>Senior Reviewing Biostatistician | Signature | Date<br>(DD-Mmm-YYYY) |
| PPD , Senior Pharmacokineticist | PPD | 04-Oct-2023 |
| Name, Title<br>Lead Pharmacokineticist | Signature | Date<br>(DD-Mmm-YYYY) |
| PPD , Medical Writer II | | 05-Oct-2023 |
| Name, Title<br>Lead Medical Writer | Signature | Date<br>(DD-Mmm-YYYY) |
| <b>Bellus Health Approval</b> | | |
| PPD , Ph.D., | PPD | |
| PPD , Head of Biostatistics | | 04-Oct-2023 |
| Name, Title<br>Sponsor Contact | Signature | Date (DD-Mmm-YYYY) |
| M.Sc., PP, Early Phase Development, PHead of Drug Development | PPD | 04-Oct-2023 |
| Name, Title<br>Sponsor Contact | Signature | Date<br>(DD-Mmm-YYYY) |
| PPD of Clinical Pharmacology | | 04-Oct-2023 |
| Name, Title<br>Sponsor Contact | Signature | Date<br>(DD-Mmm-YYYY) |

This document is confidential.

## **Table of Contents**

| Revisio | on History | .2 |
|---------|-------------------------------------------------|----|
| Approv | vals | .3 |
| Table o | of Contents | .4 |
| Glossa | ry of Abbreviations | .6 |
| 1. Pu | rpose | .8 |
| 1.1 | Responsibilities | .8 |
| 1.2 | Timings of Analyses | .8 |
| 2. Stu | udy Objectives | .8 |
| 3. Stu | udy Description | .9 |
| 3.1 | Subject Selection | .9 |
| 3.2 | Determination of Sample Size | .9 |
| 3.3 | Treatment Assignment | .9 |
| 3.4 | Randomization and Blinding | 10 |
| 3.5 | Participant Withdrawal and Replacement | 10 |
| 4. En | dpoints | 10 |
| 5. Ar | nalysis Populations | 10 |
| 5.1 | Safety Population | 11 |
| 5.2 | Pharmacokinetic Concentration Population | 11 |
| 5.3 | Pharmacokinetic Parameter Population | 11 |
| 5.4 | Pharmacogenomic Population | 11 |
| 6. Ge | eneral Aspects for Statistical Analysis | |
| 6.1 | General Methods. | 11 |
| 6.2 | Summary Statistics: | 13 |
| 6.3 | Key Definitions. | 13 |
| 6.4 | Missing Data | 14 |
| 7. Stu | udy Population | 15 |
| 7.1 | Subject Disposition. | |
| 7.2 | Protocol Deviations | 15 |
| 7.3 | Inclusion and Exclusion Criteria | |
| 7.4 | Demographics and Other Baseline Characteristics | 15 |
| 7.5 | Medical History | 16 |
| 7.6 | Medications | |
| 7.7 | Drug, Cotinine, and Alcohol Screens | |
| 7.8 | Pregnancy Screening | |
| 7.9 | Additional Screening Tests | 16 |
| 8. Ph | armacokinetic (PK) Analyses | 16 |
| 8.1 | Data Handling | |
| 8.1 | | |
| 8.1 | 1.2 Data Presentation Rules | |
| 8.2 | Pharmacokinetic (PK) Parameters | |
| 8.3 | Assessment of Rifampin Effect (Part 1) | |
| 8.4 | Assessment of Rabeprazole Effect (Part 2) | |
| 8.5 | Attainment of Steady State | 20 |

This document is confidential.


Controlled Document ID: 2805A.00, Effective Date 29-Jul-2019

| 9. Pharmacogenomic Analyses | 20 |
|---------------------------------------------------|----|
| 10. Safety | |
| 10.1 Exposure | |
| 10.2 Adverse Events (AEs) | |
| 10.3 Laboratory Evaluations | |
| 10.4 Vital Signs | |
| 10.5 Electrocardiograms (ECGs) | |
| 10.6 Physical Examination | |
| 11. Changes from Analysis Planned in the Protocol | |
| 12. Programming Considerations | |
| 12.1 General Considerations. | |
| 12.2 Table, Listing, and Figure Format | |
| 12.2.1 General | |
| 12.2.2 Headers and Footers | |
| 12.2.3 Display Titles | |
| 12.2.4 Column and Row Headings | |
| 12.2.5 Body of the Data Display | |
| 12.2.6 Footnotes | |
| 13. Quality Control | |
| 14. Reference List | |

## **Glossary of Abbreviations**

| Abbreviation | Description |
|---|---|
| AE | adverse event |
| AEMI | adverse event of medical interest |
| ANOVA | analysis of variance |
| ATC | anatomical therapeutic chemical |
| AUC | area under the concentration-time curve |
| AUC <sub>0-inf</sub> | area under the concentration-time curve from time zero to infinity, extrapolated |
| AUC <sub>0-t</sub> | area under the concentration-time curve from time zero until the last observed concentration |
| BLQ | below the lower limit of quantification |
| BMI | body mass index |
| CFR | Code of Federal Regulations |
| CI | confidence interval |
| Cl/F | apparent clearance |
| C <sub>max</sub> | maximal observed concentration |
| COVID-19 | coronavirus 2019 |
| CSR | clinical study report |
| CV | coefficient of variation |
| CYP | cytochrome P450 |
| DDI | drug-drug interaction |
| ECG | electrocardiogram |
| eCRF | electronic case report form |
| FDA | Food and Drug Administration |
| FSH | follicle-stimulating hormone |
| ICH | International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use |
| Kel | terminal elimination rate constant |
| Kel Lower | the timepoint where In-linear Kel calculation begins |
| Kel Upper | the actual sampling time of the last measurable concentration used to estimate the $K_{\text{el}}$ |
| LLOQ | lower limit of quantification |
| ln | natural logarithm |
| max | maximum |
| MedDRA® | Medical Dictionary for Regulatory Activities |

This document is confidential.


Controlled Document ID: 2805A.00, Effective Date 29-Jul-2019

| Abbreviation | Description |
|-------------------|--------------------------------------------------|
| min | minimum |
| N | number of subjects |
| n | number of observations |
| N/A | not applicable |
| NC | not calculated |
| NR | no result or not reportable |
| NS | no sample |
| PC | pharmacokinetic concentration |
| PK | pharmacokinetic(s) |
| PPI | proton-pump inhibitor |
| PT | preferred term |
| p-value | probability value |
| CCI | |
| $\mathbb{R}^2$ | R-squared |
| SAE | serious adverse event |
| SAP | statistical analysis plan |
| SD | standard deviation |
| SOC | system organ class |
| SOP | standard operation procedure |
| T½ el | terminal elimination half-life |
| TEAE | treatment-emergent adverse event |
| TFLs | tables, figures, and listings |
| $T_{\text{max}}$ | time when the maximal concentration is observed |
| V <sub>z</sub> /F | apparent volume of distribution |
| WHO DD | World Health Organization Global Drug Dictionary |

## 1. Purpose

The purpose of this statistical analysis plan (SAP) is to ensure that the data listings, summary tables, and figures which will be produced, and the statistical methodologies that will be used, are complete and appropriate to allow valid conclusions regarding the study objectives.

This SAP is based on the following documents:

- Protocol 220254 (BUS-P1-11) Final, dated 03-Apr-2023
- Protocol administrative letters dated 13-Jun-2023 and 20-Jul-2023
- Electronic case report form (eCRF) version 1.00, dated 11-Jul-2023

The plan may change due to unforeseen circumstances; any changes made after the plan has been finalized will be documented. No revision to the SAP is required for changes which do not affect the statistical analysis methods, definitions, or rules defined in this document. If additional analyses are required to supplement the planned analyses described in the SAP, the changes and justification for the changes will be outlined in the associated clinical study report (CSR). No change will be made without prior written approval of the Sponsor.

When applicable, all methodologies and related processes will be conducted according to Syneos Health's standard operating procedures (SOPs), as appropriate. Shells for all statistical tables, listings, and figures referred to in this SAP will be presented in a separate document.

#### 1.1 Responsibilities

Syneos Health will perform the statistical analyses and is responsible for the production and quality control of all tables, figures, and listings (TFLs).

## 1.2 Timings of Analyses

The final safety, tolerability, and pharmacokinetic (PK) analysis will be completed after all subjects complete the final study visit or discontinue from the study.

#### 2. Study Objectives

- Primary Objectives:
  - To assess the effect of repeated oral doses of rifampin, a cytochrome P450 (CYP) 3A4 and collection inducer (Part 1), or rabeprazole, a proton-pump inhibitor (PPI) (Part 2), on the PK of a single oral dose of camlipixant (BLU-5937), administered to healthy participants.
- Secondary Objectives:
  - o To evaluate the safety and tolerability of camlipixant when administered alone and in combination with rifampin or rabeprazole to healthy participants.

## 3. Study Description

This is a single-center, 2-part, Phase 1, open-label, fixed-sequence, drug-drug interaction (DDI) study designed to compare the PK of camlipixant when administered with and without rifampin (Part 1) or rabeprazole (Part 2) in healthy participants under fasting conditions. The start of study conduct for Part 2 is independent from Part 1 study conduct.

Participants will be enrolled to either Part 1 or Part 2. In each part, participants will receive the assigned treatment.

#### 3.1 Subject Selection

A total of 32 healthy, non-smoking participants,  $\geq$ 18 and  $\leq$ 55 years of age, with body mass index (BMI) >18.5 and  $\leq$ 30.0 kg/m², and body weight  $\geq$ 50.0 kg for males and  $\geq$ 45.0 kg for females, are planned to be enrolled in this study. In Part 1, a total of 16 healthy males and non-childbearing potential females are to be enrolled. In Part 2, a total of 16 healthy males and females are to be enrolled.

#### 3.2 Determination of Sample Size

It is planned to enroll up to 16 participants in Part 1 and 16 participants in Part 2 for participation in this study (total of 32 participants) in order to have at least 12 evaluable participants for PK analysis in each part of the study. No formal sample size calculation has been made. Based on experience from previous similar studies, a total of 32 participants (16 in each study part) was considered sufficient to adequately characterize the PK potential for a clinical DDI.

## 3.3 Treatment Assignment

In each study part, subjects will receive the assigned treatment according to the fixed-sequence scheme described below.

In Part 1, subjects will receive a single oral dose of camlipixant on Day 1, followed by a 3-day washout period. Repeated oral doses of rifampin will be administered continuous on Days 4 through 12, with co-administration of a single oral dose of camlipixant with rifampin on Day 11.

In Part 2, subjects will receive a single oral dose of camlipixant on Day 1, followed by a 3-day washout period. Common oral doses of rabeprazole will be administered on Days 4 through 11, with co-administration of a single oral dose of camlipixant with rabeprazole on Day 10.

The planned dose levels and regimens are summarized in Table 3.3-1, below.

**Table 3.3-1: Treatment Regimen** 

| <b>Study Part</b> | Study Day(s) | Treatment(s) |
|---|---|---|
| Day 1 | | 1 x 50 mg camlipixant tablet |
| Part 1 | Days 4-12 | mg rifampin capsules (total dose cor mg) |
| rait i | Day 11 | mg rifampin capsules (total dose col mg) col and 1 x 50 mg camlipixant tablet [1 hour (± 2 minutes) after rifampin] |
| Day 1 | | 1 x 50 mg camlipixant tablet |
| Part 2 | Days 4-11 | mg rabeprazole enteric-coated tablets |

This document is confidential.


Controlled Document ID: 2805A.00, Effective Date 29-Jul-2019



#### 3.4 Randomization and Blinding

This study will be an open-label study due to the objective nature of the data. Thus, no randomization and blinding measures will be applied. Participants will be administered each treatment according to the fixed-sequence scheme.

### 3.5 Participant Withdrawal and Replacement

Participants will be advised that they are free to withdraw from the study at any time. Over the course of the study, the Sponsor and the Investigator or designee may withdraw any participant from the study for one of the reasons described below; participant withdrawal will be done in accordance with the clinical site's SOP:

- Safety reason;
- Non-compliance with protocol requirements;
- Significant protocol deviation;
- Positive pregnancy test, drug screen, cotinine test, or alcohol breath test.

Participants who withdraw or are withdrawn from the study after dosing will not be replaced. However, in the event that the number of drop-outs exceeds initial expectations, participants who withdraw or are withdrawn might be replaced at the discretion of the Sponsor. Such replacement resulting in dosing more participants than planned in this protocol would be documented in a protocol amendment.

#### 4. Endpoints

- Primary Endpoints:
  - PK parameters: Area under the concentration-time curve from time zero to infinity, extrapolated (AUC<sub>0-inf</sub>), area under the concentration-time curve from time zero until the last observed concentration (AUC<sub>0-t</sub>), and maximal observed concentration (C<sub>max</sub>).
- Secondary Endpoints:
  - O PK parameters: Time when the maximal concentration is observed  $(T_{max})$ , terminal elimination half-life  $(T_{'2} \, el)$ , residual area, terminal elimination rate constant  $(K_{el})$ , apparent clearance (Cl/F), and apparent volume of distribution  $(V_z/F)$ .
  - Safety evaluation: Adverse events (AEs), serious AEs (SAEs), AEs of medical interest (AEMIs), vital signs measurements (blood pressure, heart rate, respiratory rate, and oral temperature), 12-lead electrocardiogram (ECG) recordings, physical examinations, and clinical laboratory test results, including hematology, biochemistry, coagulation, and urinalysis.


## 5. Analysis Populations

All participants' inclusion status into each analysis population will be determined after database lock and before the final analysis. Participants will be analyzed according to the treatment received.

This document is confidential.


Controlled Document ID: 2805A.00, Effective Date 29-Jul-2019

## 5.1 Safety Population

The safety population is defined as all participants who receive at least one dose of any study drug. The safety population will be used for all safety and tolerability summaries and analyses.

#### 5.2 Pharmacokinetic Concentration Population

The pharmacokinetic concentration (PC) population for camlipixant will include all participants who received at least one dose of camlipixant at Day 1 or Day 11 (Part 1)/Day 10 (Part 2) and have at least one reportable concentration. The PC population will be used for listing of concentrations.

### 5.3 Pharmacokinetic Parameter Population

The PK parameter population will include all participants for whom the Day 1 and Day 11 (Part 1) or Day 10 (Part 2) PK profiles of the victim drug, camlipixant, can be adequately characterized, specifically, when administered alone and in combination with rifampin (Part 1) or rabeprazole (Part 2). The PK parameters population will be used for all PK parameter summaries and analyses.

Any participant who experienced emesis during the sampling interval will be evaluated on a case-by-case basis in order to determine whether the participant will be excluded from the descriptive statistics and statistical analyses. Individual PK parameters from participant excluded from the PK parameter population will be presented in the listing but will be excluded from the descriptive statistics and statistical analyses.

Here are some aspects to be considered (but not to be limited to) when determining data availability for the PK population: inclusion and exclusion criteria, acceptable times for study days/timepoints and measurements, compliance with camlipixant treatment, compliance with rifampin (Part 1) or rabeprazole (Part 2) treatment impacting camlipixant PK (number of doses received equal to 9 [Part 1] or 8 [Part 2]), 1-hour time interval between rifampin and camlipixant dosing on Day 11 of Part 1 or 1-hour time interval between rabeprazole and camlipixant dosing on Day 10 of Part 2, the nature and quality of the data, withdrawal, and any protocol deviation. The final responsibility of deciding which participants are to be included or excluded lies with the Investigator and/or the Sponsor.

#### 5.4 Pharmacogenomic Population

The pharmacogenomic population will include all participants in the safety population who had at least one pharmacogenomic measurement data available.

#### 6. General Aspects for Statistical Analysis

#### 6.1 General Methods

software release 9.4 (or more recent version) will be used to perform all statistical analyses. All relevant data in the database will be presented in the data listings. Unless otherwise stated, all listings will be sorted by study part, subject number, and assessment date/time. All summaries will be presented separately for each study part. Unless otherwise stated, the descriptions of the analyses which follow will apply to all study parts.

This document is confidential.


Controlled Document ID: 2805A.00, Effective Date 29-Jul-2019

The following labels for treatment will be used on all tabulations where the results are displayed by treatment, in the following order:

- Part 1:
  - o Camlipixant
  - o Rifampin
  - o Camlipixant + Rifampin
- Part 2:
  - o Camlipixant
  - o Rabeprazole
  - Camlipixant + Rabeprazole

For Part 1, where applicable, the treatment phases considered for the safety summaries will be:

- Camlipixant alone from Day 1 post-dose until Day 4 pre-dose of rifampin;
- Rifampin alone from Day 4 dosing until Day 11 pre-dose of camlipixant;
- Rifampin + Camlipixant from camlipixant dosing on Day 11 until end of study.

For Part 2, where applicable, the treatment phases considered for the safety summaries will be:

- Camlipixant alone from Day 1 post-dose until Day 4 pre-dose of rabeprazole;
- Rabeprazole alone from Day 4 dosing until Day 10 pre-dose of camlipixant;
- Rabeprazole + Camlipixant from camlipixant dosing on Day 10 until end of study.

## **6.2** Summary Statistics:

Unless otherwise stated, continuous variables will be summarized using the number of observations (n), and the statistics mean, median, standard deviation (SD), minimum (min) and maximum (max). The min and max values will be presented to the same number of significant digits as recorded in the eCRF, mean and median will be presented to one more significant digit than the raw data, and the SD will be presented to two more significant digits than the raw data.

Summaries of change from baseline variables will include only subjects who have both a baseline value and corresponding value at the timepoint of interest. Categorical and binary variables will be summarized with frequency counts and percentages. Percentages will be rounded to one decimal place, with the denominator being the number of participants (N) in the relevant population, unless otherwise stated.

All digits will be used for PK and statistical calculations. For PK tables and listings, the final reportable results or data will be presented by rounding off to two decimal digits, except for the following situations (this applies to individual data and descriptive statistics):

- K<sub>el</sub> and R-squared (R<sup>2</sup>) adjusted data shall be rounded off to four decimal digits.
- PK parameters related to time, such as T<sub>max</sub>, the timepoint where In-linear K<sub>el</sub> calculation begins (K<sub>el Lower</sub>), and the actual sampling time of the last measurable concentration used to estimate the K<sub>el</sub> (K<sub>el Upper</sub>), must be reported with the same precision as the actual sampling time, rounded to three decimal digits.
- Concentration versus time data, as well as C<sub>max</sub> shall be reported as they appear in the corresponding dataset.
- Ratios and 90% CIs, intra- and inter-subject coefficients of variation (CV), and CV (%) will be presented to two decimal places.

Only data from protocol scheduled ("nominal") visits will be included in the summary tables. Data from unscheduled visits will not be included in the summary tables (unless they were used as baseline) but will be included in the listings.

#### 6.3 Key Definitions

#### Baseline:

Unless stated otherwise, baseline will be determined for each subject and will be defined as the last non-missing measurement (including repeated and unscheduled assessments) obtained prior to the first study drug administration. Post baseline will be considered as all measurements collected after first study drug administration. "Unknown", "Not Done", "Not Applicable" and other classifications of missing data will not be considered when calculating baseline observations unless the finding is a valid categorical observation.

#### Study Day:

Study day will be calculated using first study drug administration date as the reference date. If the date of interest occurs on or after the first study drug administration date, study day will be calculated as (date of interest – first study drug administration date) + 1. If the date of interest occurs prior to the first study drug administration date, study day will be calculated as (date of interest – first study drug administration date). There will be no study Day 0.

#### Prior and Concomitant Medications:

Prior medications are defined as medications that start and stop prior to the first dose of study drug. All other medications will be defined as concomitant medications including those that start prior to the first dose of study drug and continue thereafter. Any medications with an unknown start or stop date will be assumed to be concomitant medications unless a partial start or stop date indicates otherwise.

### 6.4 Missing Data

There will be no imputation for missing data, unless otherwise specified. Missing data shall be presented in subject listings as either "-" (unknown or not evaluated) or "N/A" (not applicable), with the corresponding definition in the footnotes. Missing descriptive statistics, or probability values (p-values), which cannot be estimated shall be presented as "-".

The listings will include the reported date/time, and the imputations rules below will be used if needed to classify as prior or concomitant medication, to determine if an AE is non-TEAE or TEAE, or to attribute to a particular treatment for the summaries.

For inclusion in concomitant medication tables, incomplete start and stop dates on the eCRF will be imputed as follows:

- If the start date is incomplete, the following rules will be applied:
  - o Missing day: Assume the first day of the month; however, if the partial date and the date of first study drug administration lie within the same month and year and the date of first study drug administration is not after the stop date of the event/medication, set to the date of study drug administration. Otherwise, set to the stop date of the event/medication.
  - O Missing day and month: Assume January 1<sup>st</sup>; however, if the partial date and the date of first study drug administration lie within the same year and the date of first study drug administration is not after the stop date of the event/medication, set to the date of first study drug administration. Otherwise, set to the stop date of the event/medication.
  - Missing day, month, and year: Assume date of first study drug administration if it
    is not after the stop date for the event/medication. Otherwise, set to the stop date
    for the event/medication.
- If the stop date is incomplete, the following rules will be applied:
  - o Missing day: Assume the last day of the month
  - o Missing day and month: Assume the last day of the year

This document is confidential.


Controlled Document ID: 2805A.00, Effective Date 29-Jul-2019

- o Missing day, month, and year: Assume that the event/medication is continuing
- o In the case of the death of a subject, and if the imputed end date is after the date of death, the end date will be imputed as the date of death.
- If the stop date is incomplete, imputed end date will be used instead of reported end date.

AEs without an onset date or time, or AEs with an onset date on the date of first study drug administration but without an onset time, will be defined as treatment-emergent, unless an incomplete date (e.g., month and year) clearly indicates that the event started prior to the first study drug administration, or the AE stop date indicates that the event started and stopped prior to the first study drug administration.

In the case of withdrawal of consent, all data from participants who withdraw from the study will be included in all summaries up to the time of withdrawal. For all other withdrawals, all data captured will be included in the safety summaries.

For PK analysis, only observed concentration data will be used in the data analysis except for concentration values below the lower limit of quantification (BLQ); see section 8.1. No attempt will be made to extrapolate or interpolate estimates for missing data.

## 7. Study Population

### 7.1 Subject Disposition

The number of participants who were screened, enrolled, dosed, completed the study, and discontinued from the study, along with reasons for discontinuation, will be summarized. The data will be presented by study part, treatment, and overall (frequency counts and the percentage) and presented by participant in a data listing.

#### 7.2 Protocol Deviations

Participant data will be examined for evidence of protocol deviations. All protocol deviations will be categorized (as critical, major or minor and important/non-important as per ICH E3 definition) and presented by participant in a data listing.

#### 7.3 Inclusion and Exclusion Criteria

All recorded inclusion and exclusion criteria status will be presented by participant in a data listing. Participant's inclusion or exclusion from each analysis population will also be presented in a data listing.

## 7.4 Demographics and Other Baseline Characteristics

All demographics and baseline body measurements will be summarized by study part and treatment for the safety, and PC and PK parameter populations (if different from safety population). All demographic characteristics will be presented by participant in a data listing.

Descriptive statistics (n, mean, SD, min, median, and max) will be calculated for continuous variables using the last results obtained (scheduled or unscheduled) prior to the first study drug administration. Frequency counts and percentages will be tabulated for categorical and binary variables.

This document is confidential.


Controlled Document ID: 2805A.00, Effective Date 29-Jul-2019

#### 7.5 Medical History

Medical history will be presented by participant in a data listing. The Medical Dictionary for Regulatory Activities (MedDRA), Version 26.0 (or more recent version) will be used to classify medical history terms by system organ class (SOC) and preferred term (PT). Output data will include the MedDRA version used in the study.

#### 7.6 Medications

Medications taken by participants that start and stop before first dosing will be documented as prior medications whereas medications taken by participants after dosing (including those that start prior to the first dosing and continue thereafter) up to follow-up phone call will be documented as concomitant medications. Prior and concomitant medications will be presented by participant in a data listing. The World Health Organization Global Drug Dictionary (WHO DD), Version B3, March 2023 (or more recent version) will be used to classify medications by anatomical therapeutic chemical (ATC) classification code (3rd level) and preferred name. When 3rd level classification code is not available, 2nd level classification will be used instead. Output data will include the WHO DD version used in the study.

#### 7.7 Drug, Cotinine, and Alcohol Screens

The results of urine drug, urine cotinine, and alcohol breath screen tests will be presented by participant in data listings.

#### 7.8 Pregnancy Screening

Pregnancy tests will be performed for all females. The follicle-stimulating hormone (FSH) level will be tested in postmenopausal females only. All results will be presented by participant in data listings.

#### 7.9 Additional Screening Tests

The results of serology tests and coronavirus 2019 (COVID-19) tests will be presented by participant in data listings.

#### 8. Pharmacokinetic (PK) Analyses

Phoenix® WinNonlin® software, Version 8.3.4 (or more recent version) will be used for all PK analyses. Statistical analyses will be performed using SAS for Windows software. Bioanalysis of all samples should be completed prior to the initiation of the PK and statistical analyses.

All PK concentration and PK parameter analyses will be conducted on the PK concentration population and PK parameter population, respectively.

PK concentrations, actual times, date/time of study drug administration and sample collection will be listed for the PK concentration population by nominal time for each study part, study day, participant and treatment, and summarized for the PC population for each study part by treatment and timepoint, using descriptive statistics (n, number of BLQs, arithmetic and geometric means, SD, geometric SD, CV%, geometric mean CV%, min, max, and median). Individual, mean (±SD) concentration, and overlay of individual plasma concentration versus time profile will be presented for both linear and semi-logarithmic scales for each study part by treatment for the PC population. For ease of presentation, actual and nominal sampling times will be used to present results for individual and mean figures, respectively.

PK parameters will be presented in data listings and summarized in tables for each study part by treatment (or day), using descriptive statistics (n, arithmetic mean, SD, %CV, geometric mean, geometric SD, geometric mean CV%, minimum, median, and maximum).

### 8.1 Data Handling

#### 8.1.1 PK Parameters Calculation Rules

For all PK analyses, concentration values BLQ that occur before the first measurable concentration of the study drug will be set to "0.00"; BLQ values that occur after first measurable concentration will be set to "missing". No imputations will be made on BLQ concentrations.

Invalid concentration values (due to bioanalytical or clinical issues) that occur prior to dosing will be replaced by "0.00". Invalid concentration values that occur after dosing will be set to "missing" for tabulation, graphical representation, and calculation purposes.

The actual clock time for dosing and the actual clock time for each PK sample collection will be recorded. For all sampling times, the actual sampling duration will be calculated as the difference between the sample collection actual clock time and the actual clock time of dosing. The actual post-dose sampling times, expressed in hours and rounded off to three decimal digits, will be used to calculate the PK parameters. Pre-dose sampling times will always be reported as zero (0.000), regardless of the time difference. Nominal sampling times will be used in concentration tables and mean graphs, while actual sampling times for post-dose samples will be used in the individual graphs. Actual sampling times for post-dose samples also will be used for PK parameter derivation, unless the actual sampling time is missing, in which case, the nominal time will be used.

#### 8.1.2 Data Presentation Rules

Non-measurable values reported in the plasma concentration data (i.e. values that are BLQ), will be entered as zero for the determination of summary statistics with the exception of geometric mean, geometric SD, and geometric CV%, where BLQ values will be imputed as half the lower limit of quantification (LLOQ) value. This also applies to any concentrations that are defined as PK parameters. Data recorded as "No Result" or "Not Reportable" (NR), "Not Calculated" (NC) or "No Sample" (NS) will be handled as missing (i.e. no assumption will be made about the actual concentration).

#### 8.2 Pharmacokinetic (PK) Parameters

The PK parameters shown in Table 8.2-1 below, will be calculated, whenever possible, by standard non-compartmental methods for camlipixant.

This document is confidential.


Controlled Document ID: 2805A.00, Effective Date 29-Jul-2019

Filing requirements: TMF 

Table 8.2-1: PK Parameters

| Parameter | Definition |
|---|---|
| AUC <sub>0-t</sub> | area under the concentration-time curve from time zero until the last observed |
| AUC <sub>0-t</sub> | concentration |
| AUC <sub>0-inf</sub> | area under the concentration-time curve from time zero to infinity (extrapolated) |
| Cl/F | apparent clearance, calculated as Dose/AUC <sub>0-inf</sub> |
| $C_{max}$ | maximal observed concentration |
| Kel | terminal elimination rate constant |
| Residual | percentage of AUC <sub>0-inf</sub> due to extrapolation from the time of the last observed |
| area | concentration to infinity, calculated as [1 - (AUC <sub>0-t</sub> /AUC <sub>0-inf</sub> )] x 100 |
| $T_{max}$ | time when the maximal concentration is observed |
| T <sub>½</sub> el | terminal elimination half-life, calculated as ln(2)/K <sub>el</sub> |
| V <sub>z</sub> /F | apparent volume of distribution, calculated as Dose/(Kel x AUC <sub>0-inf</sub> ) |

Additional PK parameters may be calculated as deemed necessary.

The following information will be presented for rifampin (Part 1): pre-dose concentrations on the morning of Days 4, 8, 9, 10, and 11. The following information will be presented for rabeprazole (Part 2): pre-dose concentrations on the morning of Days 4, 7, 8, 9, and 10. These data will be listed. Any additional PK data will be presented as appropriate.

Note: Area under the concentration-time curve (AUC) parameters will be calculated using the linear up log down trapezoidal method, where the linear trapezoidal rule is used any time the concentration data are increasing, and the logarithmic trapezoidal rule is used any time that the concentration data are decreasing.

Note:  $K_{el}$  will be the negative of the estimated slope of the linear regression of the ln-transformed plasma concentration versus time profile in the terminal elimination phase. The best fit method will be used to calculate the  $K_{el}$  from at least three concentration data points, excluding  $C_{max}$ .  $R^2$  adjusted, the goodness of fit statistic for the terminal elimination phase, adjusted for the number of points used in the estimation of  $K_{el}$  must be  $\geq 0.8$ . If the  $K_{el}$  cannot be measured (e.g.: there are fewer than three non-zero concentrations in the terminal elimination phase), the PK parameters derived from  $K_{el}$  will be presented in listing(s) but excluded from descriptive statistics in tables. All the derived parameters (i.e.,  $AUC_{0-inf}$ ,  $T_{\frac{1}{2}el}$ , Cl/F and  $V_d/F$ ) will be also flagged accordingly. The timepoint where ln-linear  $K_{el}$  calculation begins ( $K_{el}$   $L_{Ower}$ ), the actual sampling time of the last measurable concentration used to estimate the  $K_{el}$  ( $K_{el}$   $U_{Dpper}$ ), and the  $R^2$  adjusted for the ln-linear regression for the calculation of the elimination rate constant will be reported. If the Residual area is greater than 20%, the individual result should be flagged in the listing, and  $AUC_{0-inf}$ , Cl/F and  $V_d/F$ ) will be also flagged accordingly in the listing.

Some PK parameters may not be calculated for all or some participants, at the discretion of the Syneos pharmacokineticist if the concentration data is not deemed to be amenable to evaluation. Explanations for PK parameters that could not be estimated will be provided in the CSR.

This document is confidential.


Controlled Document ID: 2805A.00, Effective Date 29-Jul-2019

8.3 Assessment of Rifampin Effect (Part 1)



## 8.4 Assessment of Rabeprazole Effect (Part 2)



This document is confidential.


Controlled Document ID: 2805A.00, Effective Date 29-Jul-2019



#### 8.5 Attainment of Steady State

As supportive data, to assess attainment of steady state, descriptive statistics on pre-dose concentrations of rifampin in Part 1 (Days 9, 10, and 11) and rabeprazole in Part 2 (Days 8, 9, and 10) will be presented. If necessary, additional data may be presented.

#### 9. Pharmacogenomic Analyses

CCI

Other possible exploratory markers may be considered as deemed necessary. If applicable, a data listing will be provided for the pharmacogenomic population.

## 10. Safety

Safety and tolerability analysis will be performed for all subjects in the safety population. No inferential statistical analysis of safety data is planned.

#### 10.1 Exposure

Study drug administration will be listed by participant.

This document is confidential.


Controlled Document ID: 2805A.00, Effective Date 29-Jul-2019

## 10.2 Adverse Events (AEs)

AEs will be coded using MedDRA, Version 26.0 (or more recent version). Output data will include the MedDRA version used in the study. AEs will be grouped by SOC and PT and summarized by actual treatment phase. The summary tables will present the number and percentage of total participants and number of events by SOC and by PT.

All AE summaries will be restricted to treatment-emergent AEs (TEAEs), defined as AEs that commence on or after the time of first study drug administration. Any AE that first occurs pre-dose but worsens in severity after the first study drug administration will also be considered a TEAE. TEAEs will be attributed to the appropriate treatment phase as defined previously based on their onset date and time. TEAEs continuing after administration on the next treatment phase will be evaluated on a case-by-case basis (e.g., If there was no worsening in severity, it would be attributed to the treatment phase that coincides with the AE onset. If there was worsening in severity, it would be attributed to the treatment phase during which the worsening of the AE has occurred. The relationships could also be considered in this determination).

The relationships for each TEAE will be evaluated separately for the two drugs administered during the treatment phase of respective study part and will be classified according to the study protocol as definite, possible, probable, unlikely or not related to respective study drugs. The severity of TEAEs will be classified as mild, moderate or severe.

The number and percentage of subjects experiencing TEAEs and the number of TEAEs will be tabulated. Subjects who experience the same TEAE (in terms of MedDRA PT) more than once will only be counted once, however, the total number of events will be counted per category. This also applies to sub-categories (e.g., SOC, PT) displayed in the summaries.

The following summaries will be presented:

- Overall summary of TEAEs
- TEAEs by SOC and PT
- TEAEs by SOC, PT, and severity
- TEAEs by SOC, PT, and relationship to each study drug
- Serious AEs by SOC and PT
- AEMIs by SOC and PT

AEMIs for this study include the following, but not limited to:



All AEs will be listed. The following listings will be included: Non-TEAEs, TEAEs, serious AEs, AEMIs, CO.

This document is confidential.


Controlled Document ID: 2805A.00, Effective Date 29-Jul-2019

## 10.3 Laboratory Evaluations

Laboratory data, including biochemistry, hematology, coagulation, and urinalysis, will be listed by participant and summarized overall by study day. Observed values and changes from baseline will be presented.

In addition, a shift table representing the categorical change (low, normal, high) from baseline to each post baseline study day will be presented.

The categorical results of urinalysis will be summarized overall as number and percentage by study day.

Abnormal results will be flagged in the listings.

If more than one clinical laboratory is used, a formula that takes into consideration the relative normal ranges of each test of the laboratories will be utilized to normalize these data<sup>a</sup>. The conversion formula used for each test will depend on the typical distribution of the normal range for the test <sup>b</sup>. Prior to applying these formulas, units will be adjusted, as necessary. The laboratory which has the most results for each parameter will be considered primary in the formulas.

### 10.4 Vital Signs

Vital sign measurements will be listed by participant and summarized overall by study day. Observed values and changes from baseline will also be presented.

In addition, a shift table representing the categorical change (normal, abnormal not clinically significant, or abnormal clinically significant) from baseline to each post baseline study day will be presented.

Abnormal results will be flagged in the listings. The normal ranges as per clinical SOP (refer to the table below) will also be included in the listing and the summary tables.

| Vital Sign Parameters | Normal Ranges (inclusive) |
|--------------------------|---------------------------|
| Systolic blood pressure | 90 to 140 mmHg |
| Diastolic blood pressure | 50 to 90 mmHg |
| Hearth rate | 50 to 100 beats/min |
| Respiratory rate | 8 to 20 breaths/min |
| Oral temperature | 35.8 to 37.6 °C |

## 10.5 Electrocardiograms (ECGs)

ECG values will be listed by participant and summarized overall by study day. Observed values and changes from baseline will be presented.

In addition, a shift table representing the categorical change in overall interpretation (normal, abnormal not clinically significant, or abnormal clinically significant) from baseline to each post baseline study day will be presented.

Abnormal results will be flagged in the listings. The normal ranges as per clinical SOP (refer to the table below) will also be included in the listing and the summary tables.

This document is confidential.


Controlled Document ID: 2805A.00, Effective Date 29-Jul-2019

| ECG Parameters | Normal Ranges (inclusive) |
|----------------|---------------------------|
| Hearth rate | 50 to 100 beats/min |
| PR interval | 120 to 200 msec |
| QRS interval | 70 to 110 msec |
| QT interval | ≤ 450 msec |
| QTcF interval | ≤ 450 msec |

## 10.6 Physical Examination

The results of physical examinations will be listed by participant. Abnormal results will be flagged in the listings.

## 11. Changes from Analysis Planned in the Protocol

No changes were made to planned analyses.

## 12. Programming Considerations

All TFLs and statistical analyses will be generated using release 9.4 (or more recent version) (CCI ) software in accordance with Food and Drug Administration (FDA) guidelines. (CCI ) will be used for all PK analyses. This software was validated by Syneos in compliance with US 21 CFR Part 11 regulation.

#### 12.1 General Considerations

- One CCI program can create several outputs.
- Each output will be stored in a separate file.
- Output files will be delivered in rich text format that can be manipulated in MS Word.
- Numbering of TFLs will follow International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use (ICH) guideline E3°.

## 12.2 Table, Listing, and Figure Format

#### **12.2.1** General

- TFLs will be produced in landscape format. The orientation may be changed to portrait, as necessary to allow additional rows to be presented.
- TFLs will be produced using the Times New Roman font, size 9. The font size may be reduced as necessary to allow additional columns to be presented, but not at the expense of clarity.
- The data display for all TFLs will have a minimum blank 1-inch margin on all four sides.
- Unless otherwise specified, TFLs will be in black and white (no color).
- Specialized text styles, such as bolding, italics, borders, shading, and superscripted and subscripted text, will not be used in the TFLs, unless otherwise specified. On some occasions, superscripts 1, 2, or 3 may be used; see below.
- Standard keyboard characters will be used in the TFLs. Special characters, such as non-printable control characters, printer-specific, or font-specific characters, will not be used. Hexadecimal-derived characters will be used, where possible, if they are appropriate to help display math symbols (e.g.,  $\mu$ ). Certain subscripts and superscripts (e.g., cm<sup>2</sup>, C<sub>max</sub>) will be employed on a case-by-case basis.
- TFLs will be produced using sentence case, unless otherwise specified.

#### 12.2.2 Headers and Footers

- Times New Roman font, size 9 will be used for TFL headers and footers.
- All outputs will have the following at the top of each page: Bellus Health Protocol: 220254 (BUS-P1-11).
- All outputs will have page x of y at the top or bottom right corner of each page. TFLs are individually paginated in relation to total length (i.e., the page number appears sequentially as page x of y, where y is the total number of pages in the output).
- The data source will be included in the footer, as applicable.
- The date and time the output was generated will appear, along with the program name, at the bottom of each page.

## 12.2.3 Display Titles

Each display title includes the appropriate designation ("Table", "Figure", or "Listing") and a numeral, along with a descriptive name (e.g., Table 14.1-1 Subject Enrollment and Disposition). The analysis population should also be included in each title. ICH E3 numbering is strongly recommended, but Sponsor preferences are obtained for final determination. Display titles are left aligned, single spaced, and presented in title case. A solid line spanning the margins will separate display titles from column headings.

#### 12.2.4 Column and Row Headings

- Column and row headings are presented in title case, with the exception of complete sentences, which will be presented in sentence case.
- In efficacy or pharmacokinetic tables, the variable (or characteristic) column will be on the far left, followed by the group columns and overall column (if applicable). P-values may be presented under the overall column or in separate p-value column (if applicable). Within-treatment comparisons may have p-values presented in a row beneath the summary statistics for that treatment.
- Column and row headings will include "Unit" for numeric variables, as appropriate.
- Column and row headings will include the number of subjects in the analysis population for each group, presented as (N=xx). This is different from the 'n' used in descriptive statistics, which represents the number of observations.
- The order of treatments in the tables and listings will be placebo first, in placebo-controlled studies, and active comparators first, in active comparator trials, with "overall" (if applicable) last.

#### 12.2.5 Body of the Data Display

#### 12.2.5.1 General Conventions

Data in columns of a table or listing are formatted as follows:

• Alphanumeric values are left aligned.

This document is confidential.


Controlled Document ID: 2805A.00, Effective Date 29-Jul-2019

• Whole numbers (e.g., counts) or numerical data are centered aligned.

#### 12.2.5.2 Table Conventions

- Units will be included, where available.
- If the categories of a parameter are ordered, all categories between the maximum and minimum category are presented in the table, even if n=0 for all groups in a category between the minimum and maximum level for that parameter. See the example for the frequency distribution for symptom severity below. If percentages are presented in these tables, 0% will not be presented, therefore, counts of zero will be presented as "0", not "0 (0%)".

| Severity Rating | N |
|-----------------|---|
| Severe | 0 |
| Moderate | 8 |
| Mild | 3 |

- Where the categories are not ordered (e.g., Reason for Discontinuation), only those categories for which there is at least one subject represented will be included.
- An "Unknown" or "Missing" category will be added to each parameter for which information is unavailable for one or more subjects.
- P-values are presented in the format: 0.xxxx, where xxxx is the value. If the p-value is less than 0.0001, it will be presented as "<0.0001." If the p-value is >0.999, it will be presented as ">0.999."
- Percentage values are presented in parentheses with no spaces, one space after the count [e.g., 7 (12.8%), 13 (5.4%)]. Unless otherwise noted, for all percentages, the denominator will be the number of subjects in the analysis population for the group that has an observation. Percentages after zero counts are not displayed, and percentages equating to 100% are presented as "100%" (without decimal places).
- Unless otherwise noted, tabular displays of data for medical history, prior/concomitant medications, and AEs data are presented in alphabetical order.
- The percentage of subjects is typically calculated as a proportion of the number of subjects
  assessed in the relevant group (or overall) for the analysis population presented; however,
  careful consideration is required in many instances, due to the complicated nature of
  selecting the denominator. Details of this will be presented in footnotes or programming
  notes.
- In categorical summaries where a subject can be included in more than one category, a
  footnote or programming note will specify whether the subject is included in the summary
  statistics for all relevant categories or just one category and the criteria for selecting the
  category.

• Where a category with a subheading (such as SOC) must be split over more than one page, present the subheading followed by "(cont.)" at the top of each subsequent page. The overall summary statistics for the subheading will only be presented on the first relevant page.

## 12.2.5.3 Listing Conventions

- Unless otherwise noted, listings will be sorted for presentation in order of participant number, visit/collection day, visit/collection time, and parameter (alphabetic order).
- Dates are printed in DATE9.format (e.g., "ddMMMyyyy": 01JUL2000). Missing portions of dates are represented on subject listings as dashes (e.g.,--JUL2000). Dates that are missing because they are not applicable for the subject are presented as "N/A", unless otherwise specified.
- All observed time values are presented using a 24-hour clock HH:MM:SS or HH:MM format (e.g., 11:26:45, or 11:26). Time will only be reported if it was measured as part of the study.
- Units will be included, where available.

#### 12.2.5.4 Figure Conventions

- For safety figures, study visits will be displayed on the X-axis and endpoint (e.g., treatment mean change from baseline) values will be displayed on the Y-axis, unless otherwise specified.
- Legends will be used for all figures with more than one variable, group, or item displayed.
- Units will be included, where available.

#### 12.2.6 Footnotes

- A solid line spanning the margins will separate the body of the data display from the footnotes.
- All footnotes will be left aligned, with single spacing, immediately below the solid line beneath the data display.
- Informational footnotes begin with "Note:". Reference footnotes begin with a reference number or letter (e.g., 1, 2, 3 or a, b, c).
- Each new footnote starts on a new line, where possible.
- Subject-specific footnotes are avoided, where possible.
- Footnotes will be used sparingly and add value to the table, figure, or data listing. If more than six lines of footnotes are planned, a cover page may be used to display footnotes, and only those essential to comprehension of the data will be repeated on each page.

## 13. Quality Control

programs are developed to produce outputs such as analysis data sets, summary tables, data listings, figures, and statistical analyses. These are developed and undergo quality control in accordance with the latest versions of SOP 2800<sup>d</sup> and SOP 2801<sup>e</sup>.

#### 14. Reference List

<sup>a</sup>Chuang-Stein, C., PhD, Research Support Biostatistics Unit, 9164–32–2, The Upjohn Company, Kalamazoo, Michigan. (1992). Summarizing Laboratory Data with Different Reference Ranges in Multi-Center Clinical Trials. Drug Information Journal, 26(1), 77-84. doi:10.1177/009286159202600108

<sup>b</sup>Karvanen, J., Signal Processing Laboratory, Helsinki University of Technology, Helsinki, Finland. (2003). The Statistical Basis of Laboratory Data Normalization. Drug Information Journal, 37(1), 101-107. doi:10.1177/009286150303700112

<sup>c</sup>International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use (ICH). (1996). Guideline for Industry, Structure and Content of Clinical Study Reports (ICH E3).

End of document

This document is confidential.


Controlled Document ID: 2805A.00, Effective Date 29-Jul-2019

Statistical Analysis Plan (Table/Figure/Listing Shells) Version 1.0 dated 26-OCT-2023



## Statistical Analysis Plan (Table/ Figure/Listing Shells)

**Sponsor Name:** Bellus Health

Protocol Number: 220254 (BUS-P1-11)

**Protocol Title:** A Phase 1, 2-Part, Open-label, Fixed-sequence Study Evaluating the Effect of Rifampin (Part 1) and Rabeprazole (Part 2) on the Pharmacokinetics of a Single Dose of Camlipixant (BLU-5937) 50 mg Tablet in Healthy Participants under Fasting Conditions

**Protocol Version and Date:** Final, 03-Apr-2023

**Sponsor Study Number:** BUS-P1-11

Authors: PPD , Sr. Principal Biostatistician , Technical Writer

#### **Notice of Confidential and Proprietary Information:**

The information contained in this document is confidential belonging to Bellus Health. Acceptance of this document constitutes agreement by the recipient that no information contained herein will be published or disclosed without prior written authorization from an official of Bellus Health. However, this document may be disclosed to the appropriate Institutional Review Board and ethics committees or duly authorized representatives of a national regulatory authority under the condition that they are requested to keep it confidential. In the event of an actual or suspected breach of this obligation, Syneos Health should be notified promptly.

26-Oct-2023 (Final 1.0) 

Statistical Analysis Plan (Table/Figure/Listing Shells)

Bellus Health Protocol 220254 (BUS-P1-11)

## **Revision History**

| Version | Date<br>(DD-Mmm-YYYY) | <b>Document Owner</b> | Revision Summary |
|-----------|-----------------------|-----------------------|------------------|
| Final 1.0 | 26-Oct-2023 | PPD | Final version |



## Approvals

I confirm that I have reviewed this document and agree with the content.

| Syneos Health Approval | | |
|----------------------------------|---------------|------------------|
| PPD | | |
| PPD , | | 30-Oct-2023 |
| Sr. Principal Biostatistician | _ | |
| Name, Title | Signature | Date |
| Lead Biostatistician | PPD | (DD-Mmm-YYYY) |
| PPD Manager Statistical | | 21 0 - 1 2022 |
| Programming | | 31-Oct-2023 |
| Name, Title | Signature | Date |
| Lead Statistical Programmer | PPD | (DD-Mmm-YYYY) |
| PPD , Sr. Biostatistician | | 31-Oct-2023 |
| Name, Title | Signature | Date |
| Senior Reviewing Biostatistician | 218111111 | (DD-Mmm-YYYY) |
| PPD PPD | | |
| PPD | | |
| Senior Pharmacokineticist | | 30-Oct-2023 |
| Name, Title | Signature | Date |
| Lead Pharmacokineticist | Signature | (DD-Mmm-YYYY) |
| Lead I Harmacokineticist | PPD | (DD Millin 1111) |
| Modical Weiter H | | 02-Nov-2023 |
| , Medical Writer II | - G: | D / |
| Name, Title | Signature | Date |
| Lead Medical Writer | (DD-Mmm-YYYY) | |


## **Table of Contents**

| 1. Tables | 9 |
|---|---|
| Table 14.1-1.1 Subject Enrollment and Disposition - Part 1 | 10 |
| Table 14.1-1.2 Subject Enrollment and Disposition - Part 2 | 12 |
| Table 14.1-1.3 Analysis Populations - Part 1 | |
| Table 14.1-1.4 Analysis Populations - Part 2 | |
| Table 14.1-2.1 Demographics and Baseline Body Measurements (Safety Population) - Part 1 | 16 |
| Table 14.1-2.2 Demographics and Baseline Body Measurements (Safety Population) - Part 2 | 19 |
| Table 14.2-1.1 Plasma Concentrations (ng/mL) of Camlipixant (PK Concentration Population) - Part 1 | |
| Table 14.2-1.2 Plasma Concentrations (ng/mL) of Camlipixant (PK Concentration Population) - Part 2 | |
| Table 14.2-2.1 Plasma PK Parameters of Camlipixant (PK Parameter Population) - Part 1 | |
| Table 14.2-2.2 Plasma PK Parameters of Camlipixant (PK Parameter Population) - Part 2 | |
| Table 14.2-3 Assessment of Rifampin Effect: DDI (PK Parameter Population) - Part 1 | |
| Table 14.2-4 Assessment of Rabeprazole Effect: DDI (PK Parameter Population) - Part 2 | 31 |
| Table 14.2-5 Non-Parametric Assessment of Rifampin Effect (PK Parameter Population) - Part 1 | |
| Table 14.2-6 Non-Parametric Assessment of Rabeprazole Effect (PK Parameter Population) - Part 2 | |
| Table 14.2-7.1 Attainment of Steady State (ng/mL) (PK Concentration Population) - Part 1 | |
| Table 14.2-7.2 Attainment of Steady State (ng/mL) (PK Concentration Population) - Part 2 | |
| Table 14.3.1-1.1 Overall Summary of TEAEs (Safety Population) - Part 1 | |
| Table 14.3.1-1.2 Overall Summary of TEAEs (Safety Population) - Part 2 | |
| Table 14.3.1-2.1 TEAEs by SOC and PT (Safety Population) - Part 1 | |
| Table 14.3.1-2.2 TEAEs by SOC and PT (Safety Population) - Part 2 | |
| Table 14.3.1-3.1 TEAEs by Severity (Safety Population) - Part 1 | |
| Table 14.3.1-3.2 TEAEs by Severity (Safety Population) - Part 2 | 42 |
| Table 14.3.1-4.1 TEAEs by Relationship to Study Drug (Camlipixant) (Safety Population) - Part 1 | 44 |
| Table 14.3.1-4.2 TEAEs by Relationship to Study Drug (Rifampin) (Safety Population) – Part 1 | 46 |
| Table 14.3.1-4.3 TEAEs by Relationship to Study Drug (Camlipixant) (Safety Population) - Part 2 | |
| Table 14.3.1-4.4 TEAEs by Relationship to Study Drug (Rabeprazole) (Safety Population) - Part 2 | |
| Table 14.3.1-5.1 Serious TEAEs (Safety Population) - Part 1 | |
| Table 14.3.1-5.2 Serious TEAEs (Safety Population) – Part 2 | |
| Table 14.3.1-6.1 Treatment-emergent AEMIs (Safety Population) - Part 1 | |
| Table 14.3.1-6.2 Treatment-emergent AEMIs (Safety Population) - Part 2 | |
| Table 14.3.4-1.1 Biochemistry (Safety Population) - Part 1 | |
| Table 14.3.4-1.2 Biochemistry (Safety Population) - Part 2 | |
| Table 14.3.4-2.1 Biochemistry Shifts from Baseline (Safety Population) - Part 1 | |
| Table 14.3.4-2.2 Biochemistry Shifts from Baseline (Safety Population) - Part 2 | |
| Table 14.3.4-3.1 Hematology (Safety Population) - Part 1 | |
| Table 14.3.4-3.2 Hematology (Safety Population) - Part 2 | |
| Table 14.3.4-4.1 Hematology Shifts from Baseline (Safety Population) - Part 1 | |
| Table 14.3.4-4.2 Hematology Shifts from Baseline (Safety Population) - Part 2 | |
| Table 14.3.4-5.1 Coagulation (Safety Population) - Part 1 | |
| Table 14.3.4-5.2 Coagulation (Safety Population) - Part 2 | |
| Table 14.3.4-6.1 Coagulation Shifts from Baseline (Safety Population) - Part 1 | |
| Table 14.3.4-6.2 Coagulation Shifts from Baseline (Safety Population) - Part 2 | |
| Table 14.3.4-7.1 Urinalysis: Quantitative (Safety Population) - Part 1 | |
| Table 14.3.4-7.2 Urinalysis: Quantitative (Safety Population) - Part 2 | |
| Table 14.3.4-8.1 Urinalysis: Quantitative Shifts from Baseline (Safety Population) - Part 1 | |
| Table 14.3.4-8.2 Urinalysis: Quantitative Shifts from Baseline (Safety Population) - Part 2 | |
| Table 14.3.4-9.1 Urinalysis: Categorical (Safety Population) - Part 1 | |
| Table 14.3.4-9.2 Urinalysis: Categorical (Safety Population) - Part 2 | |
| Table 14.3.4-10.1 Vital Signs (Safety Population) - Part 1 | |
| Table 14.3.4-10.2 Vital Signs (Safety Population) - Part 2 | |
| Table 14.3.4-11.1 Vital Signs Shifts from Baseline (Safety Population) - Part 1 | |
| $oldsymbol{arphi}$ | |

| Table 14.3.4-11.2 Vi | tal Signs Shifts from Baseline (Safety Population) - Part 2 | 77 |
|---|---|---|
| Table 14.3.4-12.1 EC | CGs: Quantitative (Safety Population) - Part 1 | 78 |
| | CGs: Quantitative (Safety Population) - Part 2 | |
| | CGs: Interpretation Shifts from Baseline (Safety Population) - Part 1 | |
| | CGs: Interpretation Shifts from Baseline (Safety Population) - Part 2 | |
| 2. Figures | | 82 |
| | ividual Plasma Concentrations of Camlipixant - Linear Scale (PK Concentration Population | |
| | ividual Plasma Concentrations of Camlipixant – Linear Scale (PK Concentration Populati | |
| | ividual Plasma Concentrations of Camlipixant - Semi-Log Scale (PK Concentration Popu | |
| | ''' IN O AA' CO I'' A G 'I G I MYO AA' | 85 |
| | ividual Plasma Concentrations of Camlipixant – Semi-Log Scale (PK Concentration | 96 |
| | an (±SD) Plasma Concentrations of Camlipixant - Linear Scale (PK Concentration Popula | |
| | an (±SD) Frasma Concentrations of Caminpixant - Linear Scale (FK Concentration Popula | |
| | an (±SD) Plasma Concentrations of Camlipixant - Linear Scale (PK Concentration Popula | |
| | an (±5D) Hasina Concentrations of Caminpixant - Emear Searc (FR Concentration Fopula | |
| | an (±SD) Plasma Concentrations of Camlipixant - Semi-Log Scale (PK Concentration | |
| Population) - Part 1 | (-22) T. M. M. C. | 89 |
| | an (±SD) Plasma Concentrations of Camlipixant - Semi-Log Scale (PK Concentration | |
| | 1 5 | 90 |
| | erlay of Individual Plasma Concentrations of Camlipixant - Linear Scale (PK Concentration | |
| | * | |
| Figure 14.2-18.2 Ove | erlay of Individual Plasma Concentrations of Camlipixant – Linear Scale (PK Concentrati | ion |
| | erlay of Individual Plasma Concentrations of Camlipixant - Semi-Log Scale (PK Concent | |
| Population) - Part 1 | | 93 |
| | erlay of Individual Plasma Concentrations of Camlipixant – Semi-Log Scale (PK Concent | |
| | LO 4 4 A CD'C ' ECC 4 DDU ANOVA (DV D 4 D 14' ) ] | |
| | Output: Assessment of Rifampin Effect: DDI by ANOVA (PK Parameter Population) - | |
| | Output: Assessment of Rabeprazole Effect: DDI by ANOVA (PK Parameter Population) | |
| | Output. Assessment of Kaoeprazole Effect. DDI by ANOVA (FK Farameter Fopulation) | |
| | Output: Non-Parametric Assessment of Rifampin Effect (PK Parameter Population) - Pa | |
| CCI<br>CCI | Output: Non-Parametric Assessment of Rabeprazole Effect (PK Parameter Population) - | |
| | output 1 on 1 manager 1 aparticular of 1 mospitalists Entrol (1 111 manager 1 open mion) | |
| Listing 16.2.1.1-1 Su | bject Enrollment (Safety Population) - Part 1 | |
| | bject Enrollment (Safety Population) - Part 2 | |
| | bject Disposition (Safety Population) - Part 1 | |
| | bject Disposition (Safety Population) - Part 2 | |
| Listing 16.2.2.1-1 Pro | otocol Deviations (Safety Population) - Part 1 | 104 |
| Listing 16.2.2.1-2 Pro | otocol Deviations (Safety Population) - Part 2 | 105 |
| | clusion and Exclusion Criteria (Safety Population) - Part 1 | |
| | clusion and Exclusion Criteria (Safety Population) - Part 2 | |
| | ssignment to Analysis Populations - Part 1 | |
| | ssignment to Analysis Populations - Part 2 | |
| | emographics (Safety Population) - Part 1 | |
| | emographics (Safety Population) - Part 2 | |
| | ody Measurements (Safety Population) - Part 1 | |
| | ody Measurements (Safety Population) - Part 2 | 113 |
| I ISTING IN / A 3-1 N/L | edical History (Natery Pobliation) - Part I | 114 |



| Listing | 16.2.4.3-2 Medical History (Safety Population) - Part 2 | 15 |
|---------|--------------------------------------------------------------|----|
| | 10121 HD 2 1/1001001 1115001 (Suret) 1 op utwich) 1 of the 2 | |

| Listing 16.2.4.5-1 Prior and Concomitant Medications (Safety Population) - Part 1 | |
|---|---|
| Listing 16.2.4.5-2 Prior and Concomitant Medications (Safety Population) - Part 2 | |
| Listing 16.2.4.6-1 Urine Drug Screen (Safety Population) - Part 1 | |
| Listing 16.2.4.6-2 Urine Drug Screen (Safety Population) - Part 2 | |
| Listing 16.2.4.7-1 Alcohol Breath Test (Safety Population) - Part 1 | |
| Listing 16.2.4.7-2 Alcohol Breath Test (Safety Population) - Part 2 | |
| Listing 16.2.4.8-1 Urine Cotinine Test (Safety Population) - Part 1 | |
| Listing 16.2.4.8-2 Urine Cotinine Test (Safety Population) - Part 2 | |
| Listing 16.2.4.9-1 Pregnancy Test (Safety Population) - Part 1 | |
| Listing 16.2.4.9-2 Pregnancy Test (Safety Population) - Part 2 | |
| Listing 16.2.4.10-1 Follicle Stimulating Hormone Test (Safety Population) - Part 1 | |
| Listing 16.2.4.10-2 Follicle Stimulating Hormone Test (Safety Population) - Part 2 | |
| Listing 16.2.4.11-1 Serology (Safety Population) - Part 1 | |
| Listing 16.2.4.11-2 Serology (Safety Population) - Part 2 | |
| Listing 16.2.4.12-1 COVID-19 Test (Safety Population) - Part 1 | |
| Listing 16.2.4.12-2 COVID-19 Test (Safety Population) - Part 2 | |
| Listing 16.2.5.1-1 Study Drug Administration (Safety Population) - Part 1 | |
| Listing 16.2.5.1-2 Study Drug Administration (Safety Population) - Part 2 | |
| Listing 16.2.6.1-1 Plasma PK Concentrations (PK Concentration Population) - Part 1 | 136 |
| Listing 16.2.6.1-2 Plasma PK Concentrations (PK Concentration Population) - Part 2 | 137 |
| Listing 16.2.6.2-1 Plasma PK Parameters of (PK Parameter Population) - Part 1 | 138 |
| Listing 16.2.6.2-2 Plasma PK Parameters of (PK Parameter Population) - Part 2 | 139 |
| Listing 16.2.7.1-1 Non-TEAEs (Safety Population) - Part 1 | 140 |
| Listing 16.2.7.1-2 Non-TEAEs (Safety Population) - Part 2 | 141 |
| Listing 16.2.7.2-1 TEAEs (Safety Population) - Part 1 | 142 |
| Listing 16.2.7.2-2 TEAEs (Safety Population) - Part 2 | 143 |
| Listing 16.2.7.3-1 Serious AEs (Safety Population) - Part 1 | 144 |
| Listing 16.2.7.3-2 Serious AEs (Safety Population) - Part 2 | 145 |
| Listing 16.2.7.4-1 AEMIs (Safety Population) - Part 1 | 146 |
| Listing 16.2.7.4-2 AEMIs (Safety Population) - Part 2 | 147 |
| Listing 16.2.7.5-1 CCI | 148 |
| Listing 16.2.7.5-2 gej | |
| Listing 16.2.7.6-1 Oral Hypoesthesia, Oral Paresthesia AE Questionnaire (Safety Population) - Part 1 | 150 |
| Listing 16.2.7.6-2 Oral Hypoesthesia, Oral Paresthesia AE Questionnaire (Safety Population) - Part 2 | 151 |
| Listing 16.2.8.1-1 Biochemistry (Safety Population) - Part 1 | 152 |
| Listing 16.2.8.1-2 Biochemistry (Safety Population) - Part 2 | |
| Listing 16.2.8.2-1 Hematology (Safety Population) - Part 1 | |
| Listing 16.2.8.2-2 Hematology (Safety Population) - Part 2 | |
| Listing 16.2.8.3-1 Coagulation (Safety Population) - Part 1 | |
| Listing 16.2.8.3-2 Coagulation (Safety Population) - Part 2 | 157 |
| Listing 16.2.8.4-1 Urinalysis: Quantitative (Safety Population) - Part 1 | |
| Listing 16.2.8.4-2 Urinalysis: Quantitative (Safety Population) - Part 2 | |
| Listing 16.2.8.5-1 Urinalysis: Categorical (Safety Population) - Part 1 | |
| Listing 16.2.8.5-2 Urinalysis: Categorical (Safety Population) - Part 2 | |
| Listing 16.2.8.6-1 Vital Signs (Safety Population) - Part 1 | |
| Listing 16.2.8.6-2 Vital Signs (Safety Population) - Part 2 | |
| Listing 16.2.8.7-1 ECGs (Safety Population) - Part 1 | |
| Listing 16.2.8.7-2 ECGs (Safety Population) - Part 2 | |



| Listing 16.2.8.8-1 Physical Examination (Safety Population) - Part 1 | 166 |
|---|---|
| Listing 16.2.8.8-2 Physical Examination (Safety Population) - Part 2 | |
| Listing 16.2.8.8-3 Pharmacogenomic Measurements (Pharmacogenomic Population) - Part 1 | 168 |
| Listing 16.2.8.8-4 Pharmacogenomic Measurements (Pharmacogenomic Population) - Part 2 | 169 |

Bellus Health Protocol 220254 (BUS-P1-11)

# 1. Tables

Bellus Health Protocol 220254 (BUS-P1-11)

Table 14.1-1.1 Subject Enrollment and Disposition - Part 1

| Catagamy | Camlipixant | Rifampin | Camlipixant + Rifampin | Overall |
|---|---|---|---|---|
| Category | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| G 1 | | | | |
| Screened, n | - | - | - | XX |
| Screening Failures <sup>[a][b]</sup> , n (%) | - | - | - | xx (xx.x) |
| Not Enrolled <sup>[a][c]</sup> , n (%) | - | - | - | xx (xx.x) |
| Enrolled <sup>[a][d]</sup> , n (%) | - | - | - | xx (xx.x) |
| Dosed [e], n | XX | XX | XX | XX |
| Not Dosed, n | XX | XX | XX | - |
| Completed [f][g], n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Did Not Complete [g], n (%) | xx(xx.x) | xx (xx.x) | xx(xx.x) | xx (xx.x) |
| Reason For Non-completion <sup>[h]</sup> , n (%): | | | | |
| Adverse Event | xx (xx.x) | xx (xx.x) | xx (xx.x) | _ |
| Death | xx (xx.x) | xx (xx.x) | xx (xx.x) | - |
| Lost To Follow-up | xx (xx.x) | xx (xx.x) | xx (xx.x) | - |
| Non-Compliance With Study Drug | xx (xx.x) | xx (xx.x) | xx (xx.x) | - |
| Physician Decision | xx (xx.x) | xx (xx.x) | xx (xx.x) | - |
| Pregnancy | xx (xx.x) | xx (xx.x) | xx (xx.x) | - |
| Protocol Deviation | xx (xx.x) | xx (xx.x) | xx (xx.x) | - |
| Site Terminated By Sponsor | xx (xx.x) | xx (xx.x) | xx (xx.x) | - |
| Study Terminated By Sponsor | xx (xx.x) | xx (xx.x) | xx (xx.x) | - |
| Technical Problems | xx (xx.x) | xx (xx.x) | xx (xx.x) | - |
| Withdrawal by Participant | xx (xx.x) | xx (xx.x) | xx (xx.x) | - |
| Withdrawal of Consent | xx (xx.x) | xx (xx.x) | xx (xx.x) | - |
| Other | xx (xx.x) | xx (xx.x) | xx (xx.x) | - |

Abbreviations: N=Number of participants in the population; n=Number of participants; n (%)= number and percent of participants

<sup>[</sup>a] Percentage is based on the number of screened volunteers.

<sup>[</sup>b] Screening failures include volunteers who did not meet study criteria.

Not enrolled include volunteers who were judged eligible but decided not to participate on study or who were not selected to participate in the study since there was already a sufficient number of volunteers.

<sup>[</sup>d] Enrolled includes volunteers who were judged eligible and accepted to participate in the trial after having signed the approved final version of the study informed consent form and those identified as standby who may replace participants who withdraw from the study before dosing.

<sup>[</sup>e] Includes all participants who received at least one dose of the study drug.

CCI

Statistical Analysis Plan (Table/Figure/Listing Shells)

Bellus Health Protocol 220254 (BUS-P1-11)

Note: The overall column includes participants from all treatment groups.

Treatment sequence: camlipixant 50 mg SD on Day 1, rifampin cor mg ground from Day 4 to Day 10, rifampin cor mg ground from Day 11 to 12 with co-administration of camlipixant 50 mg SD on Day 11.

Data Sources: Listing 16.2.1.1-1, Listing 16.2.1.2-1, Listing 16.2.3.1-1, and Listing 16.2.5.1-1.

<sup>[</sup>f] Number of participants who completed the respective treatment phase.

<sup>[</sup>g] Percentage is based on the number of dosed participants.

<sup>[</sup>h] Percentage is based on the number of participants that did not complete the study.

Bellus Health Protocol 220254 (BUS-P1-11)

Table 14.1-1.2 Subject Enrollment and Disposition - Part 2

| Catagory | Camlipixant | Rabeprazole | Camlipixant + Rabeprazole | Overall |
|---|---|---|---|---|
| Category | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Screened, n | - | - | - | XX |
| Screening Failures <sup>[a][b]</sup> , n (%) | - | - | - | xx(xx.x) |
| Not Enrolled <sup>[a][c]</sup> , n (%) | - | - | - | xx(xx.x) |
| Enrolled <sup>[a][d]</sup> , n (%) | - | - | - | xx (xx.x) |
| Dosed [e], n | XX | XX | XX | xx |
| Not Dosed, n | XX | XX | XX | - |
| Completed [f][g], n (%) | XX | XX | XX | xx (xx.x) |
| Did Not Complete [g], n (%) | XX | XX | XX | xx (xx.x) |
| Reason For Non-completion <sup>[h]</sup> , n (%): | | | | |
| Adverse Event | xx (xx.x) | xx (xx.x) | xx (xx.x) | - |
| Death | xx (xx.x) | xx (xx.x) | xx (xx.x) | - |
| Lost To Follow-up | xx (xx.x) | xx (xx.x) | xx (xx.x) | - |
| Non-Compliance With Study Drug | xx (xx.x) | xx (xx.x) | xx (xx.x) | - |
| Physician Decision | xx (xx.x) | xx (xx.x) | xx (xx.x) | - |
| Pregnancy | xx (xx.x) | xx (xx.x) | xx (xx.x) | - |
| Protocol Deviation | xx (xx.x) | xx (xx.x) | xx (xx.x) | - |
| Site Terminated By Sponsor | xx (xx.x) | xx (xx.x) | xx (xx.x) | - |
| Study Terminated By Sponsor | xx (xx.x) | xx (xx.x) | xx (xx.x) | - |
| Technical Problems | xx (xx.x) | xx (xx.x) | xx (xx.x) | - |
| Withdrawal by Participant | xx (xx.x) | xx (xx.x) | xx (xx.x) | - |
| Withdrawal of Consent | xx (xx.x) | xx (xx.x) | xx (xx.x) | - |
| Other | xx (xx.x) | xx (xx.x) | xx (xx.x) | - |

Abbreviations: N=Number of participants in the population; n=Number of participants; n (%)= number and percent of participants

<sup>[</sup>a] Percentage is based on the number of screened volunteers.

<sup>[</sup>b] Screening failures include volunteers who did not meet study criteria.

Not enrolled include volunteers who were judged eligible but decided not to participate on study or who were not selected to participate in the study since there was already a sufficient number of volunteers.

<sup>[</sup>d] Enrolled includes volunteers who were judged eligible and accepted to participate in the trial after having signed the approved final version of the study informed consent form and those identified as standby who may replace participants who withdraw from the study before dosing.

<sup>[</sup>e] Includes all participants who received at least one dose of the study drug.



Bellus Health Protocol 220254 (BUS-P1-11)

Note: The overall column includes participants from all treatment groups.

Treatment sequence: camlipixant 50 mg SD on Day 1, rabeprazole remg rem from Day 4 to Day 9, rabeprazole remg rem from Day 10 to 11 with coadministration of camlipixant 50 mg SD on Day 10.

Data Sources: Listing 16.2.1.1-2, Listing 16.2.1.2-2, Listing 16.2.3.1-2, and Listing 16.2.5.1-2.

<sup>[</sup>f] Number of participants who completed the respective treatment phase.

<sup>[</sup>g] Percentage is based on the number of dosed participants.

<sup>[</sup>h] Percentage is based on the number of participants that did not complete the study.



Bellus Health Protocol 220254 (BUS-P1-11)

**Table 14.1-1.3 Analysis Populations - Part 1** 

| Analysis Population | Overall<br>(N=xx) |
|------------------------------------|-------------------|
| Safety Population, n (%) | xx (xx.x) |
| PK Concentration Population, n (%) | xx (xx.x) |
| PK Parameter Population, n (%) | xx (xx.x) |
| Pharmacogenomic Population, n (%) | xx (xx.x) |

Abbreviations: N=Number of participants dosed; n=Number of participants; n (%)= number and percent of participants



Bellus Health Protocol 220254 (BUS-P1-11)

**Table 14.1-1.4 Analysis Populations - Part 2** 

| Analysis Population | Overall<br>(N=xx) |
|---|---|
| Safety Population, n (%) PK Concentration Population, n (%) PK Parameter Population, n (%) Pharmacogenomic Population, n (%) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) |

Abbreviations: N=Number of participants dosed; n=Number of participants; n (%)= number and percent of participants



Table 14.1-2.1 Demographics and Baseline Body Measurements (Safety Population) - Part 1

| Category | Camlipixant | Rifampin | Camlipixant + Rifampin | Overall |
|---|---|---|---|---|
| Category | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Age (years) | | | | |
| n | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | xx.x |
| SD | XX.XX | XX.XX | XX.XX | xx.xx |
| Min | XX | XX | XX | XX |
| Median | XX.X | XX.X | XX.X | XX.X |
| Max | XX | XX | XX | XX |
| Sex n (%) | | | | |
| Male | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Female | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Childbearing Potential <sup>[a]</sup> , n (%) | | | | |
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | xx(xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Reason for Non-Childbearing Potential <sup>[b]</sup> , n (%) | | | | |
| Pre-Menopause | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Menopause | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Post-Menopause | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Surgically Sterile | xx(xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Ethnicity, n (%) | | | | |
| Hispanic or Latino | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Not Hispanic or Latino | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Not Reported | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Unknown | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |



Bellus Health Protocol 220254 (BUS-P1-11)

| Category | Camlipixant | Rifampin | Camlipixant + Rifampin | Overall |
|---|---|---|---|---|
| Category | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| (cont.) | | | | |
| Race, n (%) | | | | |
| Am Indian | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Asian | xx (xx.x) | xx (xx.x) | XX (XX.X) | xx (xx.x) |
| Black | xx (xx.x) | xx (xx.x) | xx (xx.x) | XX (XX.X) |
| Hawaiian | xx (xx.x) | xx (xx.x) | XX (XX.X) | xx (xx.x) |
| White | | | | xx (xx.x)<br>xx (xx.x) |
| | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| Not Reported | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Unknown | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Multiple | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Height (cm) | | | | |
| n | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX |
| Min | XX | XX | XX | XX |
| Median | XX.X | XX.X | XX.X | XX.X |
| Max | XX | XX | XX | XX |
| Weight (kg) | | | | |
| n | XX | XX | XX | XX |
| Mean | XX.XX | XX.XX | XX.XX | XX.XX |
| SD | XX.XXX | XX.XXX | XX.XXX | XX.XXX |
| Min | XX.X | XX.X | XX.X | XX.X |
| Median | XX.XX | XX.XX | XX.XX | XX.XX |
| Max | xx.x | XX.X | XX.X | XX.X |
| BMI (kg/m²) | | | | |
| n | XX | XX | XX | XX |
| Mean | XX.XX | XX.XX | XX.XX | XX.XX |
| SD | XX.XXX | XX.XXX | XX.XXX | XX.XXX |
| Min | XX.X | XX.X | XX.X | XX.X |
| Median | XX.X<br>XX.XX | XX.XX | XX.XX | XX.XX<br>XX.XX |
| Max | XX.XX<br>XX.X | | | |
| IVIAA | АА.А | XX.X | XX.X | XX.X |



Bellus Health Protocol 220254 (BUS-P1-11)

Abbreviations: Am Indian= American Indian or Alaskan native; Black= Black or African American; BMI= body mass index; Hawaiian= native Hawaiian or other pacific islander; N=Number of participants in the population; n (%)=Number and percent of participants; n= number of observations; max= maximum; min= minimum; SD= standard deviation

Note: The last result (scheduled or unscheduled) obtained prior to the first study drug administration was used to generate this table.

Treatment sequence: camlipixant 50 mg SD on Day 1, rifampin regimg from Day 4 to Day 10, rifampin regimg from Day 11 to 12 with coadministration of camlipixant 50 mg SD on Day 11.

Data Source: Listing 16.2.4.1-1 and Listing 16.2.4.2-1

Note: if N is different for safety and PC / PK populations, please include a Demographics and Baseline Body measurements table for PC / PK populations.

<sup>[</sup>a] Percentage is based on the number of females.

<sup>[</sup>b] Percentage is based on the number of females of non-childbearing potential.

Table 14.1-2.2 Demographics and Baseline Body Measurements (Safety Population) - Part 2

| Category | Camlipixant (N=xx) | Rabeprazole (N=xx) | Camlipixant + Rabeprazole (N=xx) | Overall (N=xx) |
|---|---|---|---|---|
| | | , | , | , |
| Age (years) | | | | |
| n | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX |
| Min | XX | XX | XX | XX |
| Median | XX.X | XX.X | XX.X | XX.X |
| Max | XX | XX | XX | XX |
| Sex, n (%) | | | | |
| Male | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Female | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Childbearing Potential <sup>[a]</sup> , n (%) | | | | |
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Reason for Non-Childbearing Potential <sup>[b]</sup> , n (%) | | | | |
| Pre-Menopause | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Menopause | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Post-Menopause | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Surgically Sterile | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Ethnicity, n (%) | | | | |
| Hispanic or Latino | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Not Hispanic or Latino | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Not Reported | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Unknown | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |



| Category | Camlipixant | Rabeprazole | Camlipixant + Rabeprazole | Overall |
|---|---|---|---|---|
| Category | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| (cont.) | | | | |
| Race, n (%) | | | | |
| Am Indian | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Asian | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Black | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Hawaiian | xx (xx.x) | xx (xx.x) | XX (XX.X) | xx (xx.x) |
| White | xx (xx.x) | xx (xx.x) | XX (XX.X) | xx (xx.x) |
| Not Reported | ` ′ | | * * | ` ' |
| Unknown | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Multiple | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Height (cm) | | | | |
| n | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX |
| Min | XX | XX | XX | XX |
| Median | XX.X | XX.X | XX.X | XX.X |
| Max | XX | XX | xx | XX |
| Weight (kg) | | | | |
| n (kg) | XX | XX | XX | XX |
| Mean | XX.XX | XX.XX | XX.XX | XX.XX |
| SD | XX.XXX | XX.XXX | XX.XXX | XX.XXX |
| Min | XX.X | XX.X | XX.X | XX.X |
| Median | XX.XX | | XX.XX | XX.XX |
| Max | | XX.XX | | |
| Max | XX.X | XX.X | XX.X | XX.X |
| BMI $(kg/m^2)$ | | | | |
| n | XX | XX | XX | XX |
| Mean | XX.XX | XX.XX | XX.XX | XX.XX |
| SD | XX.XXX | XX.XXX | XX.XXX | XX.XXX |
| Min | XX.X | XX.X | XX.X | XX.X |
| Median | XX.XX | XX.XX | XX.XX | XX.XX |
| Max | XX.X | XX.X | XX.X | XX.X |



Bellus Health Protocol 220254 (BUS-P1-11)

Abbreviations: Am Indian= American Indian or Alaskan native; Black= Black or African American; BMI= body mass index; Hawaiian= native Hawaiian or other pacific islander; N=Number of participants in the population; n (%)=Number and percent of participants; n= number of observations; max= maximum; min= minimum; SD= standard deviation

Note: The last result (scheduled or unscheduled) obtained prior to the first study drug administration was used to generate this table.

Treatment sequence: camlipixant 50 mg SD on Day 1, rabeprazolege mg get from Day 4 to Day 9, rabeprazole en mg get from Day 10 to 11 with co-administration of camlipixant 50 mg SD on Day 10.

Data Source: Listing 16.2.4.1-2 and Listing 16.2.4.2-2

Note: if N is different for safety and PC / PK populations, please include a Demographics and Baseline Body measurements table for PC / PK populations.

<sup>[</sup>c] Percentage is based on the number of females.

<sup>[</sup>d] Percentage is based on the number of females of non-childbearing potential.



Bellus Health Protocol 220254 (BUS-P1-11)

Table 14.2-1.1 Plasma Concentrations (ng/mL) of Camlipixant (PK Concentration Population) - Part 1

| Γimepoint Γ | Camlipixant (Day 1) | Camlipixant + Rifampin (Day 11) |
|----------------|---------------------|---------------------------------|
| Statistic | (N=xx) | (N=xx) |
| Pre-dose | | |
| n | XX | XX |
| Number of BLQs | XX | XX |
| Mean | XXXX.XX | XXXX.XX |
| SD | XXXX.XX | XXXX.XX |
| CV% | XXX.XX | XXX.XX |
| Geometric Mean | XXXX.XX | XXXX.XX |
| Geometric SD | XXXX.XX | XXXX.XX |
| Geometric CV% | XXX.XX | XXX.XX |
| Min | XXXX.XX | XXXX.XX |
| Median | XXXX.XX | XXXX.XX |
| Max | XXXX.XX | XXXX.XX |
| X.XX | | |
| n | XX | XX |
| Number of BLQs | XX | XX |
| Mean | XXXX.XX | XXXX.XX |
| SD | XXXX.XX | XXXX.XX |
| CV% | XXX.XX | XXX.XX |
| Geometric Mean | XXXX.XX | XXXX.XX |
| Geometric SD | XXXX.XX | XXXX.XX |
| Geometric CV% | XXX.XX | XXX.XX |
| Min | XXXX.XX | XXXX.XX |
| Median | XXXX.XX | XXXX.XX |
| Max | XXXX.XX | XXXX.XX |

• • •

Abbreviations: BLQ=Below lower limit of quantification; CV%=Coefficient of variation (percent); max=Maximum; min=Minimum; N=Number of participants in the population; n=Number of observations; PK=Pharmacokinetic(s); SD=Standard deviation; '-'=Not calculated

Note: BLQ values were entered as zero for the determination of summary statistics with the exception of geometric mean, geometric SD, and geometric CV%, where BLQ values were imputed as half the lower limit of quantification (LLOQ) value. The LLOQ for camlipixant was 1 ng/mL.



- Programming Notes:
  1) Sort by timepoint.
  2) Present all scheduled timepoints.



Bellus Health Protocol 220254 (BUS-P1-11)

Table 14.2-1.2 Plasma Concentrations (ng/mL) of Camlipixant (PK Concentration Population) - Part 2

| Timepoint | Camlipixant (Day 1) | Camlipixant + Rabeprazole (Day 10) |
|----------------|---------------------|------------------------------------|
| Statistic | (N=xx) | (N=xx) |
| Pre-dose | | |
| n | XX | XX |
| Number of BLQs | XX | XX |
| Mean | XXXX.XX | XXXX.XX |
| SD | XXXX.XX | XXXX.XX |
| CV% | XXX.XX | XXX.XX |
| Geometric Mean | XXXX.XX | XXXX.XX |
| Geometric SD | XXXX.XX | XXXX.XX |
| Geometric CV% | XXX.XX | XXX.XX |
| Min | XXXX.XX | XXXX.XX |
| Median | XXXX.XX | XXXX.XX |
| Max | XXXX.XX | XXXX.XX |
| X.XX | | |
| n | XX | XX |
| Number of BLQs | XX | XX |
| Mean | XXXX.XX | XXXX.XX |
| SD | XXXX.XX | XXXX.XX |
| CV% | XXX.XX | XXX.XX |
| Geometric Mean | XXXX.XX | XXXX.XX |
| Geometric SD | XXXX.XX | XXXX.XX |
| Geometric CV% | XXX.XX | XXX.XX |
| Min | XXXX.XX | XXXX.XX |
| Median | XXXX.XX | XXXX.XX |
| Max | XXXX.XX | XXXX.XX |

Abbreviations: BLQ=Below lower limit of quantification; CV%=Coefficient of variation (percent); max=Maximum; min=Minimum; N=Number of participants in the population; n=Number of observations; PK=Pharmacokinetic(s); SD=Standard deviation; '-'=Not calculated

Note: BLQ values were entered as zero for the determination of summary statistics with the exception of geometric mean, geometric SD, and geometric CV%, where BLQ values were imputed as half the lower limit of quantification (LLOQ) value. The LLOQ for cambipixant was 1 ng/mL.



- Programming Notes:
  1) Sort by timepoint.
  2) Present all scheduled timepoints.



Bellus Health Protocol 220254 (BUS-P1-11)

Table 14.2-2.1 Plasma PK Parameters of Camlipixant (PK Parameter Population) - Part 1

| Parameter (unit) | Camlipixant (Day 1) | Camlipixant + Rifampin (Day 11) |
|-------------------|---------------------|---------------------------------|
| Statistic | (N=xx) | (N=xx) |
| AUG (-) | | |
| $AUC_{0-t}(xx)$ | | |
| n | XX | XX |
| Mean | XXXX.XX | XXXX.XX |
| SD | XXXX.XX | XXXX.XX |
| CV% | XXX.XX | XXX.XX |
| Geometric Mean | XXXX.XX | XXXX.XX |
| Geometric SD | XXXX.XX | XXXX.XX |
| Geometric CV% | XXX.XX | XXX.XX |
| Min | XXXX.XX | XXXX.XX |
| Median | XXXX.XX | XXXX.XX |
| Max | XXXX.XX | XXXX.XX |
| $AUC_{0-inf}(xx)$ | | |
| n | XX | XX |
| Mean | XXXX.XX | XXXX.XX |
| SD | XXXX.XX | XXXX.XX |
| CV% | XXX.XX | XXX.XX |
| Geometric Mean | XXXX.XX | XXXX.XX |
| Geometric SD | XXXX.XX | XXXX.XX |
| Geometric CV% | XXX.XX | XXX.XX |
| Min | XXXX.XX | XXXX.XX |
| Median | XXXX.XX | XXXX.XX |
| Max | XXXX.XX | XXXX.XX |

Abbreviations: CV%=Coefficient of variation (percent); max=Maximum; min=Minimum; N=Number of participants in the population; n=Number of observations; PK=Pharmacokinetic(s); SD=Standard deviation; '-'=Not calculated

Data Source: Listing 16.2.6.2-1

### Programming Notes:

1) Geometric mean will be set to "-" if minimum is zero.



- 2) Present all PK parameters in the order in which they are presented in the corresponding listing.
- 3) Add abbreviations used in the table to the footnotes.

Bellus Health Protocol 220254 (BUS-P1-11)

Table 14.2-2.2 Plasma PK Parameters of Camlipixant (PK Parameter Population) - Part 2

| Parameter (unit) | Camlipixant (Day 1) | Camlipixant + Rabeprazole (Day 10) |
|---|---|---|
| Statistic | (N=xx) | (N=xx) |
| $AUC_{0-t}(xx)$ | | |
| n | XX | XX |
| Mean | XXXX.XX | XXXX.XX |
| SD | XXXX.XX | XXXX.XX |
| CV% | XXX.XX | XXX.XX |
| Geometric Mean | XXXX.XX | XXXX.XX |
| Geometric SD | XXXX.XX | XXXX.XX |
| Geometric CV% | XXX.XX | XXX.XX |
| Min | XXXX.XX | XXXX.XX |
| Median | XXXX.XX | XXXX.XX |
| Max | XXXX.XX | XXXX.XX |
| $AUC_{0-inf}(xx)$ | | |
| n | XX | XX |
| Mean | XXXX.XX | XXXX.XX |
| SD | XXXX.XX | XXXX.XX |
| CV% | XXX.XX | XXX.XX |
| Geometric Mean | XXXX.XX | XXXX.XX |
| Geometric SD | XXXX.XX | XXXX.XX |
| Geometric CV% | XXX.XX | XXX.XX |
| Min | XXXX.XX | XXXX.XX |
| Median | XXXX.XX | XXXX.XX |
| Max | XXXX.XX | XXXX.XX |

Abbreviations: CV%=Coefficient of variation (percent); max=Maximum; min=Minimum; N=Number of participants in the population; n=Number of observations; PK=Pharmacokinetic(s); SD=Standard deviation; '-'=Not calculated

Data Source: Listing 16.2.6.2-2

## Programming Notes:

- 1) Geometric mean will be set to "-" if minimum is zero.
- 2) Present all PK parameters in the order in which they are presented in the corresponding listing.



Bellus Health Protocol 220254 (BUS-P1-11)

3) Add abbreviations used in the table to the footnotes.

Bellus Health Protocol 220254 (BUS-P1-11)

Table 14.2-3 Assessment of Rifampin Effect: DDI (PK Parameter Population) - Part 1

| Parameter (unit) | Treatment / Treatment<br>Comparison | Geometric<br>LSM | Geometric<br>LSM Ratio<br>(%) <sup>[a]</sup> | 90% CIs for the<br>Geometric LSM<br>Ratio (%) <sup>b]</sup> | Was the criteria for no DDI met? | Intra-<br>Subject<br>CV (%) <sup>[d]</sup> | Inter-<br>Subject<br>CV (%) <sup>[e]</sup> | p-value<br>Treatment |
|---|---|---|---|---|---|---|---|---|
| $\begin{array}{c} AUC_{0\text{-t}}(xx) \\ (n=xx) \end{array}$ | Camlipixant<br>Camlipixant + Rifampin<br>Camlipixant + Rifampin vs<br>Camlipixant | XXX.XX<br>XXX.XX | xx.xx | xx.xx, xx.xx | Yes | xxx.xx | xxx.xx | 0.xxxx |
| $\begin{array}{l} AUC_{0\text{-inf}}(xx)\\ (n=xx) \end{array}$ | Camlipixant Camlipixant + Rifampin Camlipixant + Rifampin vs Camlipixant | XXX.XX<br>XXX.XX | XX.XX | xx.xx, xx.xx | Yes | xxx.xx | xxx.xx | 0.xxxx |
| $C_{max}(xx)$ $(n=xx)$ | Camlipixant Camlipixant + Rifampin Camlipixant + Rifampin vs Camlipixant | XXX.XX<br>XXX.XX | xx.xx | xx.xx, xx.xx | Yes | xxx.xx | xxx.xx | 0.xxxx |

Abbreviations: ANOVA=Analysis of variance; CI=Confidence interval; CV=Coefficient of variation; DDI=Drug-drug interaction; exp=Exponential; df=Degrees of freedom; LSM=Least square means; n=Number of participants included in the analysis; p-value=Probability value; PK=Pharmacokinetic(s); SE=Standard error; SQRT=Square root; vs=Versus.

<sup>[</sup>a] The geometric LSM ratio (camlipixant + rifampin/camlipixant) is calculated using LSM according to the following formula: exp (DIFFERENCE) \* 100.

<sup>[</sup>b] The 90% geometric CI is calculated according to the following formula: exp (DIFFERENCE ± t<sub>(dfResidual)</sub>\* SE<sub>DIFFERENCE</sub>) \* 100.

<sup>[</sup>c] The ratio of geometric means (camlipixant + rifampin/camlipixant) and 90% CIs for the ratio of geometric means, based on least squares means from the repeated measure ANOVA of the ln transformed AUC<sub>0-inf</sub>, AUC<sub>0-inf</sub>, and C<sub>max</sub> must be within 80 % to 125 % to demonstrate no DDI.

<sup>[</sup>d] Calculated according to formula: SQRT (exp (residual variance) -1) \* 100.

<sup>[</sup>e] Calculated according to formula: SQRT (exp (subject variance) – 1) \* 100.



Bellus Health Protocol 220254 (BUS-P1-11)

Table 14.2-4 Assessment of Rabeprazole Effect: DDI (PK Parameter Population) - Part 2

| Parameter (unit) | Treatment / Treatment<br>Comparison | Geometric<br>LSM | Geometric<br>LSM Ratio<br>(%) <sup>[a]</sup> | 90% CIs for the<br>Geometric LSM<br>Ratio (%) <sup>b]</sup> | Was the criteria for no DDI met? [c] | Intra-<br>Subject<br>CV (%) <sup>[d]</sup> | Inter-<br>Subject<br>CV (%) <sup>[e]</sup> | p-value<br>Treatment |
|---|---|---|---|---|---|---|---|---|
| $\begin{array}{c} AUC_{0-t}(xx) \\ (n=xx) \end{array}$ | Camlipixant Camlipixant + Rabeprazole Camlipixant + Rabeprazole vs Camlipixant | XXX.XX<br>XXX.XX | xx.xx | xx.xx, xx.xx | Yes | xxx.xx | xxx.xx | 0.xxxx |
| $\begin{array}{c} AUC_{0\text{-inf}}(xx)\\ (n=xx) \end{array}$ | Camlipixant Camlipixant + Rabeprazole Camlipixant + Rabeprazole vs Camlipixant | XXX.XX<br>XXX.XX | xx.xx | xx.xx, xx.xx | Yes | xxx.xx | xxx.xx | 0.xxxx |
| $C_{max}(xx)$ $(n=xx)$ | Camlipixant Camlipixant + Rabeprazole Camlipixant + Rabeprazole vs Camlipixant | XXX.XX<br>XXX.XX | xx.xx | xx.xx, xx.xx | Yes | xxx.xx | xxx.xx | 0.xxxx |

Abbreviations: ANOVA=Analysis of variance; CI=Confidence interval; CV=Coefficient of variation; DDI=Drug-drug interaction; exp=Exponential; df=Degrees of freedom; LSM=Least square means; n=Number of participants included in the analysis; p-value=Probability value; PK=Pharmacokinetic(s); SE=Standard error; SQRT=Square root; vs=Versus.

<sup>[</sup>a] The geometric LSM ratio (camlipixant + rabeprazole/camlipixant) is calculated using LSM according to the following formula: exp (DIFFERENCE) \* 100.

<sup>[</sup>b] The 90% geometric CI is calculated according to the following formula: exp (DIFFERENCE ± t<sub>(dIResidual)</sub>\* SE<sub>DIFFERENCE</sub>) \* 100.

<sup>[</sup>c] The ratio of geometric means (camlipixant + rabeprazole/camlipixant) and 90% CIs for the ratio of geometric means, based on least squares means from the repeated measure ANOVA of the ln transformed AUC<sub>0-t</sub>, AUC<sub>0-inf</sub>, and C<sub>max</sub> must be within 80 % to 125 % to demonstrate no DDI.

<sup>[</sup>d] Calculated according to formula: SQRT (exp (residual variance) – 1) \* 100.

<sup>[</sup>e] Calculated according to formula: SQRT (exp (subject variance) – 1) \* 100.



Bellus Health Protocol 220254 (BUS-P1-11)

## Table 14.2-5 Non-Parametric Assessment of Rifampin Effect (PK Parameter Population) - Part 1

| Plasma PK<br>Parameter (unit) | Number of Participants Included in the Analysis | Treatment Comparison | Median of Paired Difference | Signed-Rank p-value |
|---|---|---|---|---|
| T <sub>max</sub> (unit) | XX | Camlipixant + Rifampin vs Camlipixant | xx.xxx | x.xxxx |

Abbreviations: p-value=Probability value



Bellus Health Protocol 220254 (BUS-P1-11)

Table 14.2-6 Non-Parametric Assessment of Rabeprazole Effect (PK Parameter Population) - Part 2

| Plasma PK Parameter (unit) | Number of<br>Participants<br>Included in the<br>Analysis | Treatment Comparison | Median of Paired Difference | Signed-Rank p-value |
|---|---|---|---|---|
| T <sub>max</sub> (unit) | xx | Camlipixant + Rabeprazole vs Camlipixant | xx.xxx | x.xxxx |

Abbreviations: p-value=Probability value



Bellus Health Protocol 220254 (BUS-P1-11)

Table 14.2-7.1 Attainment of Steady State (ng/mL) (PK Concentration Population) - Part 1

| Analyte | Statistic | Day 9 Pre-dose (N=xx) | Day 10 Pre-dose (N=xx) | Day 11 Pre-dose (N=xx) |
|---|---|---|---|---|
| Rifampin | n | XX | XX | XX |
| N<br>M<br>S<br>C<br>G<br>G<br>G | Number of BLQs | XX | XX | XX |
| | Mean | XXXX.XX | xxxx.xx | XXXX.XX |
| | SD | xxxx.xx | xxxx.xx | XXXX.XX |
| | CV% | XXX.XX | XXX.XX | xxx.xx |
| | Geometric Mean | xxxx.xx | xxxx.xx | XXXX.XX |
| | Geometric SD | xxxx.xx | xxxx.xx | XXXX.XX |
| | Geometric CV% | XXX.XX | XXX.XX | xxx.xx |
| | Min | xxxx.xx | xxxx.xx | XXXX.XX |
| | Median | xxxx.xx | xxxx.xx | XXXX.XX |
| | Max | xxxx.xx | xxxx.xx | XXXX.XX |

Abbreviations: BLQ=Below lower limit of quantification; CV%=Coefficient of variation (percent); max=Maximum; min=Minimum; N=Number of participants in the population; n=Number of observations; PK=Pharmacokinetic(s); SD=Standard deviation; '-'=Not calculated

Note: BLQ values were entered as zero for the determination of summary statistics with the exception of geometric mean, geometric SD, and geometric CV%, where BLQ values were imputed as half the lower limit of quantification (LLOQ) value. The LLOQ for rifampin was 5 ng/mL.



Bellus Health Protocol 220254 (BUS-P1-11)

Table 14.2-7.2 Attainment of Steady State (ng/mL) (PK Concentration Population) - Part 2

| Analyte | Statistic | Day 8 Pre-dose (N=xx) | Day 9 Pre-dose<br>(N=xx) | Day 10 Pre-dose<br>(N=xx) |
|---|---|---|---|---|
| Rabeprazole | n | XX | XX | XX |
| · | Number of BLQs | XX | XX | XX |
| | Mean | xxxx.xx | xxxx.xx | XXXX.XX |
| | SD | XXXX.XX | XXXX.XX | xxxx.xx |
| | CV% | XXX.XX | XXX.XX | XXX.XX |
| | Geometric Mean | XXXX.XX | XXXX.XX | xxxx.xx |
| | Geometric SD | XXXX.XX | XXXX.XX | xxxx.xx |
| | Geometric CV% | XXX.XX | XXX.XX | XXX.XX |
| | Min | xxxx.xx | xxxx.xx | xxxx.xx |
| | Median | xxxx.xx | xxxx.xx | XXXX.XX |
| | Max | xxxx.xx | xxxx.xx | XXXX.XX |

Abbreviations: BLQ=Below lower limit of quantification; CV%=Coefficient of variation (percent); max=Maximum; min=Minimum; N=Number of participants in the population; n=Number of observations; PK=Pharmacokinetic(s); SD=Standard deviation; '-'=Not calculated

Note: BLQ values were entered as zero for the determination of summary statistics with the exception of geometric mean, geometric SD, and geometric CV%, where BLQ values were imputed as half the lower limit of quantification (LLOQ) value. The LLOQ for rabeprazole was 0.5 ng/mL.

Bellus Health Protocol 220254 (BUS-P1-11)

Table 14.3.1-1.1 Overall Summary of TEAEs (Safety Population) - Part 1

| Category | Statistic | Camlipixant <sup>[b]</sup><br>(N=xx) | Rifampin <sup>[c]</sup><br>(N=xx) | Camlipixant + Rifampin $^{[d]}$ (N=xx) | Overall (N=xx) |
|---|---|---|---|---|---|
| TEAEs | n (%) E | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x |
| Study drug-related <sup>[a]</sup> TEAEs | n (%) E | x(xx.x)x | x ( xx.x) x | x (xx.x)x | x ( xx.x) x |
| Severe TEAEs | n (%) E | x(xx.x)x | x ( xx.x) x | x (xx.x)x | x(xx.x)x |
| Serious TEAEs | n (%) E | x(xx.x)x | x(xx.x)x | x ( xx.x) x | x ( xx.x) x |
| TEAEs leading to discontinuation | n (%) E | x(xx.x)x | x(xx.x)x | x ( xx.x) x | x ( xx.x) x |
| TEAEs leading to death | n (%) E | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x |

Abbreviations: E=Event; N=Number of participants in the population; n (%)=Number and percent of participants with TEAEs; TEAE=Treatment-emergent adverse event

Note: Each participant contributes once to each of the incidence rates, regardless of the number of occurrences.

The overall column includes participants from all treatment groups.

Treatment sequence: camlipixant 50 mg SD on Day 1, rifampin color mg color from Day 4 to Day 10, rifampin color mg color from Day 11 to 12 with co-administration of camlipixant 50 mg SD on Day 11.

Data Source: Listing 16.2.7.2-1 and Listing 16.2.7.3-1

<sup>[</sup>a] Study drug-related events are events to which the relationship is categorized as "Definite", "Probable", or "Possible"

<sup>[</sup>b] Attributed from Day 1 post-dose until Day 4 pre-dose of rifampin

<sup>[</sup>c] Attributed from Day 4 dosing until Day 11 pre-dose of camlipixant

<sup>[</sup>d] Attributed from camlipixant dosing on Day 11 until end of study



Bellus Health Protocol 220254 (BUS-P1-11)

Table 14.3.1-1.2 Overall Summary of TEAEs (Safety Population) - Part 2

| Category | Statistic | Camlipixant <sup>[b]</sup><br>(N=xx) | Rabeprazole [c]<br>(N=xx) | Camlipixant + Rabeprazole [d] (N=xx) | Overall (N=xx) |
|---|---|---|---|---|---|
| TEAEs | n (%) E | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x |
| Study drug-related <sup>[a]</sup> TEAEs | n (%) E | x(xx.x)x | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x |
| Severe TEAEs | n (%) E | x(xx.x)x | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x |
| Serious TEAEs | n (%) E | x(xx.x)x | x (xx.x) x | x ( xx.x) x | x(xx.x)x |
| TEAEs leading to discontinuation | n (%) E | x(xx.x)x | x (xx.x) x | x ( xx.x) x | x(xx.x)x |
| TEAEs leading to death | n (%) E | x ( xx.x) x | x ( xx.x) x | x(xx.x)x | x (xx.x) x |

Abbreviations: E=Event; N=Number of participants in the population; n (%)=Number and percent of participants with TEAEs; TEAE=Treatment-emergent adverse event

Note: Each participant contributes once to each of the incidence rates, regardless of the number of occurrences.

The overall column includes participants from all treatment groups.

Treatment sequence: camlipixant 50 mg SD on Day 1, rabeprazole mg ggg from Day 4 to Day 9, rabeprazole gg mg ggg from Day 10 to 11 with co-administration of camlipixant 50 mg SD on Day 10.

Data Source: Listing 16.2.7.2-2 and Listing 16.2.7.3-2

<sup>[</sup>a] Study drug-related events are events to which the relationship is categorized as "Definite", "Probable", or "Possible"

<sup>[</sup>b] Attributed from Day 1 post-dose until Day 4 pre-dose of rabeprazole

<sup>[</sup>c] Attributed from Day 4 dosing until Day 10 pre-dose of camlipixant

<sup>[</sup>d] Attributed from camlipixant dosing on Day 10 until end of study



Bellus Health Protocol 220254 (BUS-P1-11)

Table 14.3.1-2.1 TEAEs by SOC and PT (Safety Population) - Part 1

| Statistic | Camlipixant <sup>[a]</sup><br>(N=xx) | Rifampin <sup>[b]</sup> (N=xx) | Camlipixant +<br>Rifampin <sup>[c]</sup><br>(N=xx) | Overall<br>(N=xx) |
|---|---|---|---|---|
| n (%) E | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x |
| n (%) E | x(xx.x)x | x ( xx.x) x | x ( xx.x) x | x(xx.x)x |
| n (%) E | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x |
| n (%) E | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x |
| n (%) E | x(xx.x)x | x ( xx.x) x | x ( xx.x) x | x(xx.x)x |
| n (%) E | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x | x (xx.x) x |
| | n (%) E<br>n (%) E<br>n (%) E<br>n (%) E<br>n (%) E | n (%) E | n (%) E x (xx.x) x x (xx.x) x n (%) E x (xx.x) x x (xx.x) x n (%) E x (xx.x) x x (xx.x) x n (%) E x (xx.x) x x (xx.x) x n (%) E x (xx.x) x x (xx.x) x n (%) E x (xx.x) x x (xx.x) x | n (%) E x (xx.x) x x (xx.x) x x (xx.x) x n (%) E x (xx.x) x x (xx.x) x x (xx.x) x n (%) E x (xx.x) x x (xx.x) x x (xx.x) x n (%) E x (xx.x) x x (xx.x) x x (xx.x) x n (%) E x (xx.x) x x (xx.x) x x (xx.x) x n (%) E x (xx.x) x x (xx.x) x x (xx.x) x |

. . .

Abbreviations: E=Event; MedDRA=Medical Dictionary for Regulatory Activities; N=Number of participants in the population; n (%)=Number and percent of participants with TEAEs; PT=Preferred term; SOC=System organ class; TEAE=Treatment-emergent adverse event

Note: Each participant could only contribute once to each of the incidence rates within a system organ class and within a preferred term, regardless of the number of occurrences.

The overall column includes participants from all treatment groups.

Treatment sequence: camlipixant 50 mg SD on Day 1, rifampin color mg color from Day 4 to Day 10, rifampin color mg color from Day 11 to 12 with co-administration of camlipixant 50 mg SD on Day 11.

Adverse events were coded using MedDRA version X.X.

Data Source: Listing 16.2.7.2-1

#### Programming Notes:

- 1) SOC will be presented in descending order of overall incidence rate in terms of frequency of subjects and then in frequency of events (alphabetical order will be used in case of equal rates). For each SOC, PT will be presented the same way.
- 2) Refer to footnotes for additional instructions.
- 3) In the footnote, replace "X.X" with the actual MedDRA version used in the study.

<sup>[</sup>a] Attributed from Day 1 post-dose until Day 4 pre-dose of rifampin

<sup>[</sup>b] Attributed from Day 4 dosing until Day 11 pre-dose of camlipixant

<sup>[</sup>c] Attributed from camlipixant dosing on Day 11 until end of study

Bellus Health Protocol 220254 (BUS-P1-11)

Table 14.3.1-2.2 TEAEs by SOC and PT (Safety Population) - Part 2

| MedDRA® System Organ Class<br>MedDRA Preferred Term | Statistic | Camlipixant <sup>[a]</sup> (N=xx) | Rabeprazole <sup>[b]</sup> (N=xx) | Camlipixant + Rabeprazole <sup>[c]</sup> (N=xx) | Overall (N=xx) |
|---|---|---|---|---|---|
| SOC 1 | n (%) E | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x |
| PT 1 | n (%) E | x ( xx.x) x | x(xx.x)x | x(xx.x)x | x ( xx.x) x |
| PT 2 | n (%) E | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x |
| OC 1 | n (%) E | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x |
| PT 1 | n (%) E | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x |
| PT 2 | n (%) E | x ( xx.x) x | x(xx.x)x | x(xx.x)x | x ( xx.x) x |

. . .

Abbreviations: E=Event; MedDRA=Medical Dictionary for Regulatory Activities; N=Number of participants in the population; n (%)=Number and percent of participants with TEAEs; PT=Preferred term; SOC=System organ class; TEAE=Treatment-emergent adverse event

Note: Each participant could only contribute once to each of the incidence rates within a system organ class and within a preferred term, regardless of the number of occurrences.

The overall column includes participants from all treatment groups.

Treatment sequence: camlipixant 50 mg SD on Day 1, rabeprazole mg mg from Day 4 to Day 9, rabeprazole mg mg from Day 10 to 11 with coadministration of camlipixant 50 mg SD on Day 10.

Adverse events were coded using MedDRA version X.X.

Data Source: Listing 16.2.7.2-2

#### Programming Notes:

- 1) SOCs will be presented in descending order of overall incidence rate in terms of frequency of subjects and then in frequency of events (alphabetical order will be used in case of equal rates). For each SOC, PT will be presented the same way.
- 2) Refer to footnotes for additional instructions.
- 3) In the footnote, replace "X.X" with the actual MedDRA version used in the study.

<sup>[</sup>a] Attributed from Day 1 post-dose until Day 4 pre-dose of rabeprazole

<sup>[</sup>b] Attributed from Day 4 dosing until Day 10 pre-dose of camlipixant

<sup>[</sup>c] Attributed from camlipixant dosing on Day 10 until end of study
Bellus Health Protocol 220254 (BUS-P1-11)

Table 14.3.1-3.1 TEAEs by Severity (Safety Population) - Part 1

| MedDRA® System Organ Class MedDRA Preferred Term Severity | Statistic | Camlipixant <sup>[a]</sup><br>(N=xx) | Rifampin <sup>[b]</sup> (N=xx) | Camlipixant + Rifampin <sup>[c]</sup> (N=xx) | Overall (N=xx) |
|---|---|---|---|---|---|
| All TEAEs | n (%) E | x ( xx.x) x | x (xx.x) x | x ( xx.x) x | x ( xx.x) x |
| Mild | n (%) E | x ( xx.x) x | x(xx.x)x | x ( xx.x) x | x ( xx.x) x |
| Moderate | n (%) E | x ( xx.x) x | x(xx.x)x | x ( xx.x) x | x ( xx.x) x |
| Severe | n (%) E | x ( xx.x) x | x (xx.x) x | x ( xx.x) x | x ( xx.x) x |
| SOC 1 | n (%) E | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x |
| Mild | n (%) E | x ( xx.x) x | x (xx.x) x | x ( xx.x) x | x ( xx.x) x |
| Moderate | n (%) E | x ( xx.x) x | x(xx.x)x | x ( xx.x) x | x ( xx.x) x |
| Severe | n (%) E | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x |
| PT 1 | n (%) E | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x |
| Mild | n (%) E | x ( xx.x) x | x(xx.x)x | x ( xx.x) x | x (xx.x)x |
| Moderate | n (%) E | x ( xx.x) x | x (xx.x) x | x ( xx.x) x | x ( xx.x) x |
| Severe | n (%) E | x ( xx.x) x | x (xx.x) x | x ( xx.x) x | x ( xx.x) x |

Abbreviations: E=Event; MedDRA=Medical Dictionary for Regulatory Activities; N=Number of participants in the population; n (%)=Number and percent of participants with TEAEs; TEAE=Treatment-emergent adverse event

Note: Each participant could only contribute once to each of the incidence rates within a system organ class and within a preferred term, regardless of the number of occurrences using the highest reported severity.

The overall column includes participants from all treatment groups.

Treatment sequence: camlipixant 50 mg SD on Day 1, rifampin regimg from Day 4 to Day 10, rifampin regimg from Day 11 to 12 with co-administration of camlipixant 50 mg SD on Day 11.

Adverse events were coded using MedDRA version X.X.

Data Source: Listing 16.2.7.2-1

#### Programming Notes:

1) SOCs will be presented in descending order of overall incidence rate in terms of frequency of subjects and then in frequency of events (alphabetical order will be used in case of equal rates). For each SOC, PT will be presented the same way.

<sup>[</sup>a] Attributed from Day 1 post-dose until Day 4 pre-dose of rifampin

<sup>[</sup>b] Attributed from Day 4 dosing until Day 11 pre-dose of camlipixant

<sup>[</sup>c] Attributed from camlipixant dosing on Day 11 until end of study



Bellus Health Protocol 220254 (BUS-P1-11)

- 2) Refer to footnotes for additional instructions.
- 3) Add abbreviations used in the table to the footnotes.
- 4) In the footnote, replace "X.X" with the actual MedDRA version used in the study.

Bellus Health Protocol 220254 (BUS-P1-11)

Table 14.3.1-3.2 TEAEs by Severity (Safety Population) - Part 2

| MedDRA® System Organ Class<br>MedDRA Preferred Term<br>Severity | Statistic | Camlipixant <sup>[a]</sup><br>(N=xx) | Rabeprazole <sup>[b]</sup> (N=xx) | Camlipixant + Rabeprazole <sup>[c]</sup> (N=xx) | Overall (N=xx) |
|---|---|---|---|---|---|
| All TEAEs | n (%) E | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x |
| Mild | n (%) E | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x | x (xx.x) x<br>x (xx.x) x |
| Moderate | n (%) E | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x | x (xx.x) x |
| Severe | n (%) E | x ( xx.x) x | x (xx.x) x | x (xx.x) x | x (xx.x) x |
| SOC 1 | n (%) E | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x |
| Mild | n (%) E | x ( xx.x) x | x (xx.x)x | x (xx.x) x | x ( xx.x) x |
| Moderate | n (%) E | x(xx.x)x | x ( xx.x) x | x (xx.x) x | x ( xx.x) x |
| Severe | n (%) E | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x |
| PT 1 | n (%) E | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x |
| Mild | n (%) E | x ( xx.x) x | x (xx.x)x | x (xx.x) x | x ( xx.x) x |
| Moderate | n (%) E | x(xx.x)x | x (xx.x)x | x (xx.x) x | x ( xx.x) x |
| Severe | n (%) E | x ( xx.x) x | x (xx.x)x | x (xx.x) x | x (xx.x)x |

Abbreviations: E=Event; MedDRA=Medical Dictionary for Regulatory Activities; N=Number of participants in the population; n (%)=Number and percent of participants with TEAEs; TEAE=Treatment-emergent adverse event

Note: Each participant could only contribute once to each of the incidence rates within a system organ class and within a preferred term, regardless of the number of occurrences using the highest reported severity.

The overall column includes participants from all treatment groups.

Treatment sequence: camlipixant 50 mg SD on Day 1, rabeprazole common graph from Day 4 to Day 9, rabeprazole common graph from Day 10 to 11 with co-administration of camlipixant 50 mg SD on Day 10.

Adverse events were coded using MedDRA version X.X.

Data Source: Listing 16.2.7.2-2

#### Programming Notes:

1) SOCs will be presented in descending order of overall incidence rate in terms of frequency of subjects and then in frequency of events (alphabetical order will be used in case of equal rates). For each SOC, PT will be presented the same way.

<sup>[</sup>a] Attributed from Day 1 post-dose until Day 4 pre-dose of rabeprazole

<sup>[</sup>b] Attributed from Day 4 dosing until Day 10 pre-dose of camlipixant

<sup>[</sup>c] Attributed from camlipixant dosing on Day 10 until end of study



Bellus Health Protocol 220254 (BUS-P1-11)

- 2) Refer to footnotes for additional instructions.
- 3) Add abbreviations used in the table to the footnotes.
- 4) In the footnote, replace "X.X" with the actual MedDRA version used in the study.

Bellus Health Protocol 220254 (BUS-P1-11)

Table 14.3.1-4.1 TEAEs by Relationship to Study Drug (Camlipixant) (Safety Population) - Part 1

| | | Relationship to Ca | mlipixant | |
|---|---|---|---|---|
| MedDRA® System Organ Class<br>MedDRA Preferred Term<br>Relationship | Statistic | Camlipixant <sup>[a]</sup><br>(N=xx) | Camlipixant + Rifampin <sup>[b]</sup> (N=xx) | Overall (N=xx) |
| All TEAEs | n (%) E | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x |
| Definite | n (%) E | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x |
| Probable | n (%) E | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x |
| Possible | n (%) E | x (xx.x) x | x ( xx.x) x | x ( xx.x) x |
| Unlikely | n (%) E | x(xx.x)x | x(xx.x)x | x ( xx.x) x |
| Not Related | n (%) E | x ( xx.x) x | x (xx.x) x | x ( xx.x) x |
| SOC 1 | n (%) E | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x |
| Definite | n (%) E | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x |
| Probable | n (%) E | x(xx.x)x | x(xx.x)x | x ( xx.x) x |
| Possible | n (%) E | x ( xx.x) x | x(xx.x)x | x ( xx.x) x |
| Unlikely | n (%) E | x ( xx.x) x | x(xx.x)x | x ( xx.x) x |
| Not Related | n (%) E | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x |
| PT 1 | n (%) E | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x |
| Definite | n (%) E | x(xx.x)x | x(xx.x)x | x ( xx.x) x |
| Probable | n (%) E | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x |
| Possible | n (%) E | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x |
| Unlikely | n (%) E | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x |
| Not Related | n (%) E | x(xx.x)x | x ( xx.x) x | x ( xx.x) x |

Abbreviations: E=Event; MedDRA=Medical Dictionary for Regulatory Activities; N=Number of participants in the population; n (%)=Number and percent of participants with TEAEs; TEAE=Treatment-emergent adverse event

Note: Each participant could only contribute once to each of the incidence rates within a system organ class and within a preferred term, regardless of the number of occurrences using the worst reported relationship.

The overall column includes participants from all treatment groups.

Treatment sequence: camlipixant 50 mg SD on Day 1, rifampin col mg col from Day 4 to Day 10, rifampin col mg col from Day 11 to 12 with coadministration of camlipixant 50 mg SD on Day 11.

Adverse events were coded using MedDRA version X.X.

<sup>[</sup>a] Attributed from Day 1 post-dose until Day 4 pre-dose of rifampin [b] Attributed from camlipixant dosing on Day 11 until end of study



Bellus Health Protocol 220254 (BUS-P1-11)

Data Source: Listing 16.2.7.2-1

- 1) SOCs will be presented in descending order of overall incidence rate in terms of frequency of subjects and then in frequency of events (alphabetical order will be used in case of equal rates). For each SOC, PT will be presented the same way.
- 2) Refer to footnotes for additional instructions.
- 3) Add abbreviations used in the table to the footnotes.
- 4) In the footnote, replace "X.X" with the actual MedDRA version used in the study.

Bellus Health Protocol 220254 (BUS-P1-11)

Table 14.3.1-4.2 TEAEs by Relationship to Study Drug (Rifampin) (Safety Population) – Part 1

| | · | Relationship to R | Lifampin | <del></del> |
|---|---|---|---|---|
| MedDRA <sup>®</sup> System Organ Class<br>MedDRA Preferred Term<br>Relationship | Statistic | Rifampin <sup>[a]</sup><br>(N=xx) | Camlipixant + Rifampin <sup>[b]</sup> (N=xx) | Overall (N=xx) |
| All TEAEs | n (%) E | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x |
| Definite | n (%) E | x ( xx.x) x | x (xx.x) x | x ( xx.x) x |
| Probable | n (%) E | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x |
| Possible | n (%) E | x (xx.x) x | x(xx.x)x | x ( xx.x) x |
| Unlikely | n (%) E | x (xx.x) x | x(xx.x)x | x ( xx.x) x |
| Not Related | n (%) E | x ( xx.x) x | x (xx.x) x | x ( xx.x) x |
| SOC 1 | n (%) E | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x |
| Definite | n (%) E | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x |
| Probable | n (%) E | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x |
| Possible | n (%) E | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x |
| Unlikely | n (%) E | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x |
| Not Related | n (%) E | x ( xx.x) x | x (xx.x) x | x ( xx.x) x |
| PT 1 | n (%) E | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x |
| Definite | n (%) E | x (xx.x) x | x(xx.x)x | x ( xx.x) x |
| Probable | n (%) E | x ( xx.x) x | x(xx.x)x | x ( xx.x) x |
| Possible | n (%) E | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x |
| Unlikely | n (%) E | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x |
| Not Related | n (%) E | x ( xx.x) x | x ( xx.x) x | x(xx.x)x |

Abbreviations: E=Event; MedDRA=Medical Dictionary for Regulatory Activities; N=Number of participants in the population; n (%)=Number and percent of participants with TEAEs; TEAE=Treatment-emergent adverse event

Note: Each participant could only contribute once to each of the incidence rates within a system organ class and within a preferred term, regardless of the number of occurrences using the worst reported relationship.

The overall column includes participants from all treatment groups.

Treatment sequence: camlipixant 50 mg SD on Day 1, rifampin col mg col from Day 4 to Day 10, rifampin col mg col from Day 11 to 12 with coadministration of camlipixant 50 mg SD on Day 11.

Adverse events were coded using MedDRA version X.X.

<sup>[</sup>a] Attributed from Day 4 dosing until Day 11 pre-dose of camlipixant [b] Attributed from camlipixant dosing on Day 11 until end of study



Bellus Health Protocol 220254 (BUS-P1-11)

Data Source: Listing 16.2.7.2-1

- 1) SOCs will be presented in descending order of overall incidence rate in terms of frequency of subjects and then in frequency of events (alphabetical order will be used in case of equal rates). For each SOC, PT will be presented the same way.
- 2) Refer to footnotes for additional instructions.
- 3) Add abbreviations used in the table to the footnotes.
- 4) In the footnote, replace "X.X" with the actual MedDRA version used in the study.

Bellus Health Protocol 220254 (BUS-P1-11)

Table 14.3.1-4.3 TEAEs by Relationship to Study Drug (Camlipixant) (Safety Population) - Part 2

| | | Relationship to Ca | ımlipixant | |
|---|---|---|---|---|
| MedDRA® System Organ Class<br>MedDRA Preferred Term<br>Relationship | Statistic | Camlipixant <sup>[a]</sup><br>(N=xx) | Camlipixant + Rabeprazole <sup>[b]</sup> (N=xx) | Overall (N=xx) |
| All TEAEs | n (%) E | x ( xx.x) x | x ( xx.x) x | x (xx.x) x |
| Definite | n (%) E | x ( xx.x) x | x ( xx.x) x | x(xx.x) |
| Probable | n (%) E | x ( xx.x) x | x ( xx.x) x | x(xx.x) |
| Possible | n (%) E | x ( xx.x) x | x(xx.x)x | x(xx.x)x |
| Unlikely | n (%) E | x(xx.x)x | x ( xx.x) x | x(xx.x)x |
| Not Related | n (%) E | x(xx.x)x | x ( xx.x) x | x ( xx.x) x |
| SOC 1 | n (%) E | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x |
| Definite | n (%) E | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x |
| Probable | n (%) E | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x |
| Possible | n (%) E | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x |
| Unlikely | n (%) E | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x |
| Not Related | n (%) E | x(xx.x)x | x ( xx.x) x | x (xx.x) x |
| PT 1 | n (%) E | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x |
| Definite | n (%) E | x (xx.x) x | x ( xx.x) x | x (xx.x) x |
| Probable | n (%) E | x (xx.x)x | x ( xx.x) x | x (xx.x) x |
| Possible | n (%) E | x (xx.x)x | x ( xx.x) x | x (xx.x) x |
| Unlikely | n (%) E | x (xx.x)x | x ( xx.x) x | x ( xx.x) x |
| Not Related | n (%) E | x (xx.x)x | x ( xx.x) x | x (xx.x) x |

Abbreviations: E=Event; MedDRA=Medical Dictionary for Regulatory Activities; N=Number of participants in the population; n (%)=Number and percent of participants with TEAEs; TEAE=Treatment-emergent adverse event

Note: Each participant could only contribute once to each of the incidence rates within a system organ class and within a preferred term, regardless of the number of occurrences using the worst reported relationship.

The overall column includes participants from all treatment groups.

Treatment sequence: camlipixant 50 mg SD on Day 1, rabeprazole comg confrom Day 4 to Day 9, rabeprazole comg confrom Day 10 to 11 with coadministration of camlipixant 50 mg SD on Day 10.

Adverse events were coded using MedDRA version X.X.

<sup>[</sup>a] Attributed from Day 1 post-dose until Day 4 pre-dose of rabeprazole
[b] Attributed from camlipixant dosing on Day 10 until end of study



Bellus Health Protocol 220254 (BUS-P1-11)

Data Source: Listing 16.2.7.2-2

- 1) SOCs will be presented in descending order of overall incidence rate in terms of frequency of subjects and then in frequency of events (alphabetical order will be used in case of equal rates). For each SOC, PT will be presented the same way.
- 2) Refer to footnotes for additional instructions.
- 3) Add abbreviations used in the table to the footnotes.
- 4) In the footnote, replace "X.X" with the actual MedDRA version used in the study.

Bellus Health Protocol 220254 (BUS-P1-11)

Table 14.3.1-4.4 TEAEs by Relationship to Study Drug (Rabeprazole) (Safety Population) - Part 2

| | | Relationship to Ra | beprazole | |
|---|---|---|---|---|
| MedDRA® System Organ Class<br>MedDRA Preferred Term<br>Relationship | Statistic | Rabeprazole <sup>[a]</sup><br>(N=xx) | Camlipixant + Rabeprazole <sup>[b]</sup> (N=xx) | Overall (N=xx) |
| All TEAEs | n (%) E | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x |
| Definite | n (%) E | x(xx.x)x | x ( xx.x) x | x ( xx.x) x |
| Probable | n (%) E | x(xx.x)x | x ( xx.x) x | x ( xx.x) x |
| Possible | n (%) E | x(xx.x)x | x ( xx.x) x | x ( xx.x) x |
| Unlikely | n (%) E | x(xx.x)x | x ( xx.x) x | x ( xx.x) x |
| Not Related | n (%) E | x(xx.x)x | x ( xx.x) x | x ( xx.x) x |
| SOC 1 | n (%) E | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x |
| Definite | n (%) E | x ( xx.x) x | x(xx.x)x | x ( xx.x) x |
| Probable | n (%) E | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x |
| Possible | n (%) E | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x |
| Unlikely | n (%) E | x(xx.x)x | x(xx.x)x | x ( xx.x) x |
| Not Related | n (%) E | x(xx.x)x | x ( xx.x) x | x(xx.x)x |
| PT 1 | n (%) E | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x |
| Definite | n (%) E | x (xx.x)x | x(xx.x)x | x ( xx.x) x |
| Probable | n (%) E | x (xx.x)x | x(xx.x)x | x ( xx.x) x |
| Possible | n (%) E | x (xx.x)x | x(xx.x)x | x ( xx.x) x |
| Unlikely | n (%) E | x(xx.x)x | x(xx.x)x | x ( xx.x) x |
| Not Related | n (%) E | x(xx.x)x | x(xx.x)x | x ( xx.x) x |

Abbreviations: E=Event; MedDRA=Medical Dictionary for Regulatory Activities; N=Number of participants in the population; n (%)=Number and percent of participants with TEAEs; TEAE=Treatment-emergent adverse event

Note: Each participant could only contribute once to each of the incidence rates within a system organ class and within a preferred term, regardless of the number of occurrences using the worst reported relationship.

The overall column includes participants from all treatment groups.

Treatment sequence: camlipixant 50 mg SD on Day 1, rabeprazole colmg col from Day 4 to Day 9, rabeprazole colmg col from Day 10 to 11 with coadministration of camlipixant 50 mg SD on Day 10.

Adverse events were coded using MedDRA version X.X.

<sup>[</sup>a] Attributed from Day 4 dosing until Day 10 pre-dose of camlipixant [b] Attributed from camlipixant dosing on Day 10 until end of study



Bellus Health Protocol 220254 (BUS-P1-11)

Data Source: Listing 16.2.7.2-2

- 1) SOCs will be presented in descending order of overall incidence rate in terms of frequency of subjects and then in frequency of events (alphabetical order will be used in case of equal rates). For each SOC, PT will be presented the same way.
- 2) Refer to footnotes for additional instructions.
- 3) Add abbreviations used in the table to the footnotes.
- 4) In the footnote, replace "X.X" with the actual MedDRA version used in the study.

Bellus Health Protocol 220254 (BUS-P1-11)

Table 14.3.1-5.1 Serious TEAEs (Safety Population) - Part 1

| MedDRA® System Organ Class<br>MedDRA Preferred Term | Statistic | Camlipixant <sup>[a]</sup><br>(N=xx) | Rifampin <sup>[b]</sup><br>(N=xx) | Camlipixant +<br>Rifampin <sup>[c]</sup><br>(N=xx) | Overall (N=xx) |
|---|---|---|---|---|---|
| SOC 1 | n (%) E | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x |
| PT 1 | n (%) E | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x |
| PT 2 | n (%) E | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x |
| SOC 1 | n (%) E | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x |
| PT 1 | n (%) E | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x |
| PT 2 | n (%) E | x(xx.x)x | x ( xx.x) x | x(xx.x)x | x ( xx.x) x |

Abbreviations: E=Event; MedDRA=Medical Dictionary for Regulatory Activities; N=Number of participants in the population; n (%)=Number and percent of participants with TEAEs; TEAE=Treatment-emergent adverse event

Note: Each participant could only contribute once to each of the incidence rates within a system organ class and within a preferred term, regardless of the number of occurrences.

The overall column includes participants from all treatment groups.

Treatment sequence: camlipixant 50 mg SD on Day 1, rifampin color mg color from Day 4 to Day 10, rifampin color mg color from Day 11 to 12 with co-administration of camlipixant 50 mg SD on Day 11.

Adverse events were coded using MedDRA version X.X.

Data Source: Listing 16.2.7.3-1

- 1) SOCs will be presented in descending order of overall incidence rate in terms of frequency of subjects and then in frequency of events (alphabetical order will be used in case of equal rates). For each SOC, PT will be presented the same way.
- 2) Refer to footnotes for additional instructions.
- 3) Add abbreviations used in the table to the footnotes.
- 4) In the footnote, replace "X.X" with the actual MedDRA version used in the study.

<sup>[</sup>a] Attributed from Day 1 post-dose until Day 4 pre-dose of rifampin

<sup>[</sup>b] Attributed from Day 4 dosing until Day 11 pre-dose of camlipixant

<sup>[</sup>c] Attributed from camlipixant dosing on Day 11 until end of study

Bellus Health Protocol 220254 (BUS-P1-11)

Table 14.3.1-5.2 Serious TEAEs (Safety Population) - Part 2

| MedDRA® System Organ Class<br>MedDRA Preferred Term | Statistic | Camlipixant <sup>[a]</sup><br>(N=xx) | Rabeprazole <sup>[b]</sup> (N=xx) | Camlipixant + Rabeprazole <sup>[c]</sup> (N=xx) | Overall (N=xx) |
|---|---|---|---|---|---|
| SOC 1 | n (%) E | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x |
| PT 1 | n (%) E | x ( xx.x) x | x ( xx.x) x | x(xx.x)x | x ( xx.x) x |
| PT 2 | n (%) E | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x |
| SOC 1 | n (%) E | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x |
| PT 1 | n (%) E | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x |
| PT 2 | n (%) E | x(xx.x)x | x(xx.x)x | x(xx.x)x | x ( xx.x) x |

. . .

Abbreviations: E=Event; MedDRA=Medical Dictionary for Regulatory Activities; N=Number of participants in the population; n (%)=Number and percent of participants with TEAEs; TEAE=Treatment-emergent adverse event

Note: Each participant could only contribute once to each of the incidence rates within a system organ class and within a preferred term, regardless of the number of occurrences.

The overall column includes participants from all treatment groups.

Treatment sequence: camlipixant 50 mg SD on Day 1, rabeprazole mg mg from Day 4 to Day 9, rabeprazole mg mg from Day 10 to 11 with coadministration of camlipixant 50 mg SD on Day 10.

Adverse events were coded using MedDRA version X.X.

Data Source: Listing 16.2.7.3-2

- 1) SOCs will be presented in descending order of overall incidence rate in terms of frequency of subjects and then in frequency of events (alphabetical order will be used in case of equal rates). For each SOC, PT will be presented the same way.
- 2) Refer to footnotes for additional instructions.
- 3) Add abbreviations used in the table to the footnotes.
- 4) In the footnote, replace "X.X" with the actual MedDRA version used in the study.

<sup>[</sup>a] Attributed from Day 1 post-dose until Day 4 pre-dose of rabeprazole

<sup>[</sup>b] Attributed from Day 4 dosing until Day 10 pre-dose of camlipixant

<sup>[</sup>c] Attributed from camlipixant dosing on Day 10 until end of study

Bellus Health Protocol 220254 (BUS-P1-11)

Table 14.3.1-6.1 Treatment-emergent AEMIs (Safety Population) - Part 1

| MedDRA® System Organ Class<br>MedDRA Preferred Term | Statistic | Camlipixant <sup>[a]</sup><br>(N=xx) | Rifampin <sup>[b]</sup> (N=xx) | Camlipixant +<br>Rifampin <sup>[c]</sup><br>(N=xx) | Overall (N=xx) |
|---|---|---|---|---|---|
| SOC 1 | n (%) E | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x |
| PT 1 | n (%) E | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x |
| PT 2 | n (%) E | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x |
| SOC 1 | n (%) E | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x |
| PT 1 | n (%) E | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x |
| PT 2 | n (%) E | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x |

Abbreviations: AEMI=Adverse events of medical interest; E=Event; MedDRA=Medical Dictionary for Regulatory Activities; N=Number of participants in the population; n (%)=Number and percent of participants with TEAEs

Note: Each participant could only contribute once to each of the incidence rates within a system organ class and within a preferred term, regardless of the number of occurrences.

The overall column includes participants from all treatment groups.

Treatment sequence: camlipixant 50 mg SD on Day 1, rifampin common management of mg SD on Day 11 to 12 with co-administration of camlipixant 50 mg SD on Day 11.

Adverse events were coded using MedDRA version X.X.

Data Source: Listing 16.2.7.4-1

- 1) SOCs will be presented in descending order of overall incidence rate in terms of frequency of subjects and then in frequency of events (alphabetical order will be used in case of equal rates). For each SOC, PT will be presented the same way.
- 2) Refer to footnotes for additional instructions.
- 3) Add abbreviations used in the table to the footnotes.
- 4) In the footnote, replace "X.X" with the actual MedDRA version used in the study.

<sup>[</sup>a] Attributed from Day 1 post-dose until Day 4 pre-dose of rifampin

<sup>[</sup>b] Attributed from Day 4 dosing until Day 11 pre-dose of camlipixant

<sup>[</sup>c] Attributed from camlipixant dosing on Day 11 until end of study

Bellus Health Protocol 220254 (BUS-P1-11)

Table 14.3.1-6.2 Treatment-emergent AEMIs (Safety Population) - Part 2

| MedDRA® System Organ Class<br>MedDRA Preferred Term | Statistic | Camlipixant <sup>[a]</sup><br>(N=xx) | Rabeprazole <sup>[b]</sup> (N=xx) | Camlipixant + Rabeprazole <sup>[c]</sup> (N=xx) | Overall (N=xx) |
|---|---|---|---|---|---|
| SOC 1 | n (%) E | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x |
| PT 1 | n (%) E | x ( xx.x) x | x(xx.x)x | x(xx.x)x | x ( xx.x) x |
| PT 2 | n (%) E | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x |
| SOC 1 | n (%) E | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x |
| PT 1 | n (%) E | x ( xx.x) x | x(xx.x)x | x(xx.x)x | x ( xx.x) x |
| PT 2 | n (%) E | x(xx.x)x | x(xx.x)x | x(xx.x)x | x(xx.x)x |

. . .

Abbreviations: AEMI=Adverse events of medical interest; E=Event; MedDRA=Medical Dictionary for Regulatory Activities; N=Number of participants in the population; n (%)=Number and percent of participants with TEAEs

Note: Each participant could only contribute once to each of the incidence rates within a system organ class and within a preferred term, regardless of the number of occurrences.

The overall column includes participants from all treatment groups.

Treatment sequence: camlipixant 50 mg SD on Day 1, rabeprazole comg mg from Day 4 to Day 9, rabeprazole comg mg from Day 10 to 11 with coadministration of camlipixant 50 mg SD on Day 10.

Adverse events were coded using MedDRA version X.X.

Data Source: Listing 16.2.7.4-2

- 1) SOCs will be presented in descending order of overall incidence rate in terms of frequency of subjects and then in frequency of events (alphabetical order will be used in case of equal rates). For each SOC, PT will be presented the same way.
- 2) Refer to footnotes for additional instructions.
- 3) Add abbreviations used in the table to the footnotes.
- 4) In the footnote, replace "X.X" with the actual MedDRA version used in the study.

<sup>[</sup>a] Attributed from Day 1 post-dose until Day 4 pre-dose of rabeprazole

<sup>[</sup>b] Attributed from Day 4 dosing until Day 10 pre-dose of camlipixant

<sup>[</sup>c] Attributed from camlipixant dosing on Day 10 until end of study

Bellus Health Protocol 220254 (BUS-P1-11)

## Table 14.3.4-1.1 Biochemistry (Safety Population) - Part 1

| Parameter (unit) Normal Range Study Day Statistic | Overall<br>(N=xx) |
|---------------------------------------------------|-------------------|
| xxxxxxx (xx)<br>xxx-xxx | |
| AAA-AAA | |
| Day x (Baseline) | |
| n | XX |
| Mean | XX.X |
| SD | XX.XX |
| Min | XX.X |
| Median | XX.X |
| Max | XX.X |
| Day x | |
| n | XX |
| Mean | XX.X |
| SD | XX.XX |
| Min | XX.X |
| Median | XX.X |
| Max | XX.X |
| Day x - CFB | |
| n | XX |
| Mean | XX.X |
| SD | XX.XX |
| Min | XX.X |
| Median | XX.X |
| Max | XX.X |

Abbreviations: CFB=Change from baseline; max=Maximum; min=Minimum; N=Number of participants in the population; n=Number of observations; SD=Standard deviation

Note: Baseline is defined as the last result (scheduled or unscheduled) obtained prior to first study drug administration on Day 1.

# Data Source: Listing 16.2.8.1-1

- 1) Sort by parameter, in alphabetical order, and study day, in chronological order.
- 2) Present all parameters.
  - a. Start a new page for each parameter.
- 3) Present all scheduled visits.
- 4) Independently for each parameter, if the baseline assessment for all subjects is on the same study day, identify the study day with "(Baseline)" [e.g., Day 1 (Baseline)]. Otherwise, the baseline would have to be summarized separately and identified as "Baseline".
- 5) Add abbreviations used in the table to the footnotes.

## Table 14.3.4-1.2 Biochemistry (Safety Population) - Part 2

| Parameter (unit) | |
|------------------|---------|
| Normal Range | Overall |
| Study Day | (N=xx) |
| Statistic | |
| xxxxxx (xx) | |
| XXX-XXX | |
| Day x (Baseline) | |
| n | XX |
| Mean | XX.X |
| SD | XX.XX |
| Min | XX.X |
| Median | XX.X |
| Max | XX.X |
| Day x | |
| n | XX |
| Mean | XX.X |
| SD | XX.XX |
| Min | XX.X |
| Median | XX.X |
| Max | XX.X |
| Day x - CFB | |
| n | XX |
| Mean | XX.X |
| SD | XX.XX |
| Min | XX.X |
| Median | XX.X |
| Max | XX.X |
| 1116/1 | AAA |
| ••• | |

Abbreviations: CFB=Change from baseline; max=Maximum; min=Minimum; N=Number of participants in the population; n=Number of observations; SD=Standard deviation

Note: Baseline is defined as the last result (scheduled or unscheduled) obtained prior to first study drug administration on Day 1.

Data Source: Listing 16.2.8.1-2

- 1) Sort by parameter, in alphabetical order, and study day, in chronological order.
- 2) Present all parameters.
  - a. Start a new page for each parameter.
- 3) Present all scheduled visits.
- 4) Independently for each parameter, if the baseline assessment for all subjects is on the same study day, identify the study day with "(Baseline)" [e.g., Day 1 (Baseline)]. Otherwise, the baseline would have to be summarized separately and identified as "Baseline".
- 5) Add abbreviations used in the table to the footnotes.

Bellus Health Protocol 220254 (BUS-P1-11)

Table 14.3.4-2.1 Biochemistry Shifts from Baseline (Safety Population) - Part 1

| | | | Post Baseline | | |
|---|---|---|---|---|---|
| Parameter (unit) | Study Day | Baseline | Low<br>n (%) | Normal<br>n (%) | High<br>n (%) |
| xxxxxxx (xx) | Day x | Low<br>Normal<br>High | x ( xx.x)<br>x ( xx.x)<br>x ( xx.x) | x ( xx.x)<br>x ( xx.x)<br>x ( xx.x) | x ( xx.x)<br>x ( xx.x)<br>x ( xx.x) |

. . .

Abbreviations: n (%)=Number and percentage of participants

Note: Percentages are based on the number of participants having available results at baseline and at post-baseline. Baseline is defined as the last result (scheduled or unscheduled) obtained prior to first study drug administration on Day 1.

Data Source: Listing 16.2.8.1-1

- 1) Sort by parameter, in alphabetical order, and study day, in chronological order.
- 2) Present all scheduled post-baseline visits.
- 3) Present all parameters.
- 4) Add abbreviations used in the table to the footnotes.

Bellus Health Protocol 220254 (BUS-P1-11)

Table 14.3.4-2.2 Biochemistry Shifts from Baseline (Safety Population) - Part 2

| | | | Post Baseline | | |
|---|---|---|---|---|---|
| Parameter (unit) | Study Day | Baseline | Low<br>n (%) | Normal<br>n (%) | High<br>n (%) |
| xxxxxxx (xx) | Day x | Low<br>Normal<br>High | x ( xx.x)<br>x ( xx.x)<br>x ( xx.x) | x ( xx.x)<br>x ( xx.x)<br>x ( xx.x) | x ( xx.x)<br>x ( xx.x)<br>x ( xx.x) |

. . .

Abbreviations: n (%)=Number and percentage of participants

Note: Percentages are based on the number of participants having available results at baseline and at post-baseline. Baseline is defined as the last result (scheduled or unscheduled) obtained prior to first study drug administration on Day 1.

Data Source: Listing 16.2.8.1-2

- 1) Sort by parameter, in alphabetical order, and study day, in chronological order.
- 2) Present all scheduled post-baseline visits.
- 3) Present all parameters.
- 4) Add abbreviations used in the table to the footnotes.

Bellus Health Protocol 220254 (BUS-P1-11)

## Table 14.3.4-3.1 Hematology (Safety Population) - Part 1

| Parameter (unit) | |
|------------------|---------|
| Normal Range | Overall |
| Study Day | (N=xx) |
| Statistic | |
| xxxxxxx (xx) | |
| XXX-XXX | |
| Day x (Baseline) | |
| n | XX |
| Mean | XX.X |
| SD | XX.XX |
| Min | XX.X |
| Median | XX.X |
| Max | XX.X |
| D | |
| Day x | |
| n<br>M | XX |
| Mean | XX.X |
| SD | XX.XX |
| Min | XX.X |
| Median | XX.X |
| Max | XX.X |
| Day x - CFB | |
| n | XX |
| Mean | XX.X |
| SD | XX.XX |
| Min | XX.X |
| Median | XX.X |
| Max | XX.X |
| ••• | |

Abbreviations: CFB=Change from baseline; max=Maximum; min=Minimum; N=Number of participants in the population; n=Number of observations; SD=Standard deviation

Note: Baseline is defined as the last result (scheduled or unscheduled) obtained prior to first study drug administration on Day 1.

Data Source: Listing 16.2.8.2-1

- 1) Sort by parameter, in alphabetical order, and study day, in chronological order.
- 2) Present all parameters.
  - a. Start a new page for each parameter.
- 3) Present all scheduled visits.
- 4) Independently for each parameter, if the baseline assessment for all subjects is on the same study day, identify the study day with "(Baseline)" [e.g., Day 1 (Baseline)]. Otherwise, the baseline would have to be summarized separately and identified as "Baseline".
- 5) Add abbreviations used in the table to the footnotes.

Bellus Health Protocol 220254 (BUS-P1-11)

## Table 14.3.4-3.2 Hematology (Safety Population) - Part 2

| Parameter (unit) Normal Range Study Day Statistic | Overall<br>(N=xx) |
|---------------------------------------------------|-------------------|
| xxxxxxx (xx)<br>xxx-xxx | |
| AAA-AAA | |
| Day x (Baseline) | |
| n | XX |
| Mean | XX.X |
| SD | XX.XX |
| Min | XX.X |
| Median | XX.X |
| Max | XX.X |
| Day x | |
| n | XX |
| Mean | XX.X |
| SD | XX.XX |
| Min | XX.X |
| Median | XX.X |
| Max | XX.X |
| Day x - CFB | |
| n | XX |
| Mean | XX.X |
| SD | XX.XX |
| Min | XX.X |
| Median | XX.X |
| Max | XX.X |

Abbreviations: CFB=Change from baseline; max=Maximum; min=Minimum; N=Number of participants in the population; n=Number of observations; SD=Standard deviation

Note: Baseline is defined as the last result (scheduled or unscheduled) obtained prior to first study drug administration on Day 1.

Data Source: Listing 16.2.8.2-2

- 1) Sort by parameter, in alphabetical order, and study day, in chronological order.
- 2) Present all parameters.
  - a. Start a new page for each parameter.
- 3) Present all scheduled visits.
- 4) Independently for each parameter, if the baseline assessment for all subjects is on the same study day, identify the study day with "(Baseline)" [e.g., Day 1 (Baseline)]. Otherwise, the baseline would have to be summarized separately and identified as "Baseline".
- 5) Add abbreviations used in the table to the footnotes.

Bellus Health Protocol 220254 (BUS-P1-11)

Table 14.3.4-4.1 Hematology Shifts from Baseline (Safety Population) - Part 1

| | | | Post Baseline | | |
|---|---|---|---|---|---|
| Parameter (unit) | Study Day | Baseline | Low<br>n (%) | Normal<br>n (%) | High<br>n (%) |
| xxxxxxx (xx) | Day x | Low<br>Normal<br>High | x ( xx.x)<br>x ( xx.x)<br>x ( xx.x) | x ( xx.x)<br>x ( xx.x)<br>x ( xx.x) | x ( xx.x)<br>x ( xx.x)<br>x ( xx.x) |

. . .

Abbreviations: n (%)=Number and percentage of participants

Note: Percentages are based on the number of participants having available results at baseline and at post-baseline. Baseline is defined as the last result (scheduled or unscheduled) obtained prior to first study drug administration on Day 1.

Data Source: Listing 16.2.8.2-1

- 1) Sort by parameter, in alphabetical order, and study day, in chronological order.
- 2) Present all treatment groups.
  - a. Start a new page for each treatment group.
- 3) Present all scheduled post-baseline visits.
- 4) Present all parameters.
- 5) Add abbreviations used in the table to the footnotes.

Bellus Health Protocol 220254 (BUS-P1-11)

Table 14.3.4-4.2 Hematology Shifts from Baseline (Safety Population) - Part 2

| | | | Post Baseline | | |
|---|---|---|---|---|---|
| Parameter (unit) | Study Day | Baseline | Low<br>n (%) | Normal<br>n (%) | High<br>n (%) |
| xxxxxxx (xx) | Day x | Low<br>Normal | x ( xx.x)<br>x ( xx.x) | x ( xx.x)<br>x ( xx.x) | x ( xx.x)<br>x ( xx.x) |
| | | High | x ( xx.x) | x ( xx.x) | x(xx.x) |

. . .

Abbreviations: n (%)=Number and percentage of participants

Note: Percentages are based on the number of participants having available results at baseline and at post-baseline. Baseline is defined as the last result (scheduled or unscheduled) obtained prior to first study drug administration on Day 1.

Data Source: Listing 16.2.8.2-2

- 1) Sort by parameter, in alphabetical order, and study day, in chronological order.
- 2) Present all scheduled post-baseline visits.
- 3) Present all parameters.
- 4) Add abbreviations used in the table to the footnotes.

Bellus Health Protocol 220254 (BUS-P1-11)

## Table 14.3.4-5.1 Coagulation (Safety Population) - Part 1

| Parameter (unit) | |
|------------------|---------|
| Normal Range | Overall |
| Study Day | (N=xx) |
| Statistic | , , |
| xxxxxxx (xx) | |
| XXX-XXX | |
| Day x (Baseline) | |
| n | XX |
| Mean | XX.X |
| SD | XX.XX |
| Min | XX.X |
| Median | XX.X |
| Max | XX.X |
| Day x | |
| n | XX |
| Mean | XX.X |
| SD | XX.XX |
| Min | XX.X |
| Median | XX.X |
| Max | XX.X |
| Day x - CFB | |
| n | XX |
| Mean | XX.X |
| SD | XX.XX |
| Min | XX.X |
| Median | XX.X |
| Max | XX.X |
| ••• | |

Abbreviations: CFB=Change from baseline; max=Maximum; min=Minimum; N=Number of participants in the population; n=Number of observations; SD=Standard deviation

Note: Baseline is defined as the last result (scheduled or unscheduled) obtained prior to first study drug administration on Day 1.

Data Source: Listing 16.2.8.3-1

- 1) Sort by parameter, in alphabetical order, and study day, in chronological order.
- 2) Present all parameters.
  - a. Start a new page for each parameter.
- 3) Present all scheduled visits.
- 4) Independently for each parameter, if the baseline assessment for all subjects is on the same study day, identify the study day with "(Baseline)" [e.g., Day 1 (Baseline)]. Otherwise, the baseline would have to be summarized separately and identified as "Baseline".
- 5) Add abbreviations used in the table to the footnotes.

## Table 14.3.4-5.2 Coagulation (Safety Population) - Part 2

| Parameter (unit) | |
|------------------|---------|
| Normal Range | Overall |
| Study Day | (N=xx) |
| Statistic | |
| xxxxxxx (xx) | |
| xxx-xxx | |
| Day x (Baseline) | |
| n | XX |
| Mean | XX.X |
| SD | XX.XX |
| Min | XX.X |
| Median | XX.X |
| Max | XX.X |
| Day x | |
| n | XX |
| Mean | XX.X |
| SD | XX.XX |
| Min | XX.X |
| Median | XX.X |
| Max | XX.X |
| Day x - CFB | |
| n | XX |
| Mean | XX.X |
| SD | XX.XX |
| Min | XX.X |
| Median | XX.X |
| Max | XX.X |

Abbreviations: CFB=Change from baseline; max=Maximum; min=Minimum; N=Number of participants in the population; n=Number of observations; SD=Standard deviation

Note: Baseline is defined as the last result (scheduled or unscheduled) obtained prior to first study drug administration on Day 1.

Data Source: Listing 16.2.8.3-2

- 1) Sort by parameter, in alphabetical order, and study day, in chronological order.
- 2) Present all parameters.
  - a. Start a new page for each parameter.
- 3) Present all scheduled visits.
- 4) Independently for each parameter, if the baseline assessment for all subjects is on the same study day, identify the study day with "(Baseline)" [e.g., Day 1 (Baseline)]. Otherwise, the baseline would have to be summarized separately and identified as "Baseline".
- 5) Add abbreviations used in the table to the footnotes.

Bellus Health Protocol 220254 (BUS-P1-11)

Table 14.3.4-6.1 Coagulation Shifts from Baseline (Safety Population) - Part 1

| | | | Post Baseline | | |
|---|---|---|---|---|---|
| Parameter (unit) | Study Day | Baseline | Low<br>n (%) | Normal<br>n (%) | High<br>n (%) |
| xxxxxxx (xx) | Day x | Low<br>Normal<br>High | x ( xx.x)<br>x ( xx.x)<br>x ( xx.x) | x ( xx.x)<br>x ( xx.x)<br>x ( xx.x) | x ( xx.x)<br>x ( xx.x)<br>x ( xx.x) |

. . .

Abbreviations: n (%)=Number and percentage of participants

Note: Percentages are based on the number of participants having available results at baseline and at post-baseline. Baseline is defined as the last result (scheduled or unscheduled) obtained prior to first study drug administration on Day 1.

Data Source: Listing 16.2.8.3-1

- 1) Sort by parameter, in alphabetical order, and study day, in chronological order.
- 2) Present all scheduled post-baseline visits.
- 3) Present all parameters.
- 4) Add abbreviations used in the table to the footnotes.

Bellus Health Protocol 220254 (BUS-P1-11)

Table 14.3.4-6.2 Coagulation Shifts from Baseline (Safety Population) - Part 2

| | | | Post Baseline | | |
|---|---|---|---|---|---|
| Parameter (unit) | Study Day | Baseline | Low<br>n (%) | Normal<br>n (%) | High<br>n (%) |
| xxxxxxx (xx) | Day x | Low<br>Normal<br>High | x ( xx.x)<br>x ( xx.x)<br>x ( xx.x) | x ( xx.x)<br>x ( xx.x)<br>x ( xx.x) | x ( xx.x)<br>x ( xx.x)<br>x ( xx.x) |

. . .

Abbreviations: n (%)=Number and percentage of participants

Note: Percentages are based on the number of participants having available results at baseline and at post-baseline. Baseline is defined as the last result (scheduled or unscheduled) obtained prior to first study drug administration on Day 1.

Data Source: Listing 16.2.8.3-2

- 1) Sort by parameter, in alphabetical order, and study day, in chronological order.
- 2) Present all scheduled post-baseline visits.
- 3) Present all parameters.
- 4) Add abbreviations used in the table to the footnotes.

Bellus Health Protocol 220254 (BUS-P1-11)

## Table 14.3.4-7.1 Urinalysis: Quantitative (Safety Population) - Part 1

| Parameter (unit) Normal Range Study Day Statistic | Overall<br>(N=xx) |
|---------------------------------------------------|-------------------|
| xxxxxxx (xx)<br>xxx-xxx | |
| AAA-AAA | |
| Day x (Baseline) | |
| n | XX |
| Mean | XX.X |
| SD | XX.XX |
| Min | XX.X |
| Median | XX.X |
| Max | XX.X |
| Day x | |
| n | XX |
| Mean | XX.X |
| SD | XX.XX |
| Min | XX.X |
| Median | XX.X |
| Max | XX.X |
| Day x - CFB | |
| n | XX |
| Mean | XX.X |
| SD | XX.XX |
| Min | XX.X |
| Median | XX.X |
| Max | XX.X |

Abbreviations: CFB=Change from baseline; max=Maximum; min=Minimum; N=Number of participants in the population; n=Number of observations; SD=Standard deviation

Note: Baseline is defined as the last result (scheduled or unscheduled) obtained prior to first study drug administration on Day 1.

Data Source: Listing 16.2.8.4-1

- 1) Sort by parameter, in alphabetical order, and study day, in chronological order.
- 2) Present all parameters.
  - a. Start a new page for each parameter.
- 3) Present all scheduled visits.
- 4) Independently for each parameter, if the baseline assessment for all subjects is on the same study day, identify the study day with "(Baseline)" [e.g., Day 1 (Baseline)]. Otherwise, the baseline would have to be summarized separately and identified as "Baseline".
- 5) Add abbreviations used in the table to the footnotes.

Bellus Health Protocol 220254 (BUS-P1-11)

## Table 14.3.4-7.2 Urinalysis: Quantitative (Safety Population) - Part 2

| | · |
|------------------|---------------------------------------|
| Parameter (unit) | |
| Normal Range | Overall |
| Study Day | (N=xx) |
| Statistic | |
| xxxxxxx (xx) | |
| XXX-XXX | |
| Day x (Baseline) | |
| n | XX |
| Mean | XX.X |
| SD | XX.XX |
| Min | XX.X |
| Median | XX.X |
| Max | XX.X |
| Day x | |
| n | XX |
| Mean | XX.X |
| SD | XX.XX |
| Min | XX.X |
| Median | XX.X |
| Max | XX.X |
| Day x - CFB | |
| n | XX |
| Mean | XX.X |
| SD | XX.XX |
| Min | |
| Median | XX.X<br>XX.X |
| Max | |
| IVIAA | XX.X |
| ••• | |

Abbreviations: CFB=Change from baseline; max=Maximum; min=Minimum; N=Number of participants in the population; n=Number of observations; SD=Standard deviation

Note: Baseline is defined as the last result (scheduled or unscheduled) obtained prior to first study drug administration on Day 1.

Data Source: Listing 16.2.8.4-2

- 1) Sort by parameter, in alphabetical order, and study day, in chronological order.
- 2) Present all parameters.
  - a. Start a new page for each parameter.
- 3) Present all scheduled visits.
- 4) Independently for each parameter, if the baseline assessment for all subjects is on the same study day, identify the study day with "(Baseline)" [e.g., Day 1 (Baseline)]. Otherwise, the baseline would have to be summarized separately and identified as "Baseline".
- 5) Add abbreviations used in the table to the footnotes.

Bellus Health Protocol 220254 (BUS-P1-11)

Table 14.3.4-8.1 Urinalysis: Quantitative Shifts from Baseline (Safety Population) - Part 1

| | | | Post Baseline | | |
|---|---|---|---|---|---|
| Parameter (unit) | Study Day | Baseline | Low<br>n (%) | Normal<br>n (%) | High<br>n (%) |
| xxxxxxx (xx) | Day x | Low<br>Normal<br>High | x ( xx.x)<br>x ( xx.x)<br>x ( xx.x) | x ( xx.x)<br>x ( xx.x)<br>x ( xx.x) | x ( xx.x)<br>x ( xx.x)<br>x ( xx.x) |

. . .

Abbreviations: n (%)=Number and percentage of participants

Note: Percentages are based on the number of participants having available results at baseline and at post-baseline. Baseline is defined as the last result (scheduled or unscheduled) obtained prior to first study drug administration on Day 1.

Data Source: Listing 16.2.8.4-1

- 1) Sort by parameter, in alphabetical order, and study day, in chronological order.
- 2) Present all scheduled post-baseline visits.
- 3) Present all parameters.
- 4) Add abbreviations used in the table to the footnotes.

Bellus Health Protocol 220254 (BUS-P1-11)

Table 14.3.4-8.2 Urinalysis: Quantitative Shifts from Baseline (Safety Population) - Part 2

| | | | Post Baseline | | |
|---|---|---|---|---|---|
| Parameter (unit) | Study Day | Baseline | Low n (%) | Normal<br>n (%) | High<br>n (%) |
| xxxxxxx (xx) | Day x | Low<br>Normal<br>High | x ( xx.x)<br>x ( xx.x)<br>x ( xx.x) | x ( xx.x)<br>x ( xx.x)<br>x ( xx.x) | x ( xx.x)<br>x ( xx.x)<br>x ( xx.x) |

. . .

Abbreviations: n (%)=Number and percentage of participants

Note: Percentages are based on the number of participants having available results at baseline and at post-baseline. Baseline is defined as the last result (scheduled or unscheduled) obtained prior to first study drug administration on Day 1.

Data Source: Listing 16.2.8.4-2

- 1) Sort by parameter, in alphabetical order, and study day, in chronological order.
- 2) Present all scheduled post-baseline visits.
- 3) Present all parameters.
- 4) Add abbreviations used in the table to the footnotes.

Bellus Health Protocol 220254 (BUS-P1-11)

Table 14.3.4-9.1 Urinalysis: Categorical (Safety Population) - Part 1

| Parameter (unit) | Study Day | Result | Overall (N=xx) n (%) |
|---|---|---|---|
| xxxxxxx (xx) | Day x (Baseline) | Negative<br>Trace | x ( xx.x)<br>x ( xx.x) |
| | Day x | Negative<br>Trace | x ( xx.x)<br>x ( xx.x) |

Abbreviations: N=Number of participants in the population; n (%)=Number and percentage of participants Note: Baseline is defined as the last result (scheduled or unscheduled) obtained prior to first study drug administration on Day 1.

Data Source: Listing 16.2.8.5-1

- 1) Sort by parameter, in alphabetical order, and study day, in chronological order.
- 2) Present categorical parameters.
  - a. Start a new page for each categorical parameter.
- 3) Present all scheduled post-baseline visits.
- 4) Add abbreviations used in the table to the footnotes.

Bellus Health Protocol 220254 (BUS-P1-11)

Table 14.3.4-9.2 Urinalysis: Categorical (Safety Population) - Part 2

| Parameter (unit) | Study Day | Result | Overall (N=xx) n (%) |
|---|---|---|---|
| xxxxxxx (xx) | Day x (Baseline) | Negative<br>Trace | x ( xx.x)<br>x ( xx.x) |
| | Day x | Negative<br>Trace | x ( xx.x)<br>x ( xx.x) |
| ••• | | | |

Abbreviations: N=Number of participants in the population; n (%)=Number and percentage of participants Note: Baseline is defined as the last result (scheduled or unscheduled) obtained prior to first study drug administration on Day 1.

Data Source: Listing 16.2.8.5-2

- 1) Sort by parameter, in alphabetical order, and study day, in chronological order.
- 2) Present categorical parameters.
  - a. Start a new page for each categorical parameter.
- 3) Present all scheduled post-baseline visits.
- 4) Add abbreviations used in the table to the footnotes.

Bellus Health Protocol 220254 (BUS-P1-11)

## Table 14.3.4-10.1 Vital Signs (Safety Population) - Part 1

| Parameter (unit) | |
|------------------|---------|
| Normal Range | Overall |
| Study Day | (N=xx) |
| Statistic | |
| xxxxxxx (xx) | |
| XXX-XXX | |
| Day x (Baseline) | |
| n | XX |
| Mean | XX.X |
| SD | XX.XX |
| Min | XX.X |
| Median | XX.X |
| Max | XX.X |
| Day x | |
| n | XX |
| Mean | XX.X |
| SD | XX.XX |
| Min | XX.X |
| Median | XX.X |
| Max | XX.X |
| Day x - CFB | |
| n | XX |
| Mean | XX.X |
| SD | XX.XX |
| Min | XX.X |
| Median | XX.X |
| Max | XX.X |

Abbreviations: CFB=Change from baseline; max=Maximum; min=Minimum; N=Number of participants in the population; n=Number of observations; SD=Standard deviation

Note: Baseline is defined as the last result (scheduled or unscheduled) obtained prior to first study drug administration on Day 1.

Data Source: Listing 16.2.8.6-1

- 1) Sort by parameter, in alphabetical order, and study day, in chronological order.
- 2) Present all parameters.
  - a. Start a new page for each parameter.
- 3) Present all scheduled visits.
- 4) Independently for each parameter, if the baseline assessment for all subjects is on the same study day, identify the study day with "(Baseline)" [e.g., Day 1 (Baseline)]. Otherwise, the baseline would have to be summarized separately and identified as "Baseline".
- 5) Add abbreviations used in the table to the footnotes.

Bellus Health Protocol 220254 (BUS-P1-11)

# Table 14.3.4-10.2 Vital Signs (Safety Population) - Part 2

| Parameter (unit) | |
|------------------|---------|
| Normal Range | Overall |
| Study Day | (N=xx) |
| Statistic | |
| xxxxxxx (xx) | |
| XXX-XXX | |
| Day x (Baseline) | |
| n | XX |
| Mean | XX.X |
| SD | XX.XX |
| Min | XX.X |
| Median | XX.X |
| Max | XX.X |
| Day x | |
| n | XX |
| Mean | XX.X |
| SD | XX.XX |
| Min | XX.X |
| Median | XX.X |
| Max | XX.X |
| Day x - CFB | |
| n | XX |
| Mean | XX.X |
| SD | XX.XX |
| Min | XX.X |
| Median | XX.X |
| Max | XX.X |

Abbreviations: CFB=Change from baseline; max=Maximum; min=Minimum; N=Number of participants in the population; n=Number of observations; SD=Standard deviation

Note: Baseline is defined as the last result (scheduled or unscheduled) obtained prior to first study drug administration on Day 1.

Data Source: Listing 16.2.8.6-2

- 1) Sort by parameter, in alphabetical order, and study day, in chronological order.
- 2) Present all parameters.
  - a. Start a new page for each parameter.
- 3) Present all scheduled visits.
- 4) Independently for each parameter, if the baseline assessment for all subjects is on the same study day, identify the study day with "(Baseline)" [e.g., Day 1 (Baseline)]. Otherwise, the baseline would have to be summarized separately and identified as "Baseline".
- 5) Add abbreviations used in the table to the footnotes.
Bellus Health Protocol 220254 (BUS-P1-11)

Table 14.3.4-11.1 Vital Signs Shifts from Baseline (Safety Population) - Part 1

| | | | Post Basel | ine | | |
|---|---|---|---|---|---|---|
| Parameter (unit) | Study Day | Baseline | Normal<br>n (%) | Abnormal NCS n (%) | Abnormal CS<br>n (%) | Missing n(%) |
| xxxxxxx (xx) | Day x | Normal | x (xx.x) | x(xx.x) | x (xx.x) | x ( xx.x) |
| | | Abnormal NCS | x(xx.x) | x(xx.x) | x(xx.x) | x(xx.x) |
| | | Abnormal CS | x(xx.x) | x (xx.x) | x (xx.x) | x(xx.x) |
| | | Missing | x(xx.x) | x(xx.x) | x(xx.x) | x(xx.x) |

Abbreviations: CS=Clinically significant; n (%)=Number and percentage of participants; NCS=Not clinically significant

Note: Percentages are based on the number of participants having available results at baseline and at post-baseline. Baseline is defined as the last result (scheduled or unscheduled) obtained prior to first study drug administration on Day 1.

Data Source: Listing 16.2.8.6-1

- 1) Sort by parameter, in alphabetical order, and study day, in chronological order.
- 2) Present all scheduled post-baseline visits.
- 3) Present all parameters.
- 4) Add abbreviations used in the table to the footnotes.

Bellus Health Protocol 220254 (BUS-P1-11)

Table 14.3.4-11.2 Vital Signs Shifts from Baseline (Safety Population) - Part 2

| | | | Post Baseli | ne | • | |
|---|---|---|---|---|---|---|
| Parameter (unit) | Study Day | Baseline | Normal<br>n (%) | Abnormal NCS n (%) | Abnormal CS<br>n (%) | Missing n(%) |
| xxxxxxx (xx) | Day x | Normal<br>Abnormal NCS<br>Abnormal CS<br>Missing | x ( xx.x)<br>x ( xx.x)<br>x ( xx.x)<br>x ( xx.x) | x ( xx.x)<br>x ( xx.x)<br>x ( xx.x)<br>x ( xx.x) | x ( xx.x)<br>x ( xx.x)<br>x ( xx.x)<br>x ( xx.x) | x ( xx.x)<br>x ( xx.x)<br>x ( xx.x)<br>x ( xx.x) |

Abbreviations: CS=Clinically significant; n (%)=Number and percentage of participants; NCS=Not clinically significant

Note: Percentages are based on the number of participants having available results at baseline and at post-baseline. Baseline is defined as the last result (scheduled or unscheduled) obtained prior to first study drug administration on Day 1.

Data Source: Listing 16.2.8.6-2

- 1) Sort by parameter, in alphabetical order, and study day, in chronological order.
- 2) Present all scheduled post-baseline visits.
- 3) Present all parameters.
- 4) Add abbreviations used in the table to the footnotes.

Bellus Health Protocol 220254 (BUS-P1-11)

#### Table 14.3.4-12.1 ECGs: Quantitative (Safety Population) - Part 1

| Parameter (unit) Normal Range Study Day Statistic | Overall (N=xx) |
|---------------------------------------------------|----------------|
| xxxxxxx (xx) | |
| XXX-XXX | |
| Day x (Baseline) | |
| n | XX |
| Mean | XX.X |
| SD | XX.XX |
| Min | XX.X |
| Median | XX.X |
| Max | XX.X |
| Day x | |
| n | XX |
| Mean | XX.X |
| SD | XX.XX |
| Min | XX.X |
| Median | XX.X |
| Max | XX.X |
| Day x - CFB | |
| n | XX |
| Mean | XX.X |
| SD | XX.XX |
| Min | XX.X |
| Median | XX.X |
| Max | XX.X |

Abbreviations: CFB=Change from baseline; max=Maximum; min=Minimum; N=Number of participants in the population; n=Number of observations; SD=Standard deviation

Note: Baseline is defined as the last result (scheduled or unscheduled) obtained prior to first study drug administration on Day 1.

Data Source: Listing 16.2.8.7-1

- 1) Sort by parameter, in alphabetical order, and study day, in chronological order.
- 2) Present all parameters.
  - a. Start a new page for each parameter.
- 3) Present all scheduled visits.
- 4) Independently for each parameter, if the baseline assessment for all subjects is on the same study day, identify the study day with "(Baseline)" [e.g., Day 1 (Baseline)]. Otherwise, the baseline would have to be summarized separately and identified as "Baseline".
- 5) Add abbreviations used in the table to the footnotes.

Bellus Health Protocol 220254 (BUS-P1-11)

### Table 14.3.4-12.2 ECGs: Quantitative (Safety Population) - Part 2

| Parameter (unit) | |
|------------------|---------|
| Normal Range | Overall |
| Study Day | (N=xx) |
| Statistic | • |
| xxxxxxx (xx) | |
| XXX-XXX | |
| Day x (Baseline) | |
| n | XX |
| Mean | XX.X |
| SD | XX.XX |
| Min | XX.X |
| Median | XX.X |
| Max | XX.X |
| Day x | |
| n | XX |
| Mean | XX.X |
| SD | XX.XX |
| Min | XX.X |
| Median | XX.X |
| Max | XX.X |
| Day x - CFB | |
| n | XX |
| Mean | XX.X |
| SD | XX.XX |
| Min | XX.X |
| Median | XX.X |
| Max | XX.X |

Abbreviations: CFB=Change from baseline; max=Maximum; min=Minimum; N=Number of participants in the population; n=Number of observations; SD=Standard deviation

Note: Baseline is defined as the last result (scheduled or unscheduled) obtained prior to first study drug administration on Day 1.

Data Source: Listing 16.2.8.7-2

- 1) Sort by parameter, in alphabetical order, and study day, in chronological order.
- 2) Present all parameters.
  - a. Start a new page for each parameter.
- 3) Present all scheduled visits.
- 4) Independently for each parameter, if the baseline assessment for all subjects is on the same study day, identify the study day with "(Baseline)" [e.g., Day 1 (Baseline)]. Otherwise, the baseline would have to be summarized separately and identified as "Baseline".
- 5) Add abbreviations used in the table to the footnotes.

Bellus Health Protocol 220254 (BUS-P1-11)

Table 14.3.4-13.1 ECGs: Interpretation Shifts from Baseline (Safety Population) - Part 1

| Study Day | Baseline | Normal<br>n (%) | Abnormal NCS<br>n (%) | Abnormal CS<br>n (%) | Missing<br>n (%) |
|---|---|---|---|---|---|
| Day x | Normal | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) |
| | Abnormal NCS | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) |
| | Abnormal CS | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) |
| | Missing | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) |

Abbreviations: CS=Clinically significant; n (%)=Number and percentage of participants; NCS=Not clinically significant;

Note: Percentages are based on the number of participants having available results at baseline and at post-baseline. Baseline is defined as the last result (scheduled or unscheduled) obtained prior to first study drug administration on Day 1.

Data Source: Listing 16.2.8.7-1

- 1) Sort by parameter, in alphabetical order, and study day, in chronological order.
- 2) Present all scheduled post-baseline visits.
- 3) Present all parameters.
- 4) Add abbreviations used in the table to the footnotes.

Bellus Health Protocol 220254 (BUS-P1-11)

Table 14.3.4-13.2 ECGs: Interpretation Shifts from Baseline (Safety Population) - Part 2

| Study Day | Baseline | Post Baseline<br>Normal<br>n (%) | Abnormal NCS<br>n (%) | Abnormal CS<br>n (%) | Missing n (%) |
|---|---|---|---|---|---|
| Day x | Normal | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) |
| | Abnormal NCS | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) |
| | Abnormal CS | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) |
| | Missing | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) |

Abbreviations: CS=Clinically significant; n (%)=Number and percentage of participants; NCS=Not clinically significant

Note: Percentages are based on the number of participants having available results at baseline and at post-baseline. Baseline is defined as the last result (scheduled or unscheduled) obtained prior to first study drug administration on Day 1.

Data Source: Listing 16.2.8.7-2

- 1) Sort by parameter, in alphabetical order, and study day, in chronological order.
- 2) Present all scheduled post-baseline visits.
- 3) Present all parameters.
- 4) Add abbreviations used in the table to the footnotes.

Bellus Health Protocol 220254 (BUS-P1-11)

# 2. Figures



Bellus Health Protocol 220254 (BUS-P1-11)

# Figure 14.2-14.1 Individual Plasma Concentrations of Camlipixant - Linear Scale (PK Concentration Population) - Part 1

Plots of individual plasma concentrations over time, by treatment group for each participant.

Figure Description: The individual plasma concentrations over time will be presented by treatment group (or day) for each participant. The figure will display values for all treatment groups for a particular participant on a single page. Straight lines will connect the values for each treatment (or day). Different symbols, colors and line types will be used to distinguish between each treatment (or day).

For each figure, the X axis will be the actual timepoint. The Y axis will be the concentration, in units.

X axis title: Actual Timepoint (Hours) Y axis title: Concentration (units)

Abbreviations: PK= pharmacokinetic(s)

Data Source: Listing 16.2.6.1-1

- 1) Include all scheduled visits/timepoints.
- 2) Provide for each subject.



Bellus Health Protocol 220254 (BUS-P1-11)

# Figure 14.2-14.2 Individual Plasma Concentrations of Camlipixant – Linear Scale (PK Concentration Population) – Part 2

Plots of individual plasma concentrations over time, by treatment group for each participant.

Figure Description: The individual plasma concentrations over time will be presented by treatment group (or day) for each participant. The figure will display values for all treatment groups for a particular participant on a single page. Straight lines will connect the values for each treatment (or day). Different symbols, colors and line types will be used to distinguish between each treatment (or day).

For each figure, the X axis will be the actual timepoint. The Y axis will be the concentration, in units.

X axis title: Actual Timepoint (Hours) Y axis title: Concentration (units)

Abbreviations: PK= pharmacokinetic(s)

Data Source: Listing 16.2.6.1-2

- 1) Include all scheduled visits/timepoints.
- 2) Provide for each subject.



Bellus Health Protocol 220254 (BUS-P1-11)

# Figure 14.2-15.1 Individual Plasma Concentrations of Camlipixant - Semi-Log Scale (PK Concentration Population) - Part 1

Plots of individual plasma concentrations (log scale) over time, by treatment group for each participant.

Figure Description: The individual plasma concentrations (log scale) over time will be presented by treatment group (or day) for each participant. The figure will display values for all treatment groups for a particular participant on a single page. Straight lines will connect the values for each treatment (or day). Different symbols, colors and line types will be used to distinguish between each treatment (or day).

For each figure, the X axis will be the actual timepoint. The Y axis will be the concentration, in units.

X axis title: Actual Timepoint (Hours) Y axis title: Concentration (units)

Abbreviations: PK= pharmacokinetic(s)

Data Source: Listing 16.2.6.1-1

- 1) Include all scheduled visits/timepoints.
- 2) Provide for each subject.



Bellus Health Protocol 220254 (BUS-P1-11)

# Figure 14.2-15.2 Individual Plasma Concentrations of Camlipixant – Semi-Log Scale (PK Concentration Population) – Part 2

Plots of individual plasma concentrations (log scale) over time, by treatment group for each participant.

Figure Description: The individual plasma concentrations (log scale) over time will be presented by treatment group (or day) for each participant. The figure will display values for all treatment groups for a particular participant on a single page. Straight lines will connect the values for each treatment (or day). Different symbols, colors and line types will be used to distinguish between each treatment (or day).

For each figure, the X axis will be the actual timepoint. The Y axis will be the concentration, in units.

X axis title: Actual Timepoint (Hours) Y axis title: Concentration (units)

Abbreviations: PK= pharmacokinetic(s)

Data Source: Listing 16.2.6.1-2

#### **Programming Notes:**

1) Include all scheduled visits/timepoints.

2) Provide for each subject.



Bellus Health Protocol 220254 (BUS-P1-11)

# Figure 14.2-16.1 Mean (±SD) Plasma Concentrations of Camlipixant - Linear Scale (PK Concentration Population) - Part 1

Plot of mean plasma concentrations over time

Figure Description: The mean plasma concentration over time ( $\pm$ SD) will be presented. The figure will display values for all treatment groups on a single page. Straight lines will connect the values within each treatment group. Different symbols, colors and line types will be used to distinguish between each treatment group. The SD at each point will be added.

For each figure, the X axis will be the scheduled (nominal) timepoint. The Y axis will be the concentration, in units.

X axis title: Nominal Timepoint (Hours) Y axis title: Concentration (units)

Abbreviations: SD= standard deviation; PK= pharmacokinetic(s)

Data Source: Listing 16.2.6.1-1

#### Programming Notes:



Bellus Health Protocol 220254 (BUS-P1-11)

# Figure 14.2-16.2 Mean (±SD) Plasma Concentrations of Camlipixant - Linear Scale (PK Concentration Population) - Part 2

Plot of mean plasma concentrations over time

Figure Description: The mean plasma concentration over time  $(\pm SD)$  will be presented. The figure will display values for all treatment groups on a single page. Straight lines will connect the values within each treatment group. Different symbols, colors and line types will be used to distinguish between each treatment group. The SD at each point will be added.

For each figure, the X axis will be the scheduled (nominal) timepoint. The Y axis will be the concentration, in units.

X axis title: Nominal Timepoint (Hours) Y axis title: Concentration (units)

Abbreviations: SD= standard deviation; PK= pharmacokinetic(s)

Data Source: Listing 16.2.6.1-2

#### Programming Notes:



Bellus Health Protocol 220254 (BUS-P1-11)

# Figure 14.2-17.1 Mean (±SD) Plasma Concentrations of Camlipixant - Semi-Log Scale (PK Concentration Population) - Part 1

Plot of mean plasma concentrations (log scale) over time

Figure Description: The mean plasma concentrations (log scale) over time will be presented. The figure will display values for all treatment groups on a single page. Straight lines will connect the values within each treatment group. Different symbols, colors and line types will be used to distinguish between each treatment group.

For each figure, the X axis will be the scheduled (nominal) timepoint. The Y axis will be the concentration, in units.

X axis title: Nominal Timepoint (Hours) Y axis title: Concentration (units)

Abbreviations: SD= standard deviation; PK= pharmacokinetic(s)

Data Source: Listing 16.2.6.1-1

#### **Programming Notes:**



# Figure 14.2-17.2 Mean (±SD) Plasma Concentrations of Camlipixant - Semi-Log Scale (PK Concentration Population) - Part 2

Plot of mean plasma concentrations (log scale) over time

Figure Description: The mean plasma concentrations (log scale) over time will be presented. The figure will display values for all treatment groups on a single page. Straight lines will connect the values within each treatment group. Different symbols, colors and line types will be used to distinguish between each treatment group.

For each figure, the X axis will be the scheduled (nominal) timepoint. The Y axis will be the concentration, in units.

X axis title: Nominal Timepoint (Hours) Y axis title: Concentration (units)

Abbreviations: SD= standard deviation; PK= pharmacokinetic(s)

Data Source: Listing 16.2.6.1-2

#### **Programming Notes:**



### Figure 14.2-18.1 Overlay of Individual Plasma Concentrations of Camlipixant - Linear Scale (PK Concentration Population) - Part 1

Plots of overlay individual plasma concentrations over time for all participants, by treatment group.

Figure Description: The individual plasma concentrations over time will be presented for all participants, by treatment group. The figure will display values for all participants within each treatment group on a single page. Straight lines will connect the values for each participant.

For each figure, the X axis will be the actual timepoint. The Y axis will be the concentration, in units.

X axis title: Actual Timepoint (Hours) Y axis title: Concentration (units)

Abbreviations: PK= pharmacokinetic(s)

Data Source: Listing 16.2.6.1-1

#### **Programming Notes:**



Bellus Health Protocol 220254 (BUS-P1-11)

# Figure 14.2-18.2 Overlay of Individual Plasma Concentrations of Camlipixant – Linear Scale (PK Concentration Population) – Part 2

Plots of overlay individual plasma concentrations over time for all participants, by treatment group.

Figure Description: The individual plasma concentrations over time will be presented for all participant, by treatment group. The figure will display values for all participants within each treatment group on a single page. Straight lines will connect the values for each participant.

For each figure, the X axis will be the actual timepoint. The Y axis will be the concentration, in units.

X axis title: Actual Timepoint (Hours) Y axis title: Concentration (units)

Abbreviations: PK= pharmacokinetic(s)

Data Source: Listing 16.2.6.1-2

#### **Programming Notes:**



Bellus Health Protocol 220254 (BUS-P1-11)

# Figure 14.2-19.1 Overlay of Individual Plasma Concentrations of Camlipixant – Semi-Log Scale (PK Concentration Population) - Part 1

Plots of overlay individual plasma concentrations (log scale) over time for all participants, by treatment group.

Figure Description: The individual plasma concentrations (log scale) over time will be presented for all participant, by treatment group. The figure will display values for all participant within each treatment group on a single page. Straight lines will connect the values for each participant.

For each figure, the X axis will be the actual timepoint. The Y axis will be the concentration, in units.

X axis title: Actual Timepoint (Hours) Y axis title: Concentration (units)

Abbreviations: PK= pharmacokinetic(s)

Data Source: Listing 16.2.6.1-1

#### Programming Notes:



Bellus Health Protocol 220254 (BUS-P1-11)

# Figure 14.2-19.2 Overlay of Individual Plasma Concentrations of Camlipixant – Semi-Log Scale (PK Concentration Population) – Part 2

Plots of overlay individual plasma concentrations (log scale) over time for all participants, by treatment group.

Figure Description: The individual plasma concentrations (log scale) over time will be presented for all participant, by treatment group. The figure will display values for all participants within each treatment group on a single page. Straight lines will connect the values for each participant.

For each figure, the X axis will be the actual timepoint. The Y axis will be the concentration, in units.

X axis title: Actual Timepoint (Hours) Y axis title: Concentration (units)

Abbreviations: PK= pharmacokinetic(s)

Data Source: Listing 16.2.6.1-2

#### Programming Notes:

Bellus Health Protocol 220254 (BUS-P1-11)

# 3. Listings



Bellus Health Protocol 220254 (BUS-P1-11)

# Listing 16.1.9-1 COLL Output: Assessment of Rifampin Effect: DDI by ANOVA (PK Parameter Population) - Part 1

outputs related to the Assessment of Rifampin Effect: DDI by ANOVA will be placed here.

Abbreviations: DDI=Drug-drug interaction; ANOVA=Analysis of variance

26-Oct-2023 (Final 1.0) 



Bellus Health Protocol 220254 (BUS-P1-11)

# Listing 16.1.9-2 COLO Output: Assessment of Rabeprazole Effect: DDI by ANOVA (PK Parameter Population) - Part 2

outputs related to the Assessment of Rabeprazole Effect: DDI by ANOVA will be placed here.

Abbreviations: DDI=Drug-drug interaction; ANOVA=Analysis of variance

26-Oct-2023 (Final 1.0) 



Bellus Health Protocol 220254 (BUS-P1-11)

# Listing 16.1.9-3 Output: Non-Parametric Assessment of Rifampin Effect (PK Parameter Population) - Part 1

outputs related to the Non-Parametric Assessment of Rifampin Effect will be placed here.

Abbreviations:

26-Oct-2023 (Final 1.0) 



Bellus Health Protocol 220254 (BUS-P1-11)

# Listing 16.1.9-4 COLE Output: Non-Parametric Assessment of Rabeprazole Effect (PK Parameter Population) - Part 2

outputs related to the Non-Parametric Assessment of Rabeprazole Effect will be placed here.

Abbreviations:

26-Oct-2023 (Final 1.0) 



Bellus Health Protocol 220254 (BUS-P1-11)

# **Listing 16.2.1.1-1 Subject Enrollment (Safety Population) - Part 1**

| Subject<br>Number | Date / Time<br>ICF Signed | ICF Version Date /<br>Version Number | Protocol<br>Version<br>Number | Did the Subject Reconsent? /<br>If Yes, Date / Time of<br>Reconsent | ICF Version<br>Number at Time<br>of Reconsent | Protocol Version<br>Number at Time<br>of Reconsent | Was there a new<br>addendum to the ICF? /<br>If Yes, Date / Time<br>Addendum Signed | Addendum<br>Version Date /<br>Version Number |
|---|---|---|---|---|---|---|---|---|
| xxxxx | ddmmmyyyy /<br>hh:mm | ddmmmyyyy / xx | xx | Yes /<br>ddmmmyyyy / hh:mm | xx | xx | Yes /<br>ddmmmyyyy / hh:mm | ddmmmyyyy / xx |

Abbreviations: ICF=Informed consent form

# Programming Notes:

1) Sort by subject number

26-Oct-2023 (Final 1.0) 



Bellus Health Protocol 220254 (BUS-P1-11)

# **Listing 16.2.1.1-2 Subject Enrollment (Safety Population) - Part 2**

| Subject<br>Number | Date / Time<br>ICF Signed | ICF Version Date /<br>Version Number | Protocol<br>Version<br>Number | Did the Subject Reconsent? /<br>If Yes, Date / Time of<br>Reconsent | ICF Version<br>Number at Time<br>of Reconsent | Protocol Version<br>Number at Time<br>of Reconsent | Was there a new<br>addendum to the ICF? /<br>If Yes, Date / Time<br>Addendum Signed | Addendum<br>Version Date /<br>Version Number |
|---|---|---|---|---|---|---|---|---|
| xxxxx | ddmmmyyyy /<br>hh:mm | ddmmmyyyy / xx | XX | Yes /<br>ddmmmyyyy / hh:mm | xx | xx | Yes /<br>ddmmmyyyy / hh:mm | ddmmmyyyy / xx |

Abbreviations: ICF=Informed consent form

# Programming Notes:

1) Sort by subject number

26-Oct-2023 (Final 1.0) 



Bellus Health Protocol 220254 (BUS-P1-11)

# **Listing 16.2.1.2-1 Subject Disposition (Safety Population) - Part 1**

| Subject Number | Did the subject complete the study? / If No, Reason for Non-Completion | Date of Withdrawal or Completion /<br>Last Date of Participation or Contact | Other Recorded Information |
|---|---|---|---|
| xxxxx | No / xxxxxxxxxxxxxx | ddmmmyyyy / ddmmmyyyy | xxxxxxxxxxxx |
| xxxxx | Yes | ddmmmyyyy / ddmmmyyyy | N/A |

Abbreviations: N/A=Not applicable

# Programming Notes:

1) Sort by subject number.



Bellus Health Protocol 220254 (BUS-P1-11)

# **Listing 16.2.1.2-2 Subject Disposition (Safety Population) - Part 2**

| Subject Number | Did the subject complete the study? / If No, Reason for Non-Completion | Date of Withdrawal or Completion /<br>Last Date of Participation or Contact | Other Recorded Information |
|---|---|---|---|
| xxxxx | No / xxxxxxxxxxxxxx | ddmmmyyyy / ddmmmyyyy | xxxxxxxxxxxx |
| XXXXX | Yes | ddmmmyyyy / ddmmmyyyy | N/A |

Abbreviations: N/A=Not applicable

# Programming Notes:

1) Sort by subject number.

26-Oct-2023 (Final 1.0) 



Bellus Health Protocol 220254 (BUS-P1-11)

# **Listing 16.2.2.1-1 Protocol Deviations (Safety Population) - Part 1**

| Subject<br>Number | Study Day | Date of Deviation | Deviation Category | Deviation Classification <sup>[a]</sup> /<br>Importance <sup>[b]</sup> | Description of Deviation |
|---|---|---|---|---|---|
| xxxxx | Day x | ddmmmyyyy | xxxxxxxxxxx | Minor/<br>Non-important | xxxxxxxxxxx |
| ••• | | | | | |

# Programming Notes:

1) Sort by subject number and date of deviation.

26-Oct-2023 (Final 1.0) 

<sup>[</sup>a] Critical, major or minor [b] Important or non-important as per ICH E3 definition



Bellus Health Protocol 220254 (BUS-P1-11)

# **Listing 16.2.2.1-2 Protocol Deviations (Safety Population) - Part 2**

| Subject<br>Number | Study Day | Date of Deviation | Deviation Category | Deviation Classification <sup>[a]</sup> /<br>Importance <sup>[b]</sup> | Description of Deviation |
|---|---|---|---|---|---|
| xxxxx | Day x | ddmmmyyyy | xxxxxxxxxxx | Minor/<br>Non-important | xxxxxxxxxxx |
| ••• | | | | | |

# Programming Notes:

1) Sort by subject number and date of deviation.

26-Oct-2023 (Final 1.0) 

<sup>[</sup>a] Critical, major or minor [b] Important or non-important as per ICH E3 definition



Bellus Health Protocol 220254 (BUS-P1-11)

# Listing 16.2.3.1-1 Inclusion and Exclusion Criteria (Safety Population) - Part 1

| Subject Number | Study Day | Assessment Date | Did the subject meet all eligibility criteria? / If No, Criteria Not Met:<br>Category / Criterion Short Name / Reason Criterion not Respected |
|---|---|---|---|
| xxxxx | Screening<br>Day x | ddmmmyyyy<br>ddmmmyyyy | Yes<br>No/xxxxxxxx/xxxxxxxx/xxxxxxxx |

 26-Oct-2023 (Final 1.0)

Programming Notes:
1) Sort by subject number and assessment date.



Bellus Health Protocol 220254 (BUS-P1-11)

# Listing 16.2.3.1-2 Inclusion and Exclusion Criteria (Safety Population) - Part 2

| Subject Number | Study Day | Assessment Date | Did the subject meet all eligibility criteria? / If No, Criteria Not Met:<br>Category / Criterion Short Name / Reason Criterion not Respected |
|---|---|---|---|
| xxxxx | Screening<br>Day x | ddmmmyyyy<br>ddmmmyyyy | Yes<br>No/xxxxxxxx/xxxxxxxx/xxxxxxxxx |

Programming Notes:
1) Sort by subject number and assessment date.

 26-Oct-2023 (Final 1.0)



Bellus Health Protocol 220254 (BUS-P1-11)

# **Listing 16.2.3.2-1 Assignment to Analysis Populations - Part 1**

| Subject<br>Number | Date / Time of First Study<br>Drug Administration | Is the subject included in the safety population? / If No Reason | Is the subject included in the PK concentration population? / If No Reason | Is the subject included in the PK parameter population? / If No Reason | Is the subject included in the pharmacogenomic population? / If No Reason |
|---|---|---|---|---|---|
| xxxxx | ddmmmyyyy / hh:mm | Yes | Yes | Yes | No / xxxxxxxxxxxxx |



Bellus Health Protocol 220254 (BUS-P1-11)

# **Listing 16.2.3.2-2 Assignment to Analysis Populations - Part 2**

| Subject<br>Number | Date / Time of First Study<br>Drug Administration | Is the subject included in the safety population? / If No Reason | Is the subject included in the PK concentration population? / If No Reason | Is the subject included in the PK parameter population? / If No Reason | Is the subject included in the pharmacogenomic population? / If No Reason |
|---|---|---|---|---|---|
| xxxxx | ddmmmyyyy / hh:mm | Yes | Yes | Yes | No / xxxxxxxxxxxxx |



Bellus Health Protocol 220254 (BUS-P1-11)

# **Listing 16.2.4.1-1 Demographics (Safety Population) - Part 1**

| Subject<br>Number | Age<br>(years) <sup>[a]</sup> | Sex | If female, is subject of childbearing potential? | If Female of Non-Childbearing Potential,<br>Reason for Non-Childbearing Potential | Ethnicity | Race |
|---|---|---|---|---|---|---|
| xxxxx | xx | Female | No | Post-Menopause | Not Hispanic or Latino | Am Indian |

Abbreviations: Am Indian=American Indian or Alaskan native; Black=Black or African American; Hawaiian=Native Hawaiian or other pacific islander [a] Age at the time of informed consent

### Programming Notes:

- Sort by subject number.
   Refer to footnotes for additional instructions.

26-Oct-2023 (Final 1.0) 



Bellus Health Protocol 220254 (BUS-P1-11)

# **Listing 16.2.4.1-2 Demographics (Safety Population) - Part 2**

| Subject<br>Number | Age<br>(years) <sup>[a]</sup> | Sex | If female, is subject of childbearing potential? | If Female of Non-Childbearing Potential,<br>Reason for Non-Childbearing Potential | Ethnicity | Race |
|---|---|---|---|---|---|---|
| xxxxx | xx | Female | No | Post-Menopause | Not Hispanic or Latino | Am Indian |
| ••• | | | | | | |

Abbreviations: Am Indian=American Indian or Alaskan native; Black=Black or African American; Hawaiian=Native Hawaiian or other pacific islander [b] Age at the time of informed consent

### Programming Notes:

- Sort by subject number.
   Refer to footnotes for additional instructions.

26-Oct-2023 (Final 1.0) 


Bellus Health Protocol 220254 (BUS-P1-11)

# **Listing 16.2.4.2-1 Body Measurements (Safety Population) - Part 1**

| Subject Number | Was the assessment performed? / If No, Reason | Date / Time of Assessment | Height (cm) | Weight (kg) | BMI (kg/m²) |
|---|---|---|---|---|---|
| xxxxx | Yes | ddmmmyyyy / hh:mm | xxxx | xxxx | XXXX |

Abbreviations: BMI=Body mass index

# Programming Notes:

- 1) Sort by subject number.
- 2) Refer to footnotes for additional instructions.

26-Oct-2023 (Final 1.0) 



Bellus Health Protocol 220254 (BUS-P1-11)

# Listing 16.2.4.2-2 Body Measurements (Safety Population) - Part 2

| Subject Number | Was the assessment performed? / If No, Reason | Date / Time of Assessment | Height (cm) | Weight (kg) | BMI (kg/m²) |
|---|---|---|---|---|---|
| xxxxx | Yes | ddmmmyyyy / hh:mm | xxxx | xxxx | xxxx |

Abbreviations: BMI=Body mass index

- Programming Notes:
  1) Sort by subject number.
- 2) Refer to footnotes for additional instructions.

26-Oct-2023 (Final 1.0) 



Bellus Health Protocol 220254 (BUS-P1-11)

## **Listing 16.2.4.3-1 Medical History (Safety Population) - Part 1**

| Subject<br>Number | Collection<br>Date | Medical<br>History<br>ID | | MedDRA® System Organ Class / MedDRA Preferred Term | Start Date /<br>End Date | Is the subject taking any medication related to this condition? |
|---|---|---|---|---|---|---|
| xxxxx | ddmmmyyyy | x | TERM 1 | SOC 1 /<br>PT 1 | ddmmmyyyy /<br>ddmmmyyyy | No |
| xxxxx | ddmmmyyyy | X | TERM 2 | SOC 1 /<br>PT 1 | ddmmmyyyy /<br>ONGOING | Yes |

Abbreviations: ID= identifier; MedDRA= Medical Dictionary for Regulatory Activities; PT= preferred term; SOC= system organ class Note: Medical history terms were coded using MedDRA version X.X

#### **Programming Notes:**

- 1) Sort by subject number, start date, end date, SOC, and PT.
- 2) Present SOC and term in uppercase; present PT in "propcase".
- 3) If finding is ongoing, replace end date with "ONGOING" (in uppercase).
- 4) For incomplete date display, refer to CDISC SDTM Implementation Guide according to ISO 8601 format.
- 5) Add abbreviations used in the table to the footnotes.
  - a. MedDRA SOCs: Card=Cardiac disorders; Eye=Eye disorders; Gastr=Gastrointestinal disorders; Genrl=General disorders and administration site conditions; Infec=Infections and infestations; Inj&P=Injury, poisoning and procedural complications; Inv=Investigations; Musc=Musculoskeletal and connective tissue disorders; Nerv=Nervous system disorders; Psych=Psychiatric disorders; Resp=Respiratory, thoracic and mediastinal disorders; Skin=Skin and subcutaneous tissue disorders; Vasc=Vascular disorders
- 6) In the footnote, replace "X.X" with the actual MedDRA version used in the study



Bellus Health Protocol 220254 (BUS-P1-11)

### Listing 16.2.4.3-2 Medical History (Safety Population) - Part 2

| Subject<br>Number | Collection<br>Date | Medical<br>History<br>ID | Medical History Term | MedDRA® System Organ Class /<br>MedDRA Preferred Term | Start Date / End Date | Is the subject taking any medication related to this condition? |
|---|---|---|---|---|---|---|
| xxxxx | ddmmmyyyy | x | TERM 1 | SOC 1 /<br>PT 1 | ddmmmyyyy /<br>ddmmmyyyy | No |
| xxxxx | ddmmmyyyy | x | TERM 2 | SOC 1 /<br>PT 1 | ddmmmyyyy /<br>ONGOING | Yes |

Abbreviations: ID= identifier; MedDRA= Medical Dictionary for Regulatory Activities; PT= preferred term; SOC= system organ class Note: Medical history terms were coded using MedDRA version X.X

#### **Programming Notes:**

- 1) Sort by subject number, start date, end date, SOC, and PT.
- 2) Present SOC and term in uppercase; present PT in "propcase".
- 3) If finding is ongoing, replace end date with "ONGOING" (in uppercase).
- 4) For incomplete date display, refer to CDISC SDTM Implementation Guide according to ISO 8601 format.
- 5) Add abbreviations used in the table to the footnotes.
  - a. MedDRA SOCs: Card=Cardiac disorders; Eye=Eye disorders; Gastr=Gastrointestinal disorders; Genrl=General disorders and administration site conditions; Infec=Infections and infestations; Inj&P=Injury, poisoning and procedural complications; Inv=Investigations; Musc=Musculoskeletal and connective tissue disorders; Nerv=Nervous system disorders; Psych=Psychiatric disorders; Resp=Respiratory, thoracic and mediastinal disorders; Skin=Skin and subcutaneous tissue disorders; Vasc=Vascular disorders
- 6) In the footnote, replace "X.X" with the actual MedDRA version used in the study



Bellus Health Protocol 220254 (BUS-P1-11)



26-Oct-2023 (Final 1.0) 



Bellus Health Protocol 220254 (BUS-P1-11)



26-Oct-2023 (Final 1.0) 



Bellus Health Protocol 220254 (BUS-P1-11)

## Listing 16.2.4.5-1 Prior and Concomitant Medications (Safety Population) - Part 1

| Subject<br>Number | Reported Name /<br>ATC Classification /<br>Preferred Name | Indication | Dose, Unit / Form | Frequency /<br>Route | Start Date / Time /<br>End Date / Time | Due to AE? /<br>If Yes, AE ID(s) /<br>Due to MH? /<br>If Yes, MH ID(s) | Prior or<br>Concomitant |
|---|---|---|---|---|---|---|---|
| xxxxx | Medication 1 /<br>ATC 1 /<br>Preferred Name 1 / | xxxxxxxxxx | 100 mg / Tablet | CC / Oral | ddmmmyyyy /<br>hh:mm /<br>ddmmmyyyy / hh:mm | Yes / 1 /No | Prior |

Abbreviations: AE=Adverse event; ATC=Anatomic therapeutic chemical; ID=Identifier; MH=Medical history; WHODrug=World Health Organization Global Drug Dictionary.

Note: Prior medications are defined as medications that start and stop prior to the first dose of study drug. All other medications will be defined as concomitant medications including those that start prior to the first dose of study drug and continue thereafter.

Medications were coded using WHODrug, version MMM YYYY.

#### **Programming Notes:**

- 1) Sort by subject number, start date / time, and end date / time.
- 2) If medication is ongoing, replace end date / time with "ONGOING" (in uppercase).
- 3) If start or end time is unknown, replace time with "UNKNOWN" (in uppercase).
- 4) In the footnote, replace "MMM YYYY" with the actual WHO DD version used in the study.
- 5) Add abbreviations used in the table to the footnotes.
  - a. BID=Bis in die (twice daily); TID=Ter in die (three times daily); QID=Quater in die (four times daily)



Bellus Health Protocol 220254 (BUS-P1-11)

## Listing 16.2.4.5-2 Prior and Concomitant Medications (Safety Population) - Part 2

| Subject<br>Number | Reported Name /<br>ATC Classification /<br>Preferred Name | Indication | Dose, Unit / Form | Frequency /<br>Route | Start Date / Time /<br>End Date / Time | Due to AE? /<br>If Yes, AE ID(s) /<br>Due to MH? /<br>If Yes, MH ID(s) | Prior or<br>Concomitant |
|---|---|---|---|---|---|---|---|
| xxxxx | Medication 1 /<br>ATC 1 /<br>Preferred Name 1 / | xxxxxxxxxx | 100 mg / Tablet | CC / Oral | ddmmmyyyy /<br>hh:mm /<br>ddmmmyyyy / hh:mm | Yes / 1 /No | Prior |

Abbreviations: AE=Adverse event; ATC=Anatomic therapeutic chemical; ID=Identifier; MH=Medical history; WHODrug=World Health Organization Global Drug Dictionary.

Note: Prior medications are defined as medications that start and stop prior to the first dose of study drug. All other medications will be defined as concomitant medications including those that start prior to the first dose of study drug and continue thereafter.

Medications were coded using WHODrug, version MMM YYYY.

#### **Programming Notes:**

- 1) Sort by subject number, start date / time, and end date / time.
- 2) If medication is ongoing, replace end date / time with "ONGOING" (in uppercase).
- 3) If start or end time is unknown, replace time with "UNKNOWN" (in uppercase).
- 4) In the footnote, replace "MMM YYYY" with the actual WHO DD version used in the study.
- 5) Add abbreviations used in the table to the footnotes.
  - a. BID=Bis in die (twice daily); TID=Ter in die (three times daily); QID=Quater in die (four times daily)



Bellus Health Protocol 220254 (BUS-P1-11)

# Listing 16.2.4.6-1 Urine Drug Screen (Safety Population) - Part 1

| Subject Number | Study Day | Was the sample collected? / If No, Reason | Date / Time of Collection | Result / If Positive, Test Name(s) |
|---|---|---|---|---|
| xxxxx | Screening<br>Day x | Yes<br>Yes | ddmmmyyyy / hh:mm<br>ddmmmyyyy / hh:mm | Negative<br>Positive / MDMA |

#### Abbreviations:

#### Programming Notes:

- 1) Sort by subject number, and visit.
- 2) Refer to footnotes for additional instructions.
- 3) Add abbreviations used in the table to the footnotes.
  - a. MDMA=3,4 methylenedioxymethamphetamine, PCP=Phencyclidine; THC=Tetrahydrocannabinol

26-Oct-2023 (Final 1.0) 



Bellus Health Protocol 220254 (BUS-P1-11)

# Listing 16.2.4.6-2 Urine Drug Screen (Safety Population) - Part 2

| Subject Number | Study Day | Was the sample collected? / If No, Reason | Date / Time of Collection | Result / If Positive, Test Name(s) |
|---|---|---|---|---|
| xxxxx | Screening<br>Day x | Yes<br>Yes | ddmmmyyyy / hh:mm<br>ddmmmyyyy / hh:mm | Negative<br>Positive / MDMA |

#### Abbreviations:

#### Programming Notes:

- 1) Sort by subject number, and visit.
- 2) Refer to footnotes for additional instructions.
- 3) Add abbreviations used in the table to the footnotes.
  - a. MDMA=3,4 methylenedioxymethamphetamine, PCP=Phencyclidine; THC=Tetrahydrocannabinol

26-Oct-2023 (Final 1.0) 



Bellus Health Protocol 220254 (BUS-P1-11)

# Listing 16.2.4.7-1 Alcohol Breath Test (Safety Population) - Part 1

| Subject Number | Study Day | Was the test performed? / If No, Reason | Date / Time of Collection | Result |
|---|---|---|---|---|
| xxxxx | Screening<br>Day x | Yes<br>Yes | ddmmmyyyy / hh:mm<br>ddmmmyyyy / hh:mm | Negative<br>Positive |

Programming Notes:
1) Sort by subject number, and visit.

 26-Oct-2023 (Final 1.0)



Bellus Health Protocol 220254 (BUS-P1-11)

# **Listing 16.2.4.7-2 Alcohol Breath Test (Safety Population) - Part 2**

| Subject Number | Study Day | Was the test performed? / If No, Reason | Date / Time of Collection | Result |
|---|---|---|---|---|
| xxxxx | Screening<br>Day x | Yes<br>Yes | ddmmmyyyy / hh:mm<br>ddmmmyyyy / hh:mm | Negative<br>Positive |

Programming Notes:
1) Sort by subject number, and visit.

 26-Oct-2023 (Final 1.0)



Bellus Health Protocol 220254 (BUS-P1-11)

# Listing 16.2.4.8-1 Urine Cotinine Test (Safety Population) - Part 1

| Subject Number | Study Day | Was the sample collected? /<br>If No, Reason | Date / Time of Collection | Result |
|---|---|---|---|---|
| xxxxx | Screening<br>Day x | Yes<br>Yes | ddmmmyyyy / hh:mm | Negative<br>Positive |

Abbreviations:

Programming Notes:

1) Sort by subject number, and visit.

26-Oct-2023 (Final 1.0) 



Bellus Health Protocol 220254 (BUS-P1-11)

# **Listing 16.2.4.8-2 Urine Cotinine Test (Safety Population) - Part 2**

| Subject Number | Study Day | Was the sample collected? /<br>If No, Reason | Date / Time of Collection | Result |
|---|---|---|---|---|
| xxxxx | Screening<br>Day x | Yes<br>Yes | ddmmmyyyy / hh:mm | Negative<br>Positive |

Abbreviations:

Programming Notes:

1) Sort by subject number, and visit.

26-Oct-2023 (Final 1.0) 



Bellus Health Protocol 220254 (BUS-P1-11)

# **Listing 16.2.4.9-1 Pregnancy Test (Safety Population) - Part 1**

| Subject Number | Study Day | Sample Matrix <sup>[a]</sup> | Was the sample collected? / If No, Reason | Date / Time of Collection | Result |
|---|---|---|---|---|---|
| xxxxx | Screening<br>Day x<br>Day x | Urine<br>Serum<br>Urine | Yes<br>Yes | ddmmmyyyy / hh:mm<br>ddmmmyyyy / hh:mm<br>ddmmmyyyy / hh:mm | Negative<br>Negative<br>Positive |

<sup>[</sup>a] Serum or urine

# Programming Notes:

- Sort by subject number, and visit.
   Include all visits.

26-Oct-2023 (Final 1.0) 



Bellus Health Protocol 220254 (BUS-P1-11)

# **Listing 16.2.4.9-2 Pregnancy Test (Safety Population) - Part 2**

| Subject Number | Study Day | Sample Matrix <sup>[a]</sup> | Was the sample collected? / If No, Reason | Date / Time of Collection | Result |
|---|---|---|---|---|---|
| xxxxx | Screening<br>Day x<br>Day x | Urine<br>Serum<br>Urine | Yes<br>Yes | ddmmmyyyy / hh:mm<br>ddmmmyyyy / hh:mm<br>ddmmmyyyy / hh:mm | Negative<br>Negative<br>Positive |

<sup>[</sup>a] Serum or urine

## Programming Notes:

- Sort by subject number, and visit.
   Include all visits.

26-Oct-2023 (Final 1.0) 



Bellus Health Protocol 220254 (BUS-P1-11)

# **Listing 16.2.4.10-1 Follicle Stimulating Hormone Test (Safety Population) - Part 1**

| Subject Number | Was the sample collected? / If No, Reason | Date / Time of Collection | Result (mIU/mL) | Normal Range |
|---|---|---|---|---|
| xxxxx | Yes | ddmmmyyyy / hh:mm | xxxx | xxx-xxx |

## Programming Notes:

1) Sort by subject number.

26-Oct-2023 (Final 1.0) 



Bellus Health Protocol 220254 (BUS-P1-11)

# **Listing 16.2.4.10-2 Follicle Stimulating Hormone Test (Safety Population) - Part 2**

| Subject Number | Was the sample collected? / If No, Reason | Date / Time of Collection | Result (mIU/mL) | Normal Range |
|---|---|---|---|---|
| xxxxx | Yes | ddmmmyyyy / hh:mm | xxxx | xxx-xxx |

## Programming Notes:

1) Sort by subject number.

26-Oct-2023 (Final 1.0) 



Bellus Health Protocol 220254 (BUS-P1-11)

# **Listing 16.2.4.11-1 Serology (Safety Population) - Part 1**

| Subject Number | Was the sample collected? / If No, Reason | Date / Time of Collection | Are there any clinically significant values? / If Yes, Clinically Significant Lab Analyte(s) | Corresponding AE ID(s) /<br>Corresponding MH ID(s) |
|---|---|---|---|---|
| xxxxx | Yes | ddmmmyyyy / hh:mm | Yes / HBsAg | N/A / 1 |

Abbreviations: AE=Adverse event; ID=Identifier; MH=Medical history

## Programming Notes:

- 1) Sort by subject number.
- 2) Add abbreviations used in the table to the footnotes:
  - a. HIV=Immunodeficiency virus; HCV=Hepatitis C virus; HBsAg= Hepatitis B virus surface antigen

26-Oct-2023 (Final 1.0) 



Bellus Health Protocol 220254 (BUS-P1-11)

# **Listing 16.2.4.11-2 Serology (Safety Population) - Part 2**

| Subject Number | Was the sample collected? / If No, Reason | Date / Time of Collection | Are there any clinically significant values? / If Yes, Clinically Significant Lab Analyte(s) | Corresponding AE ID(s) /<br>Corresponding MH ID(s) |
|---|---|---|---|---|
| xxxxx | Yes | ddmmmyyyy / hh:mm | Yes / HBsAg | N/A / 1 |

Abbreviations: AE=Adverse event; ID=Identifier; MH=Medical history

## Programming Notes:

- 1) Sort by subject number.
- 2) Add abbreviations used in the table to the footnotes:
  - a. HIV=Immunodeficiency virus; HCV= Hepatitis C virus; HBsAg= Hepatitis B virus surface antigen

26-Oct-2023 (Final 1.0) 



Bellus Health Protocol 220254 (BUS-P1-11)

# Listing 16.2.4.12-1 COVID-19 Test (Safety Population) - Part 1

| Subject<br>Number | Study Day | Was the test performed? / If No, Reason | Date / Time of Collection | Method | Result |
|---|---|---|---|---|---|
| xxxxx | Day x | Yes | ddmmmyyyy / hh:mm | PCR | Negative |

Abbreviations: COVID-19=Coronavirus 2019

## Programming Notes:

- 1) Sort by subject number, and visit.
- 2) Add abbreviations used in the table to the footnotes:
  - a. PCR=Polymerase chain reaction

26-Oct-2023 (Final 1.0) 



Bellus Health Protocol 220254 (BUS-P1-11)

# Listing 16.2.4.12-2 COVID-19 Test (Safety Population) - Part 2

| Subject<br>Number | Study Day | Was the test performed? / If No, Reason | Date / Time of Collection | Method | Result |
|---|---|---|---|---|---|
| xxxxx | Day x | Yes | ddmmmyyyy / hh:mm | PCR | Negative |

Abbreviations: COVID-19=Coronavirus 2019

## Programming Notes:

- 1) Sort by subject number, and visit.
- 2) Add abbreviations used in the table to the footnotes:
  - a. PCR=Polymerase chain reaction

26-Oct-2023 (Final 1.0) 



Bellus Health Protocol 220254 (BUS-P1-11)

# **Listing 16.2.5.1-1 Study Drug Administration (Safety Population) - Part 1**

| Subject<br>Number | Study Day | Was the study drug administered? / If No, Reason | Administration Date / Time | Treatment Name | Planned Dose (Unit) / Was the planned dose administered? / Dose Administered (Unit) |
|---|---|---|---|---|---|
| xxxxx | Day x | Yes | ddmmmyyyy / hh:mm | Camlipixant | xx (xx) / Yes / xx (xx) |

Note: Treatment sequence: camlipixant 50 mg SD on Day 1, rifampin col mg col from Day 4 to Day 10, rifampin col mg col from Day 11 to 12 with co-administration of camlipixant 50 mg SD on Day 11.

## Programming Notes:

1) Sort by subject number, and visit.

26-Oct-2023 (Final 1.0) 



Bellus Health Protocol 220254 (BUS-P1-11)

## Listing 16.2.5.1-2 Study Drug Administration (Safety Population) - Part 2

| Subject<br>Number | Study Day | Was the study drug administered? / If No, Reason | Administration Date / Time | Treatment Name | Planned Dose (Unit) / Was the planned dose administered? / Dose Administered (Unit) |
|---|---|---|---|---|---|
| xxxxx | Day x | Yes | ddmmmyyyy / hh:mm | Camlipixant | xx (xx) / Yes / xx (xx) |

Note: Treatment sequence: camlipixant 50 mg SD on Day 1, rabeprazole comg mg from Day 4 to Day 9, rabeprazole mg mg from Day 10 to 11 with coadministration of camlipixant 50 mg SD on Day 10.

# Programming Notes:

1) Sort by subject number, and visit.



Bellus Health Protocol 220254 (BUS-P1-11)

## Listing 16.2.6.1-1 Plasma PK Concentrations (PK Concentration Population) - Part 1

| Analyte | Subject<br>Number | Study<br>Day | Nominal Timepoint<br>(Hours) | Date / Time of Study Drug Administration /<br>Date / Time of Sample Collection | Actual Time <sup>[a]</sup> (hours) | Concentration (unit) | Excluded? /<br>If Yes, Reason |
|---|---|---|---|---|---|---|---|
| Camlipixant | xxxxx | Day 1 | Pre-Dose | ddmmmyyyy / hh:mm /<br>ddmmmyyyy / hh:mm | 0.000 | xx xx | Yes / Inconclusive |

#### Abbreviations:

#### Programming Notes:

- 1) add pre-dose concentrations of Rifampin also in this listing.
- 2) Sort by analyte, subject number, day, and timepoint.
- 3) Include all scheduled visits/timepoints.
  - a. If a sample is not collected at a scheduled visit/timepoint, collection data is presented as "-".

26-Oct-2023 (Final 1.0) 

<sup>[</sup>a] Actual time is the difference (in hours) from study drug administration to sample collection.



Bellus Health Protocol 220254 (BUS-P1-11)

## Listing 16.2.6.1-2 Plasma PK Concentrations (PK Concentration Population) - Part 2

| Analyte | Subject<br>Number | Study<br>Day | Nominal Timepoint<br>(Hours) | Date / Time of Study Drug Administration /<br>Date / Time of Sample Collection | Actual Time <sup>[a]</sup><br>(hours) | Concentration (unit) | Excluded? /<br>If Yes, Reason |
|---|---|---|---|---|---|---|---|
| Camlipixant | xxxxx | Day 1 | Pre-Dose | ddmmmyyyy / hh:mm /<br>ddmmmyyyy / hh:mm | 0.000 | xx xx | Yes / Inconclusive |

#### Abbreviations:

#### Programming Notes:

- 1) add pre-dose concentrations of Rabeprazole also in this listing.
- 2) Sort by analyte, subject number, day, and timepoint.
- 3) Include all scheduled visits/timepoints.
  - a. If a sample is not collected at a scheduled visit/timepoint, collection data is presented as "-".

26-Oct-2023 (Final 1.0) 

<sup>[</sup>a] Actual time is the difference (in hours) from study drug administration to sample collection.



Bellus Health Protocol 220254 (BUS-P1-11)

Listing 16.2.6.2-1 Plasma PK Parameters of (PK Parameter Population) - Part 1

| Analyte | Subject<br>Number | Study<br>Day | Parameter | Result | Unit | Excluded? /<br>If Yes, Reason |
|---|---|---|---|---|---|---|
| G tit | | D 1 | ATIC | 27/4 | | XX /XX 11 |
| Camlipixant | XXXXX | Day 1 | $\mathrm{AUC}_{0	ext{-t}}$ | N/A | XX | Yes / Not estimable |
| | | | $\mathrm{AUC}_{0	ext{-}\mathrm{inf}}$ | XXXXXXX | XX | No |
| | | | Cl/F | xxxxxxx | XX | No |
| | | | $C_{max}$ | xxxxxxx | XX | No |
| | | | $K_{\mathrm{el}}$ | xxxxxxx | XX | No |
| | | | Residual area | N/A | XX | Yes / Not estimable |
| | | | $T_{max}$ | xxxxxxx | XX | N |
| | | | $T_{1/2 \text{ el}}$ | xxxxxxx | XX | No |
| | | | $V_z/F$ | xxxxxxx | XX | No |
| | | | ••• | | | |
| | ••• | | | | | |

Abbreviations: PK=Pharmacokinetic(s)

## Programming Notes:

- 1) Sort by analyte, subject number and day.
- 2) Add abbreviations used in the table to the footnotes.

26-Oct-2023 (Final 1.0) 



Bellus Health Protocol 220254 (BUS-P1-11)

# Listing 16.2.6.2-2 Plasma PK Parameters of (PK Parameter Population) - Part 2

| Analyte | Subject<br>Number | Study<br>Day | Parameter | Result | Unit | Excluded? /<br>If Yes, Reason |
|---|---|---|---|---|---|---|
| | | | | **/. | | |
| Camlipixant | XXXXX | Day 1 | $\mathrm{AUC}_{0	ext{-t}}$ | N/A | XX | Yes / Not estimable |
| | | | $\mathrm{AUC}_{0	ext{-inf}}$ | XXXXXXX | XX | No |
| | | | Cl/F | xxxxxxx | XX | No |
| | | | $C_{max}$ | xxxxxxx | XX | No |
| | | | $K_{\mathrm{el}}$ | xxxxxxx | XX | No |
| | | | Residual area | N/A | XX | Yes / Not estimable |
| | | | $T_{max}$ | xxxxxxx | XX | N |
| | | | $T_{1/2 \; el}$ | xxxxxxx | XX | No |
| | | | $V_z/F$ | xxxxxxx | XX | No |

Abbreviations: PK=Pharmacokinetic(s)

## Programming Notes:

- 1) Sort by analyte, subject number and day.
- 2) Add abbreviations used in the table to the footnotes.



Bellus Health Protocol 220254 (BUS-P1-11)

## **Listing 16.2.7.1-1 Non-TEAEs (Safety Population) - Part 1**

| Subject<br>Number | MedDRA® System Organ Class /<br>MedDRA Preferred Term /<br>AE Term | Onset Date / Time / Resolution Date / Time | Severity /<br>Relationship | Action Ta Study Drug | ken Treatment | Outcome | Subject<br>Discontinued/<br>serious/AEMI | Other Recorded<br>Information |
|---|---|---|---|---|---|---|---|---|
| xxxxx | SOC 1 /<br>PT 1 /<br>TERM 1 | ddmmmyyyy / hh:mm / | xxx/xxx | Dose Not Changed | xxx | Recovered/<br>Resolved | No / No / No | xxxxxxxxxxxx |

Abbreviations: AE=Adverse event; AEMI=Adverse events of medical interest; ID=Identifier; MedDRA=Medical Dictionary for Regulatory Activities; TEAE=Treatment-emergent adverse event;

Note: AE terms were coded using MedDRA version X.X.

#### **Programming Notes:**

- 1) Sort by subject number, onset date / time, SOC, and PT.
- 2) Present SOC and term in uppercase; present PT in "propease".
- 3) Use coling "/~n" between terms to generate break lines between SOC, PT, and description.
- 4) Use gran coding "/~n" to generate a break line between dates and between Severity and Relationship.
- 5) If needed, hardcode outcome and actions to introduce break line (~n) between answer elements.
- 6) If AE is ongoing, replace resolution date / time with "ONGOING" (in uppercase).
- 7) If onset or resolution time is unknown, replace time with "UNKNOWN" (in uppercase)
- 8) For incomplete date display, refer to CDISC SDTM Implementation Guide according to ISO 8601 format.
- 9) Add abbreviations used in the table to the footnotes.
  - a. MedDRA SOCs: Card=Cardiac disorders; Eye=Eye disorders; Gastr=Gastrointestinal disorders; Genrl=General disorders and administration site conditions; Infec=Infections and infestations; Inj&P=Injury, poisoning and procedural complications; Inv=Investigations; Musc=Musculoskeletal and connective tissue disorders; Nerv=Nervous system disorders; Psych=Psychiatric disorders; Resp=Respiratory, thoracic and mediastinal disorders; Skin=Skin and subcutaneous tissue disorders; Vasc=Vascular disorders



Bellus Health Protocol 220254 (BUS-P1-11)

## **Listing 16.2.7.1-2 Non-TEAEs (Safety Population) - Part 2**

| Subject<br>Number | MedDRA® System Organ Class /<br>MedDRA Preferred Term /<br>AE Term | Onset Date / Time / Resolution Date / Time | Severity /<br>Relationship | Action Ta<br>Study Drug | ken Treatment | Outcome | Subject<br>Discontinued/<br>serious/AEMI | Other Recorded<br>Information |
|---|---|---|---|---|---|---|---|---|
| xxxxx | SOC 1 /<br>PT 1 /<br>TERM 1 | ddmmmyyyy / hh:mm / | xxx/xxx | Dose Not Changed | xxx | Recovered/<br>Resolved | No / No / No | xxxxxxxxxxxx |
| ••• | | | | | | | | |

Abbreviations: AE=Adverse event; AEMI=Adverse events of medical interest; ID=Identifier; MedDRA=Medical Dictionary for Regulatory Activities; TEAE=Treatment-emergent adverse event;

Note: AE terms were coded using MedDRA version X.X.

#### **Programming Notes:**

- 1) Sort by subject number, onset date / time, SOC, and PT.
- 2) Present SOC and term in uppercase; present PT in "propease".
- 3) Use coling "/~n" between terms to generate break lines between SOC, PT, and description.
- 4) Use gran coding "/~n" to generate a break line between dates and between Severity and Relationship.
- 5) If needed, hardcode outcome and actions to introduce break line (~n) between answer elements.
- 6) If AE is ongoing, replace resolution date / time with "ONGOING" (in uppercase).
- 7) If onset or resolution time is unknown, replace time with "UNKNOWN" (in uppercase)
- 8) For incomplete date display, refer to CDISC SDTM Implementation Guide according to ISO 8601 format.
- 9) Add abbreviations used in the table to the footnotes.
  - a. MedDRA SOCs: Card=Cardiac disorders; Eye=Eye disorders; Gastr=Gastrointestinal disorders; Genrl=General disorders and administration site conditions; Infec=Infections and infestations; Inj&P=Injury, poisoning and procedural complications; Inv=Investigations; Musc=Musculoskeletal and connective tissue disorders; Nerv=Nervous system disorders; Psych=Psychiatric disorders; Resp=Respiratory, thoracic and mediastinal disorders; Skin=Skin and subcutaneous tissue disorders; Vasc=Vascular disorders



Bellus Health Protocol 220254 (BUS-P1-11)

## **Listing 16.2.7.2-1 TEAEs (Safety Population) - Part 1**

| Subject<br>Number | Treatment<br>Phase | MedDRA® System Organ Class /<br>MedDRA Preferred Term /<br>AE Term | Onset Date / Time / Resolution Date / Time | Severity /<br>Relationship:<br>to Camlipixant /<br>to Rifampin | Actions Taken:<br>with Camlipixant /<br>with Rifampin /<br>Other | Outcome | Did the AE cause the subject to be discontinued from the study? / Is the AE serious? / Is this an AEMI? | Other Recorded<br>Information |
|---|---|---|---|---|---|---|---|---|
| xxxxx | Rifampin | SOC 1 /<br>PT 1 /<br>TERM 1 | ddmmmyyyy / hh:mm /<br>ddmmmyyyy / hh:mm | Mild /<br>Not Related /<br>Possible | Dose Not Changed /<br>Dose Not Changed /<br>None | Recovered/<br>Resolved | No / No / No | xxxxxxxxxxxx |

Abbreviations: AE=Adverse event; AEMI=Adverse events of medical interest; ID=Identifier; MedDRA=Medical Dictionary for Regulatory Activities; TEAE=Treatment-emergent adverse event;

Note: Treatment sequence: camlipixant 50 mg SD on Day 1, rifampin get mg get from Day 4 to Day 10, rifampin get mg get from Day 11 to 12 with co-administration of camlipixant 50 mg SD on Day 11.

AE terms were coded using MedDRA version X.X.

#### **Programming Notes:**

- 1) Sort by subject number, onset date / time, SOC, and PT.
- 2) Present SOC and term in uppercase; present PT in "propcase".
- 3) Use coding "/~n" between terms to generate break lines between SOC, PT, and description.
- 4) Use coding "/~n" to generate a break line between dates and between Severity and Relationship.
- 5) If needed, hardcode outcome and actions to introduce break line (~n) between answer elements.
- 6) If AE is ongoing, replace resolution date / time with "ONGOING" (in uppercase).
- 7) If onset or resolution time is unknown, replace time with "UNKNOWN" (in uppercase)
- 8) For incomplete date display, refer to CDISC SDTM Implementation Guide according to ISO 8601 format.
- 9) Add abbreviations used in the table to the footnotes.
  - a. MedDRA SOCs: Card=Cardiac disorders; Eye=Eye disorders; Gastr=Gastrointestinal disorders; Genrl=General disorders and administration site conditions; Infec=Infections and infestations; Inj&P=Injury, poisoning and procedural complications; Inv=Investigations; Musc=Musculoskeletal and connective tissue disorders; Nerv=Nervous system disorders; Psych=Psychiatric disorders; Resp=Respiratory, thoracic and mediastinal disorders; Skin=Skin and subcutaneous tissue disorders; Vasc=Vascular disorders



Bellus Health Protocol 220254 (BUS-P1-11)

#### Listing 16.2.7.2-2 TEAEs (Safety Population) - Part 2

| Subject<br>Number | Treatment<br>Phase | MedDRA® System Organ Class /<br>MedDRA Preferred Term /<br>AE Term | Onset Date / Time / Resolution Date / Time | Severity /<br>Relationship:<br>to Camlipixant /<br>to Rabeprazole | Actions Taken:<br>with Camlipixant /<br>with Rabeprazole /<br>Other | Outcome | Did the AE cause the subject to be discontinued from the study? / Is the AE serious? / Is this an AEMI? | Other Recorded<br>Information |
|---|---|---|---|---|---|---|---|---|
| xxxxx | Rabeprazole | SOC 1 /<br>PT 1 /<br>TERM 1 | ddmmmyyyy /<br>hh:mm /<br>ddmmmyyyy /<br>hh:mm | Mild /<br>Not Related /<br>Possible | Dose Not Changed /<br>Dose Not Changed /<br>None | Recovered/<br>Resolved | No / No / No | xxxxxxxxxxxx |

Abbreviations: AE=Adverse event; AEMI=Adverse events of medical interest; ID=Identifier; MedDRA=Medical Dictionary for Regulatory Activities; TEAE= Treatment-emergent adverse event;

Note: Treatment sequence: camlipixant 50 mg SD on Day 1, rabeprazole mg mg from Day 4 to Day 9, rabeprazole mg mg from Day 10 to 11 with coadministration of camlipixant 50 mg SD on Day 10.

AE terms were coded using MedDRA version X.X.

#### Programming Notes:

- 1) Sort by subject number, onset date / time, SOC, and PT.
- 2) Present SOC and term in uppercase; present PT in "propcase".
- 3) Use coding "/~n" between terms to generate break lines between SOC, PT, and description.
- 4) Use coding "/~n" to generate a break line between dates and between Severity and Relationship.
- 5) If needed, hardcode outcome and actions to introduce break line (~n) between answer elements.
- 6) If AE is ongoing, replace resolution date / time with "ONGOING" (in uppercase).
- 7) If onset or resolution time is unknown, replace time with "UNKNOWN" (in uppercase)
- 8) For incomplete date display, refer to CDISC SDTM Implementation Guide according to ISO 8601 format.
- 9) Add abbreviations used in the table to the footnotes.
  - a. MedDRA SOCs: Card=Cardiac disorders; Eye=Eye disorders; Gastr=Gastrointestinal disorders; Genrl=General disorders and administration site conditions; Infec=Infections and infestations; Inj&P=Injury, poisoning and procedural complications; Inv=Investigations; Musc=Musculoskeletal and connective tissue disorders; Nerv=Nervous system disorders; Psych=Psychiatric disorders; Resp=Respiratory, thoracic and mediastinal disorders; Skin=Skin and subcutaneous tissue disorders; Vasc=Vascular disorders



Bellus Health Protocol 220254 (BUS-P1-11)

#### Listing 16.2.7.3-1 Serious AEs (Safety Population) - Part 1

| Subject<br>Number | Treatment<br>Phase | MedDRA® System Organ Class /<br>MedDRA Preferred Term /<br>AE Term | Onset Date / Time /<br>Resolution Date / Time | Severity /<br>Relationship:<br>to Camlipixant /<br>to Rifampin | Actions Taken:<br>with Camlipixant /<br>with Rifampin /<br>Other | Outcome | Serious Reason |
|---|---|---|---|---|---|---|---|
| xxxxx | Camlipixant | SOC 1 /<br>PT 1 /<br>TERM 1 | ddmmmyyyy / hh:mm /<br>ddmmmyyyy / hh:mm | Mild /<br>Definite /<br>Not Related / | Dose Not Changed /<br>Drug Interrupted /<br>Hospitalization | Recovered/<br>Resolved | Life threatening |

Abbreviations: AE=Adverse event; MedDRA=Medical Dictionary for Regulatory Activities; TEAE=Treatment-emergent adverse event

Note: Treatment sequence: camlipixant 50 mg SD on Day 1, rifampin col mg col from Day 4 to Day 10, rifampin col mg ECI from Day 11 to 12 with co-administration of camlipixant 50 mg SD on Day 11.

AE terms were coded using MedDRA version X.X.

#### **Programming Notes:**

- 1) Sort by subject number, treatment, onset date / time, SOC, and PT.
- 2) Present SOC and term in uppercase; present PT in "propease".
- 3) Use coding "/~n" between terms to generate break lines between SOC, PT, and description.
- 4) Use coding "/~n" to generate a break line between dates and between Severity and Relationship.
- 5) If needed, hardcode outcome and actions to introduce break line (~n) between answer elements.
- 6) If AE is ongoing, replace resolution date / time with "ONGOING" (in uppercase).
- 7) If onset or resolution time is unknown, replace time with "UNKNOWN" (in uppercase).
- 8) For incomplete date display, refer to CDISC SDTM Implementation Guide according to ISO 8601 format.
- 9) Add abbreviations used in the table to the footnotes.
  - a. MedDRA SOCs: Card=Cardiac disorders; Eye=Eye disorders; Gastr=Gastrointestinal disorders; Genrl=General disorders and administration site conditions; Infec=Infections and infestations; Inj&P=Injury, poisoning and procedural complications; Inv=Investigations; Musc=Musculoskeletal and connective tissue disorders; Nerv=Nervous system disorders; Psych=Psychiatric disorders; Resp=Respiratory, thoracic and mediastinal disorders; Skin=Skin and subcutaneous tissue disorders; Vasc=Vascular disorders



Bellus Health Protocol 220254 (BUS-P1-11)

## **Listing 16.2.7.3-2 Serious AEs (Safety Population) - Part 2**

| Subject<br>Number | Treatment<br>Phase | MedDRA® System Organ Class /<br>MedDRA Preferred Term /<br>AE Term | Onset Date / Time /<br>Resolution Date / Time | Severity / Relationship: to Camlipixant / to Rabeprazole | Actions Taken:<br>with Camlipixant /<br>with Rabeprazole /<br>Other | Outcome | Serious Reason |
|---|---|---|---|---|---|---|---|
| xxxxx | Camlipixant | SOC 1 /<br>PT 1 /<br>TERM 1 | ddmmmyyyy / hh:mm /<br>ddmmmyyyy / hh:mm | Mild /<br>Definite /<br>Not Related / | Dose Not Changed /<br>Drug Interrupted /<br>Hospitalization | Recovered/<br>Resolved | Life threatening |

Abbreviations: AE=Adverse event; MedDRA=Medical Dictionary for Regulatory Activities; TEAE=Treatment-emergent adverse event

Note: Treatment sequence: camlipixant 50 mg SD on Day 1, rabeprazole compared from Day 4 to Day 9, rabeprazole compared from Day 10 to 11 with co-administration of camlipixant 50 mg SD on Day 10.

AE terms were coded using MedDRA version X.X.

#### Programming Notes:

- 1) Sort by subject number, treatment, onset date / time, SOC, and PT.
- 2) Present SOC and term in uppercase; present PT in "propease".
- 3) Use color coding "/~n" between terms to generate break lines between SOC, PT, and description.
- 4) Use coding "/~n" to generate a break line between dates and between Severity and Relationship.
- 5) If needed, hardcode outcome and actions to introduce break line (~n) between answer elements.
- 6) If AE is ongoing, replace resolution date / time with "ONGOING" (in uppercase).
- 7) If onset or resolution time is unknown, replace time with "UNKNOWN" (in uppercase).
- 8) For incomplete date display, refer to CDISC SDTM Implementation Guide according to ISO 8601 format.
- 9) Add abbreviations used in the table to the footnotes.
  - a. MedDRA SOCs: Card=Cardiac disorders; Eye=Eye disorders; Gastr=Gastrointestinal disorders; Genrl=General disorders and administration site conditions; Infec=Infections and infestations; Inj&P=Injury, poisoning and procedural complications; Inv=Investigations; Musc=Musculoskeletal and connective tissue disorders; Nerv=Nervous system disorders; Psych=Psychiatric disorders; Resp=Respiratory, thoracic and mediastinal disorders; Skin=Skin and subcutaneous tissue disorders; Vasc=Vascular disorders



Bellus Health Protocol 220254 (BUS-P1-11)

## **Listing 16.2.7.4-1 AEMIs (Safety Population) - Part 1**

| Subject<br>Number | Treatment<br>Phase | MedDRA® System Organ Class /<br>MedDRA Preferred Term /<br>AE Term | Onset Date / Time /<br>Resolution Date / Time | Severity /<br>Relationship:<br>to Camlipixant /<br>to Rifampin | Actions Taken:<br>with Camlipixant /<br>with Rifampin /<br>Other | Outcome | Type of AEMI |
|---|---|---|---|---|---|---|---|
| xxxxx | Rifampin | SOC 1 /<br>PT 1 /<br>TERM 1 | ddmmmyyyy / hh:mm /<br>ddmmmyyyy / hh:mm | Mild /<br>Not Related /<br>Unlikely | Dose Not Changed /<br>Dose Not Changed /<br>None | Recovered/<br>Resolved | Oral Hypoesthesia |

...

Abbreviations: AE=Adverse event; AEMI=Adverse events of medical interest; MedDRA=Medical Dictionary for Regulatory Activities;

Note: Treatment sequence: camlipixant 50 mg SD on Day 1, rifampin get mg get from Day 4 to Day 10, rifampin equing from Day 11 to 12 with co-administration of camlipixant 50 mg SD on Day 11.

AE terms were coded using MedDRA version X.X.

#### **Programming Notes:**

- 1) Sort by subject number, treatment, onset date / time, SOC, and PT.
- 2) Present SOC and term in uppercase; present PT in "propcase".
- 3) Use coding "/~n" between terms to generate break lines between SOC, PT, and description.
- 4) Use coding "/~n" to generate a break line between dates and between Severity and Relationship.
- 5) If needed, hardcode outcome and actions to introduce break line (~n) between answer elements.
- 6) If AE is ongoing, replace resolution date / time with "ONGOING" (in uppercase).
- 7) If onset or resolution time is unknown, replace time with "UNKNOWN" (in uppercase).
- 8) For incomplete date display, refer to CDISC SDTM Implementation Guide according to ISO 8601 format.
- 9) Add abbreviations used in the table to the footnotes.
  - a. MedDRA SOCs: Card=Cardiac disorders; Eye=Eye disorders; Gastr=Gastrointestinal disorders; Genrl=General disorders and administration site conditions; Infec=Infections and infestations; Inj&P=Injury, poisoning and procedural complications; Inv=Investigations; Musc=Musculoskeletal and connective tissue disorders; Nerv=Nervous system disorders; Psych=Psychiatric disorders; Resp=Respiratory, thoracic and mediastinal disorders; Skin=Skin and subcutaneous tissue disorders; Vasc=Vascular disorders



Bellus Health Protocol 220254 (BUS-P1-11)

#### Listing 16.2.7.4-2 AEMIs (Safety Population) - Part 2

| Subject<br>Number | Treatment<br>Phase | MedDRA® System Organ Class /<br>MedDRA Preferred Term /<br>AE Term | Onset Date / Time /<br>Resolution Date / Time | Severity / Relationship: to Camlipixant / to Rabeprazole | Actions Taken:<br>with Camlipixant /<br>with Rabeprazole /<br>Other | Outcome | Type of AEMI |
|---|---|---|---|---|---|---|---|
| xxxxx | Rabeprazole | SOC 1 /<br>PT 1 /<br>TERM 1 | ddmmmyyyy / hh:mm /<br>ddmmmyyyy / hh:mm | Mild /<br>Not Related /<br>Unlikely / | Dose Not Changed /<br>Dose Not Changed /<br>None | Recovered/<br>Resolved | Oral Hypoesthesia |

Abbreviations: AE=Adverse event; AEMI=Adverse events of medical interest; MedDRA=Medical Dictionary for Regulatory Activities;

Note: Treatment sequence: camlipixant 50 mg SD on Day 1, rabeprazole rem mg from Day 4 to Day 9, rabeprazole rem mg from Day 10 to 11 with co-administration of camlipixant 50 mg SD on Day 10.

AE terms were coded using MedDRA version X.X.

#### **Programming Notes:**

- 1) Sort by subject number, treatment, onset date / time, SOC, and PT.
- 2) Present SOC and term in uppercase; present PT in "propcase".
- 3) Use coding "/~n" between terms to generate break lines between SOC, PT, and description.
- 4) Use coding "/~n" to generate a break line between dates and between Severity and Relationship.
- 5) If needed, hardcode outcome and actions to introduce break line (~n) between answer elements.
- 6) If AE is ongoing, replace resolution date / time with "ONGOING" (in uppercase).
- 7) If onset or resolution time is unknown, replace time with "UNKNOWN" (in uppercase).
- 8) For incomplete date display, refer to CDISC SDTM Implementation Guide according to ISO 8601 format.
- 9) Add abbreviations used in the table to the footnotes.
  - a. MedDRA SOCs: Card=Cardiac disorders; Eye=Eye disorders; Gastr=Gastrointestinal disorders; Genrl=General disorders and administration site conditions; Infec=Infections and infestations; Inj&P=Injury, poisoning and procedural complications; Inv=Investigations; Musc=Musculoskeletal and connective tissue disorders; Nerv=Nervous system disorders; Psych=Psychiatric disorders; Resp=Respiratory, thoracic and mediastinal disorders; Skin=Skin and subcutaneous tissue disorders; Vasc=Vascular disorders


Bellus Health Protocol 220254 (BUS-P1-11)



## Programming Notes:

- 1) Sort by subject number.
- 2) Add abbreviations used in the table to the footnotes:
  - a. PCR=Polymerase chain reaction

26-Oct-2023 (Final 1.0) 



Statistical Analysis Plan (Table/Figure/Listing Shells)

Bellus Health Protocol 220254 (BUS-P1-11)



## Programming Notes:

- 1) Sort by subject number.
- 2) Add abbreviations used in the table to the footnotes:
  - a. PCR=Polymerase chain reaction

26-Oct-2023 (Final 1.0) 



Bellus Health Protocol 220254 (BUS-P1-11)

# Listing 16.2.7.6-1 Oral Hypoesthesia, Oral Paresthesia AE Questionnaire (Safety Population) - Part 1

| Subject<br>Number | Was the assessment performed? / If No, Reason | AE<br>ID | What type of oral hypoesthesia/paresthesia has the participant experienced? | Are there other possible contributory factors to oral hypoesthesia/paresthesia? / If yes, specify |
|---|---|---|---|---|
| xxxxx | Yes | xx | Oral Hypoesthesia | Yes / xxxxxxxxxxxx |

Abbreviations: AE=Adverse event; ID=Identifier

Note: Treatment sequence: camlipixant 50 mg SD on Day 1, rifampin graph mg graph from Day 4 to Day 10, rifampin graph mg graph from Day 11 to 12 with co-administration of camlipixant 50 mg SD on Day 11.

## Programming Notes:

1) Sort by subject number.

26-Oct-2023 (Final 1.0) 



Bellus Health Protocol 220254 (BUS-P1-11)

# Listing 16.2.7.6-2 Oral Hypoesthesia, Oral Paresthesia AE Questionnaire (Safety Population) - Part 2

| Subject<br>Number | Was the assessment performed? / If No, Reason | AE<br>ID | What type of oral hypoesthesia/paresthesia has the participant experienced? | Are there other possible contributory factors to oral hypoesthesia/paresthesia? / If yes, specify |
|---|---|---|---|---|
| xxxxx | Yes | XX | Oral Hypoesthesia | Yes / xxxxxxxxxxxx |
| ••• | | | | |

Abbreviations: AE=Adverse event; ID=Identifier

Note: Treatment sequence: camlipixant 50 mg SD on Day 1, rabeprazole reg mg reg from Day 4 to Day 9, rabeprazole reg mg reg from Day 10 to 11 with coadministration of camlipixant 50 mg SD on Day 10.

## Programming Notes:

1) Sort by subject number.

C C

26-Oct-2023 (Final 1.0) 



Bellus Health Protocol 220254 (BUS-P1-11)

## Listing 16.2.8.1-1 Biochemistry (Safety Population) - Part 1

| Subject<br>Number | Study<br>Day | Was the sample collected? / If No, Reason | Date / Time of<br>Collection | Parameter (unit) | Actual<br>Value | Actual Change<br>from Baseline <sup>[a]</sup> | Normal Range<br>(LLN-ULN) | Flag <sup>[b]</sup> | Corresponding AE ID(s) /<br>Corresponding MH ID(s) |
|---|---|---|---|---|---|---|---|---|---|
| xxxxx | Day x <sup>[a]</sup> | Yes | ddmmmyyyy / hh:mm | xxxx (xx) | xxx.x | N/A | xxx.x-xxx.x | H, CS | N/A / 1 |

...

Abbreviations: AE=Adverse event; CS=Clinically significant; H=Above normal range (high); ID=Identifier; L=Below normal range (low); LLN=Lower limit of normal; MH=Medical history; N=Within normal range; NCS=Not clinically significant; ULN=Upper limit of normal

#### **Programming Notes:**

- 1) Include all visits.
- 2) Include all parameters in alphabetical order.
- 3) Add abbreviations used in the table to the footnotes.

26-Oct-2023 (Final 1.0) 

<sup>[</sup>a] Baseline value; baseline is defined as the last result (scheduled or unscheduled) obtained prior to study drug administration.

<sup>[</sup>b] H, L, or N; if abnormal (H or L), CS or NCS



Bellus Health Protocol 220254 (BUS-P1-11)

## **Listing 16.2.8.1-2 Biochemistry (Safety Population) - Part 2**

| Subject<br>Number | Study<br>Day | Was the sample collected? / If No, Reason | Date / Time of<br>Collection | Parameter (unit) | Actual<br>Value | Actual Change from Baseline <sup>[a]</sup> | Normal Range<br>(LLN-ULN) | Flag <sup>[b]</sup> | Corresponding AE ID(s) /<br>Corresponding MH ID(s) |
|---|---|---|---|---|---|---|---|---|---|
| xxxxx | Day x <sup>[a]</sup> | Yes | ddmmmyyyy / hh:mm | xxxx (xx) | xxx.x | N/A | xxx.x-xxx.x | H, CS | N/A / 1 |

Abbreviations: AE=Adverse event; CS=Clinically significant; H=Above normal range (high); ID=Identifier; L=Below normal range (low); LLN=Lower limit of normal; MH=Medical history; N=Within normal range; NCS=Not clinically significant; ULN=Upper limit of normal

### **Programming Notes:**

- 1) Include all visits.
- 2) Include all parameters in alphabetical order.
- 3) Add abbreviations used in the table to the footnotes.

26-Oct-2023 (Final 1.0) 

<sup>[</sup>a] Baseline value; baseline is defined as the last result (scheduled or unscheduled) obtained prior to study drug administration.

<sup>[</sup>b] H, L, or N; if abnormal (H or L), CS or NCS



Bellus Health Protocol 220254 (BUS-P1-11)

# Listing 16.2.8.2-1 Hematology (Safety Population) - Part 1

| Subject<br>Number | Study<br>Day | Was the sample collected? / If No, Reason | Date / Time of<br>Collection | Parameter (unit) | Actual<br>Value | Actual Change from Baseline <sup>[a]</sup> | Normal Range<br>(LLN-ULN) | Flag <sup>[b]</sup> | Corresponding AE ID(s) /<br>Corresponding MH ID(s) |
|---|---|---|---|---|---|---|---|---|---|
| xxxxx | Day x <sup>[a]</sup> | Yes | ddmmmyyyy / hh:mm | xxxx (xx) | xxx.x | N/A | xxx.x-xxx.x | H, CS | N/A / 1 |

Abbreviations: AE=Adverse event; CS=Clinically significant; H=Above normal range (high); ID=Identifier; L=Below normal range (low); LLN=Lower limit of normal; MH=Medical history; N=Within normal range; NCS=Not clinically significant; ULN=Upper limit of normal

#### **Programming Notes:**

- 1) Include all visits.
- 2) Include all parameters in alphabetical order.
- 3) Add abbreviations used in the table to the footnotes.

26-Oct-2023 (Final 1.0) 

<sup>[</sup>a] Baseline value; baseline is defined as the last result (scheduled or unscheduled) obtained prior to study drug administration.

<sup>[</sup>b] H, L, or N; if abnormal (H or L), CS or NCS



Bellus Health Protocol 220254 (BUS-P1-11)

# Listing 16.2.8.2-2 Hematology (Safety Population) - Part 2

| Subject<br>Number | Study<br>Day | Was the sample collected? / If No, Reason | Date / Time of<br>Collection | Parameter (unit) | Actual<br>Value | Actual Change from Baseline <sup>[a]</sup> | Normal Range<br>(LLN-ULN) | Flag <sup>[b]</sup> | Corresponding AE ID(s) /<br>Corresponding MH ID(s) |
|---|---|---|---|---|---|---|---|---|---|
| xxxxx | Day x <sup>[a]</sup> | Yes | ddmmmyyyy / hh:mm | xxxx (xx) | xxx.x | N/A | xxx.x-xxx.x | H, CS | N/A / 1 |

Abbreviations: AE=Adverse event; CS=Clinically significant; H=Above normal range (high); ID=Identifier; L=Below normal range (low); LLN=Lower limit of normal; MH=Medical history; N=Within normal range; NCS=Not clinically significant; ULN=Upper limit of normal

#### **Programming Notes:**

- 1) Include all visits.
- 2) Include all parameters in alphabetical order.
- 3) Add abbreviations used in the table to the footnotes.

26-Oct-2023 (Final 1.0) 

<sup>[</sup>a] Baseline value; baseline is defined as the last result (scheduled or unscheduled) obtained prior to study drug administration.

<sup>[</sup>b] H, L, or N; if abnormal (H or L), CS or NCS



Bellus Health Protocol 220254 (BUS-P1-11)

## **Listing 16.2.8.3-1 Coagulation (Safety Population) - Part 1**

| Subject<br>Number | Study<br>Day | Was the sample collected? / If No, Reason | Date / Time of<br>Collection | Parameter (unit) | Actual<br>Value | Actual Change from Baseline <sup>[a]</sup> | Normal Range<br>(LLN-ULN) | Flag <sup>[b]</sup> | Corresponding AE ID(s) /<br>Corresponding MH ID(s) |
|---|---|---|---|---|---|---|---|---|---|
| xxxxx | Day x <sup>[a]</sup> | Yes | ddmmmyyyy / hh:mm | xxxx (xx) | xxx.x | N/A | xxx.x-xxx.x | H, CS | N/A / 1 |

Abbreviations: AE=Adverse event; CS=Clinically significant; H=Above normal range (high); ID=Identifier; L=Below normal range (low); LLN=Lower limit of normal; MH=Medical history; N=Within normal range; NCS=Not clinically significant; ULN=Upper limit of normal

#### **Programming Notes:**

- 1) Include all visits.
- 2) Include all parameters in alphabetical order.
- 3) Add abbreviations used in the table to the footnotes.

26-Oct-2023 (Final 1.0) 

<sup>[</sup>a] Baseline value; baseline is defined as the last result (scheduled or unscheduled) obtained prior to study drug administration.

<sup>[</sup>b] H, L, or N; if abnormal (H or L), CS or NCS



Bellus Health Protocol 220254 (BUS-P1-11)


## Listing 16.2.8.3-2 Coagulation (Safety Population) - Part 2

| Subject<br>Number | Study<br>Day | Was the sample collected? / If No, Reason | Date / Time of<br>Collection | Parameter (unit) | Actual<br>Value | Actual Change from Baseline <sup>[a]</sup> | Normal Range<br>(LLN-ULN) | Flag <sup>[b]</sup> | Corresponding AE ID(s) /<br>Corresponding MH ID(s) |
|---|---|---|---|---|---|---|---|---|---|
| xxxxx | Day x <sup>[a]</sup> | Yes | ddmmmyyyy / hh:mm | xxxx (xx) | xxx.x | N/A | XXX.X-XXX.X | H, CS | N/A / 1 |

Abbreviations: AE=Adverse event; CS=Clinically significant; H=Above normal range (high); ID=Identifier; L=Below normal range (low); LLN=Lower limit of normal; MH=Medical history; N=Within normal range; NCS=Not clinically significant; ULN=Upper limit of normal

#### **Programming Notes:**

- 1) Include all visits.
- 2) Include all parameters in alphabetical order.
- 3) Add abbreviations used in the table to the footnotes.

26-Oct-2023 (Final 1.0)

<sup>[</sup>a] Baseline value; baseline is defined as the last result (scheduled or unscheduled) obtained prior to study drug administration.

<sup>[</sup>b] H, L, or N; if abnormal (H or L), CS or NCS



Bellus Health Protocol 220254 (BUS-P1-11)

## Listing 16.2.8.4-1 Urinalysis: Quantitative (Safety Population) - Part 1

| Subject<br>Number | Study<br>Day | Was the sample collected? / If No, Reason | Date / Time of<br>Collection | Parameter (unit) | Actual<br>Value | Actual Change from Baseline <sup>[a]</sup> | Normal Range<br>(LLN-ULN) | Flag <sup>[b]</sup> | Corresponding AE ID(s) /<br>Corresponding MH ID(s) |
|---|---|---|---|---|---|---|---|---|---|
| xxxxx | Day x <sup>[a]</sup> | Yes | ddmmmyyyy / hh:mm | xxxx (xx) | xxx.x | N/A | xxx.x-xxx.x | H, CS | N/A / 1 |

Abbreviations: AE=Adverse event; CS=Clinically significant; H=Above normal range (high); ID=Identifier; L=Below normal range (low); LLN=Lower limit of normal; MH=Medical history; N=Within normal range; NCS=Not clinically significant; ULN=Upper limit of normal

#### **Programming Notes:**

- 1) Include all visits.
- 2) Include all parameters in alphabetical order.
- 3) Add abbreviations used in the table to the footnotes.

26-Oct-2023 (Final 1.0) 

<sup>[</sup>a] Baseline value; baseline is defined as the last result (scheduled or unscheduled) obtained prior to study drug administration.

<sup>[</sup>b] H, L, or N; if abnormal (H or L), CS or NCS



Bellus Health Protocol 220254 (BUS-P1-11)

## Listing 16.2.8.4-2 Urinalysis: Quantitative (Safety Population) - Part 2

| Subject<br>Number | Study<br>Day | Was the sample collected? / If No, Reason | Date / Time of<br>Collection | Parameter (unit) | Actual<br>Value | Actual Change from Baseline <sup>[a]</sup> | Normal Range<br>(LLN-ULN) | Flag <sup>[b]</sup> | Corresponding AE ID(s) /<br>Corresponding MH ID(s) |
|---|---|---|---|---|---|---|---|---|---|
| xxxxx | Day x <sup>[a]</sup> | Yes | ddmmmyyyy / hh:mm | xxxx (xx) | xxx.x | N/A | xxx.x-xxx.x | H, CS | N/A / 1 |

Abbreviations: AE=Adverse event; CS=Clinically significant; H=Above normal range (high); ID=Identifier; L=Below normal range (low); LLN=Lower limit of normal; MH=Medical history; N=Within normal range; NCS=Not clinically significant; ULN=Upper limit of normal

#### **Programming Notes:**

- 1) Include all visits.
- 2) Include all parameters in alphabetical order.
- 3) Add abbreviations used in the table to the footnotes.

26-Oct-2023 (Final 1.0) 

<sup>[</sup>a] Baseline value; baseline is defined as the last result (scheduled or unscheduled) obtained prior to study drug administration.

<sup>[</sup>b] H, L, or N; if abnormal (H or L), CS or NCS



Bellus Health Protocol 220254 (BUS-P1-11)


## Listing 16.2.8.5-1 Urinalysis: Categorical (Safety Population) - Part 1

| Subject<br>Number | Study Day | Was the sample collected? /<br>If No, Reason | Date / Time of Collection | Parameter (unit) | Result | Normal Range<br>(LLN-ULN) | Flag <sup>[a]</sup> | Corresponding AE ID(s) /<br>Corresponding MH ID(s) |
|---|---|---|---|---|---|---|---|---|
| xxxxx | Day x | Yes | ddmmmyyyy / hh:mm | xxxx (xx) | Trace | xxx.x-xxx.x | CS | N/A / 1 |

Abbreviations: AE=Adverse event; CS=Clinically significant; ID=Identifier; LLN=Lower limit of normal; MH=Medical history; NCS=Not clinically significant; ULN=Upper limit of normal <sup>[a]</sup> CS or NCS

## **Programming Notes:**

- 1) Include all visits.
- 2) Include all categorical parameters in alphabetical order.
- 3) Add abbreviations used in the table to the footnotes.

26-Oct-2023 (Final 1.0)



Bellus Health Protocol 220254 (BUS-P1-11)

## Listing 16.2.8.5-2 Urinalysis: Categorical (Safety Population) - Part 2

| Subject<br>Number | Study Day | Was the sample collected? /<br>If No, Reason | Date / Time of Collection | Parameter (unit) | Result | Normal Range<br>(LLN-ULN) | Flag <sup>[a]</sup> | Corresponding AE ID(s) /<br>Corresponding MH ID(s) |
|---|---|---|---|---|---|---|---|---|
| xxxxx | Day x | Yes | ddmmmyyyy / hh:mm | xxxx (xx) | Trace | xxx.x-xxx.x | CS | N/A / 1 |

Abbreviations: AE=Adverse event; CS=Clinically significant; ID=Identifier; LLN=Lower limit of normal; MH=Medical history; NCS=Not clinically significant; ULN=Upper limit of normal <sup>[a]</sup> CS or NCS

## **Programming Notes:**

- 1) Include all visits.
- 2) Include all categorical parameters in alphabetical order.
- 3) Add abbreviations used in the table to the footnotes.

26-Oct-2023 (Final 1.0) 



Bellus Health Protocol 220254 (BUS-P1-11)

# Listing 16.2.8.6-1 Vital Signs (Safety Population) - Part 1

| Subject<br>Number | Study<br>Day | Was the assessment performed? / If No, Reason | Date / Time of Assessment | Parameter (unit) | Actual Value | Normal Range | Actual Change<br>from Baseline <sup>[a]</sup> | Interpretation <sup>[b]</sup> |
|---|---|---|---|---|---|---|---|---|
| xxxxx | Day x <sup>[a]</sup> | Yes | ddmmmyyyy / hh:mm | xxxx (xx) | xxx | xxx-xxx | N/A | Normal |

Abbreviations: CS=Clinically significant; NCS=Not clinically significant

## Programming Notes:

- 1) Include all visits.
- 2) Include all parameters.
- 3) Add abbreviations used in the table to the footnotes.

26-Oct-2023 (Final 1.0) 

<sup>[</sup>a] Baseline value; baseline is defined as the last result (scheduled or unscheduled) obtained prior to study drug administration.
[b] Normal or abnormal, if abnormal, CS or NCS



Bellus Health Protocol 220254 (BUS-P1-11)

# Listing 16.2.8.6-2 Vital Signs (Safety Population) - Part 2

| Subject<br>Number | Study<br>Day | Was the assessment performed? / If No, Reason | Date / Time of Assessment | Parameter (unit) | Actual Value | Normal Range | Actual Change<br>from Baseline <sup>[a]</sup> | Interpretation <sup>[b]</sup> |
|---|---|---|---|---|---|---|---|---|
| xxxxx | Day x <sup>[a]</sup> | Yes | ddmmmyyyy / hh:mm | xxxx (xx) | xxx | xxx-xxx | N/A | Normal |

Abbreviations: CS=Clinically significant; NCS=Not clinically significant

## Programming Notes:

- 1) Include all visits.
- 2) Include all parameters.
- 3) Add abbreviations used in the table to the footnotes.

26-Oct-2023 (Final 1.0) 

<sup>[</sup>a] Baseline value; baseline is defined as the last result (scheduled or unscheduled) obtained prior to study drug administration.
[b] Normal or abnormal, if abnormal, CS or NCS



Bellus Health Protocol 220254 (BUS-P1-11)

## Listing 16.2.8.7-1 ECGs (Safety Population) - Part 1

| Subject<br>Number | Study<br>Day | Was the assessment performed? / If No, Reason | Date / Time of Assessment | ECG Position | Parameter (unit) | Actual Value | Normal Range | Actual Change<br>from Baseline <sup>[a]</sup> | Overall<br>Interpretation <sup>[b]</sup> |
|---|---|---|---|---|---|---|---|---|---|
| xxxxx | Day x <sup>[a]</sup> | Yes | ddmmmyyyy / hh:mm | Supine | xxxx (xx) | xxx | xxx-xxx | N/A | Normal |

## Programming Notes:

- 1) Include all visits.
- 2) Include all parameters.
- 3) Add abbreviations used in the table to the footnotes.

26-Oct-2023 (Final 1.0) 

Abbreviations: CS=Clinically significant; ECG=Electrocardiogram; NCS=Not clinically significant [a] Baseline value; baseline is defined as the last result (scheduled or unscheduled) obtained prior to study drug administration.

<sup>[</sup>a] Normal or abnormal, if abnormal, CS or NCS.



Bellus Health Protocol 220254 (BUS-P1-11)

# **Listing 16.2.8.7-2 ECGs (Safety Population) - Part 2**

| Subject<br>Number | Study<br>Day | Was the assessment<br>performed? /<br>If No, Reason | Date / Time of Assessment | ECG Position | Parameter (unit) | Actual Value | Normal Range | Actual Change<br>from Baseline <sup>[a]</sup> | Overall<br>Interpretation <sup>[b]</sup> |
|---|---|---|---|---|---|---|---|---|---|
| xxxxx | Day x <sup>[a]</sup> | Yes | ddmmmyyyy / hh:mm | Supine | xxxx (xx) | xxx.x | xxx-xxx | N/A | Normal |
| ••• | | | | | | | | | |

### Programming Notes:

- 1) Include all visits.
- 2) Include all parameters.3) Add abbreviations used in the table to the footnotes.

26-Oct-2023 (Final 1.0) 

Abbreviations: CS=Clinically significant; ECG=Electrocardiogram; NCS=Not clinically significant [a] Baseline value; baseline is defined as the last result (scheduled or unscheduled) obtained prior to study drug administration. [b] Normal or abnormal, if abnormal, CS or NCS.



Bellus Health Protocol 220254 (BUS-P1-11)

# **Listing 16.2.8.8-1 Physical Examination (Safety Population) - Part 1**

| Subject<br>Number | Study<br>Day | Assessment Type <sup>[a]</sup> | Was the assessment performed? / If No, Reason | Date / Time of<br>Assessment | Body System | Result <sup>[b]</sup> | Abnormal Findings |
|---|---|---|---|---|---|---|---|
| xxxxx | Day x | Complete | Yes | ddmmmyyyy / hh:mm | HEENT | Normal | N/A |

Abbreviations: CS=Clinically significant; NCS=Not clinically significant [a] Brief or complete [b] Normal or abnormal; if abnormal: CS or NCS

## Programming Notes:

- 1) Include all visits.
- 2) Include all body systems.
- 3) Add abbreviations used in the table to the footnotes.
  - a. HEENT= head, eyes, ears, nose, and throat

26-Oct-2023 (Final 1.0) 



Bellus Health Protocol 220254 (BUS-P1-11)

# Listing 16.2.8.8-2 Physical Examination (Safety Population) - Part 2

| Subject<br>Number | Study Day | Assessment Type <sup>[a]</sup> | Was the assessment performed? / If No, Reason | Date / Time of<br>Assessment | Body System | Result <sup>[b]</sup> | Abnormal Findings |
|---|---|---|---|---|---|---|---|
| xxxxx | Day x | Complete | Yes | ddmmmyyyy / hh:mm | HEENT | Normal | N/A |
| ••• | | | | | | | |

Abbreviations: CS=Clinically significant; NCS=Not clinically significant

## Programming Notes:

- 1) Include all visits.
- 2) Include all body systems.
- 3) Add abbreviations used in the table to the footnotes.
  - a. HEENT= head, eyes, ears, nose, and throat

26-Oct-2023 (Final 1.0) 

<sup>[</sup>a] Brief or complete
[b] Normal or abnormal; if abnormal: CS or NCS



Bellus Health Protocol 220254 (BUS-P1-11)

# Listing 16.2.8.8-3 Pharmacogenomic Measurements (Pharmacogenomic Population) - Part 1

| Subject Number | Study Day | Date / Time of Sample Collection | Result | Unit |
|---|---|---|---|---|
| xxxxx | Day x | ddmmmyyyy / hh:mm | xx | XX |

26-Oct-2023 (Final 1.0) 



Bellus Health Protocol 220254 (BUS-P1-11)

# Listing 16.2.8.8-4 Pharmacogenomic Measurements (Pharmacogenomic Population) - Part 2

| Subject Number | Study Day | Date / Time of Sample Collection | Result | Unit |
|---|---|---|---|---|
| xxxxx | Day x | ddmmmyyyy / hh:mm | XX | xx |
| ••• | | | | |

26-Oct-2023 (Final 1.0) 